# Statistical Analysis Plan



| Sponsor | Arcutis Biotherapeutics, Inc. |
|---|---|
| Protocol Title: | A Phase 2b, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-154 Foam 0.3% Administered QD in Adolescents and Adults with Scalp and Body Psoriasis |
| Protocol Number: | ARQ-154-204 |
| Premier Research PCN: | ARCU210101 |
| Document Version: | Final 2.0 |
| Document Date: | 09-Dec-2020 |

## Approvals

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| | Print Name: | |
| Lead<br>Biostatistician | Sign Name: | 09-Dec-2020 06:20:07 EST |
| | Print Name: | |
| | Sign Name: | |
| Premier Senior<br>Reviewer | | 09-Dec-2020 08:35:32 EST |
| | Print Name: | |
| Arcutis Biotherapeutics, Inc. Representative | Sign Name: | 09-Dec-2020 14:14:38 PST |





## **Document History**

| Version | Date | Section | Description of Change/Purpose |
|---|---|---|---|
| 1.0 | 12-Nov-2020 | N/A | N/A |
| 2.0 | 04-Dec-2020 | 8.1 | Text from this section describing the primary endpoint analysis (including sensitivity analysis) was accidentally removed when accepting changes from the redlined version of SAP draft v0.3. This text was not in redline, so the deletion was unexpected and therefore not noticed once the draft was upversioned to final v1.0. The exact text from draft v0.3 was copied back into the SAP; no other changes were made to the SAP. |





## **Table of Contents**

| Ap | provals | | 1 |
|-----|----------|--------------------------------------------------|------|
| Do | cument | History | 2 |
| Tal | ble of C | ontents | 3 |
| Lis | t of Tal | oles | 5 |
| Lis | t of Fig | ures | 5 |
| 1. | Ov | erview | 6 |
| 2. | Stu | dy Objectives and Endpoints | 6 |
| | 2.1. | Study Objectives | 6 |
| | 2.1.1. | Primary Objective | 6 |
| | 2.2. | Study Endpoints | 6 |
| | 2.2.1. | Safety Endpoints | 6 |
| | 2.2.2. | Efficacy Endpoints | 7 |
| 3. | Ov | erall Study Design and Plan | 8 |
| | 3.1. | Overall Design | 8 |
| | 3.2. | Sample Size and Power | |
| | 3.3. | Study Population | 9 |
| | 3.4. | Treatments Administered | 9 |
| | 3.5. | Method of Assigning Subjects to Treatment Groups | |
| | 3.6. | Blinding and Unblinding | 9 |
| | 3.7. | Schedule of Events | |
| 4. | Sta | tistical Analysis and Reporting | . 11 |
| | 4.1. | Introduction | . 11 |
| | 4.2. | Interim Analysis and Data Monitoring | . 11 |
| 5. | | alysis Populations | |
| 6. | | neral Issues for Statistical Analysis | |
| | 6.1. | Statistical Definitions and Algorithms | . 12 |
| | | Baseline | |
| | 6.1.2. | Adjustments for Covariates | . 13 |
| | 6.1.3. | Multiple Comparisons | |
| | 6.1.4. | Handling of Dropouts or Missing Data | |
| | 6.1.5. | Analysis Visit Windows | |
| | | Pooling of Sites | |
| | | Derived Variables | |
| | 6.1.8. | Data Adjustments/Handling/Conventions | |
| | 6.2. | Special Handling for COVID-19 Disruptions | |
| 7. | Stu | dy Subjects and Demographics | . 23 |





| | 7.1. | Disposition of Subjects and Withdrawals | 23 |
|-----|---------|-------------------------------------------------------|----|
| | 7.2. | Protocol Deviations. | 23 |
| | 7.3. | Demographics and Other Baseline Characteristics | 23 |
| | 7.4. | Exposure and Compliance | |
| 8. | Eff | ficacy Analysis | 24 |
| | 8.1. | Primary Efficacy Analysis | 24 |
| | 8.1.1. | Scalp Investigator Global Assessment (S-IGA) | 24 |
| | 8.2. | Secondary Efficacy Analysis | 26 |
| | 8.2.1. | Body Investigator Global Assessment (B-IGA) | 27 |
| | 8.2.2. | Psoriasis Scalp Severity Index (PSSI) | 27 |
| | 8.2.3. | Scalp Itch – Numeric Rating Scale (SI-NRS) | 28 |
| | 8.2.4. | Psoriasis Symptoms Diary (PSD) | 28 |
| | 8.3. | Exploratory Efficacy Analysis | 28 |
| 9. | Sat | fety and Tolerability Analysis | 29 |
| | 9.1. | Adverse Events | 29 |
| | 9.1.1. | Adverse Events Leading to Withdrawal | 30 |
| | 9.1.2. | Deaths and Serious Adverse Events | 30 |
| | 9.2. | Local Tolerability Assessments | 30 |
| | 9.3. | Clinical Laboratory Evaluations | 30 |
| | 9.4. | Vital Signs | 30 |
| | 9.5. | PHQ-8 and Modified PHQ-A | 31 |
| | 9.6. | C-SSRS | 31 |
| | 9.7. | Physical Examination | 31 |
| | 9.8. | Concomitant Medication | 31 |
| 10. | Ch | anges from Planned Analysis | 32 |
| 11. | Otl | her Planned Analysis | 33 |
| | 11.1. | Pharmacokinetic Analysis | 33 |
| 12. | Re | ferences | 33 |
| 13. | Tal | bles, Listings, and Figures | 34 |
| | 13.1. | Planned Table Descriptions | 34 |
| | 13.1.1. | Demographic Data | 34 |
| | 13.1.2. | Efficacy Data | 34 |
| | 13.1.3. | Safety Data | 40 |
| | 13.2. | Planned Listing Descriptions | 42 |
| 14. | Tal | ble, Listing, and Figure Shells | 44 |
| | 14.1. | Standard Layout for all Tables, Listings, and Figures | |
| | 14.2. | Planned Table Shells | 46 |





| Appendix 1: Premier Research Library of Abbreviations | |
|-------------------------------------------------------|----|
| List of Tables | |
| Table 1: Schedule of Events | |
| Table 2: Analysis Visit Windows | 17 |
| Table 3: S-IGA | 24 |
| Table 4: Demographic Data Summary Tables | 34 |
| Table 5: Efficacy Data Summary Tables | 34 |
| Table 6: Safety Data Summary Tables | 40 |
| Table 7: Planned Listings | 42 |
| List of Figures | |
| Figure 1: Primary and Secondary Endpoint Testing | 14 |
| Figure 2: Standardized Layout | 45 |
| Figure 3: Planned Table Shells | 47 |



#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Arcutis Biotherapeutics, Inc. protocol number ARQ-154-204 (A Phase 2b, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-154 Foam 0.3% Administered QD in Adolescents and Adults with Scalp and Body Psoriasis), dated 13-Jan-2020 Amendment Version 1.0. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>1</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>3</sup> and the Royal Statistical Society<sup>1</sup>, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to Arcutis Biotherapeutics, Inc.'s study ARQ-154-204. Any amendments to this plan that occur after unblinding for an interim analysis will be performed by a study statistician who remains blinded to treatment codes and outcomes.

ARQ-154 foam 0.3% will be described as "roflumilast foam 0.3%" throughout this document and the tables, listings, and figures (TLFs).

## 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

#### 2.1.1. Primary Objective

The primary objective is to assess the safety and efficacy of roflumilast foam 0.3% vs vehicle administered daily (QD) x 8 weeks in adolescents and adults with scalp and body plaque psoriasis.

#### 2.2. Study Endpoints

#### 2.2.1. Safety Endpoints

The safety endpoints of this study include the following:

Local tolerability assessments



- Clinical laboratory parameters
- Adverse events (AEs)
- Columbia-Suicide Severity Rating Scale (C-SSRS)
- Patient Health Questionnaire depression scale (PHQ-8)
- Modified PHQ-Adolescents (PHQ-A)
- Vital signs
- Physical examinations

## 2.2.2. Efficacy Endpoints

#### 2.2.2.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is Scalp-Investigator Global Assessment (S-IGA) Success at Week 8, defined as achievement of an S-IGA score of "Clear" or "Almost Clear" plus a 2-grade improvement from baseline.

## 2.2.2.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints of this study include the following:

- Body-IGA (B-IGA) Success at Week 8, defined as achievement of B-IGA score of "Clear" or "Almost Clear" plus a 2-grade improvement from baseline
- Psoriasis Scalp Severity Index (PSSI)-75 (subjects who achieve a 75% reduction in PSSI from Baseline) at Week 8
- For subjects with baseline Scalp Itch Numeric Rating Scale (SI-NRS) score ≥4, achievement of ≥4-point improvement from baseline in SI-NRS at Week 8
- For subjects with baseline SI-NRS score ≥4, achievement of ≥4-point improvement from baseline in SI-NRS at Week 4
- For subjects with baseline SI-NRS score ≥4, achievement of ≥4-point improvement from baseline in SI-NRS at Week 2
- Time to success in PSSI-50
- Change and percent change from baseline in total Psoriasis Symptoms Diary (PSD) score at Week 8
- Change and percent change from baseline in total PSD score at Week 4
- PSSI-90 (subjects who achieve a 90% reduction in PSSI from Baseline) at Week 8

#### 2.2.2.3. Exploratory Efficacy Endpoints

The exploratory efficacy endpoints of this study include the following:

- Psoriasis Area Severity Index (PASI)-75 (subjects who achieve a 75% reduction in PASI from Baseline) at Week 8
- Time to success in PASI-50
- Change and percent change from baseline modified PASI (mPASI) at Weeks 2, 4, 8, and 9
- For subjects with baseline Worst Itch Numeric Rating Scale (WI-NRS) score ≥4, achievement of ≥4-point improvement from baseline in WI-NRS at Weeks 2, 4, and 8
- Change and percent change from baseline in Dermatology Life Quality Index (DLQI)/ Children's DLQI (CDLQI) total scores at Weeks 2, 4, and 8



• Change and percent change from baseline in % BSA affected by disease at Weeks 2, 4, and 8

The exploratory endpoints below are not defined in the protocol explicitly but are based on other efficacy assessments collected:

- Change and percent change from baseline in SI-NRS at Weeks 2, 4, and 8
- Change and percent change from baseline in PASI at Weeks 2, 4, 8, and 9
- PASI-90 (subjects who achieve a 90% reduction in PASI from Baseline), PASI-75 (subjects who achieve a 75% reduction in PASI from Baseline), and PASI-50 (subjects who achieve a 50% reduction in PASI from Baseline) at Weeks 2, 4, 8, and 9
- Change and percent change from baseline in WI-NRS at Weeks 2, 4, and 8

## 3. Overall Study Design and Plan

#### 3.1. Overall Design

This is a parallel group, double blind, vehicle-controlled study in which roflumilast foam 0.3% or vehicle foam is applied QD x 8 weeks to adolescent and adults with scalp and body psoriasis of at least mild severity (S-IGA and B-IGA with a score of at least "2"), involving up to 25% body surface area (BSA) (scalp and body, not including palms/soles).

Approximately 300 subjects will be enrolled. After having met all inclusion criteria, and none of the exclusion criteria, subjects will be randomized in a 2:1 ratio to roflumilast foam 0.3% QD or vehicle foam QD, which will be applied to all psoriasis lesions (including the scalp, face, trunk, and intertriginous areas; palms and soles will be treated but will not be counted towards any measurements of efficacy). Screening will be for up to 4 weeks followed by an 8-week Treatment Phase, with a Follow-up Visit 1 week after last dose. The anticipated maximum duration of subject participation is approximately 13 weeks.

Subjects will have to apply the study drug once a day in the evening, with the exception of Day 0, Week 2 (Visit 3), and Week 4 (Visit 4), when the study drug is applied at the study site in the morning. Participants have to record the date and time each dose has been applied with details including missed doses and any additional comments.

#### 3.2. Sample Size and Power

There are approximately 300 subjects planned for this study. Approximately 200 subjects will receive roflumilast foam 0.3% QD; approximately 100 subjects will receive vehicle foam QD. The sample size was selected to provide an adequate number of subjects to compare the efficacy of roflumilast treatment to vehicle and to provide an adequate number of subjects needed for a safety database.

This sample size provides 96% power at the  $\alpha$ =0.05 level to detect a 22.4% difference between treatment groups for S-IGA Success at Week 8 using a 2-sided Chi-squared test. The results from a recent phase 2b study (ARQ-151-201) of roflumilast cream compared to vehicle treatment were used to estimate the treatment difference, and it is assumed that the S-IGA response in the present study are similar to IGA responses seen with roflumilast cream. Specifically, in the phase 2b trial, 32.2% of subjects reported IGA success in the roflumilast cream 0.3% group and 9.8% of subjects reported IGA success in the vehicle group.

The number of subjects to be enrolled will also provide sufficient power for most secondary

**premier** research

endpoints.

#### 3.3. Study Population

Study population consists of male and female subjects aged 12 years or older with no more than 25% BSA of scalp and body psoriasis. Subjects should have a minimum S-IGA of at least "Moderate" (3) and B-IGA of "Mild" (2) at Baseline. Note that the original protocol allowed subjects having an S-IGA of "Mild" (2) to be enrolled, and some subjects were enrolled and treated with an S-IGA of "Mild" before the amendment under which this SAP operates was put into effect (i.e., Amendment Version 1.0, dated 13-Jan-2020).

#### 3.4. Treatments Administered

Subjects who meet the eligibility criteria will be randomized to 1 of the 2 following treatment groups in a 2:1 ratio (active:vehicle):

- Roflumilast foam 0.3% QD
- Matching vehicle foam QD.

#### 3.5. Method of Assigning Subjects to Treatment Groups

Subjects will be randomized and assigned to active drug or vehicle will be made at a 2:1 ratio according to a computer-generated randomization list. Randomization will be stratified by country, baseline S-IGA (S-IGA=2 vs. S-IGA  $\geq$ 3), and baseline B-IGA (B-IGA=2 vs. B-IGA  $\geq$ 3).

#### 3.6. Blinding and Unblinding

This is a double-blind study; therefore, neither the subjects nor the investigator, clinical personnel, or sponsor will be aware of which treatment a subject has received. Emergency unblinding will be done using the study internet-based randomization system (interactive webresponse system; IWRS) system in consultation with the medical monitor and the sponsor's chief medical officer (CMO).

#### 3.7. Schedule of Events

A detailed schedule of events for the study is provided in Table 1.



#### **Table 1: Schedule of Events**

| Study Procedure | Screen | Baseline<br>Day 0 | Wk 2<br>Day 14 | Wk 4<br>Day 28 | Wk 8<br>Day 56 | Wk 9<br>Day 63 |
|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 |
| Visit Window | -4 weeks | 2 | +/- 3 days | +/- 5 days | +/- 5 days | +/- 5 days |
| Informed consent/assent | X | | | v | · | · |
| Medical history | X | | | | | |
| Physical examination <sup>a</sup> | X | X | | | X | |
| I/E criteria | X | X | | | | |
| Randomization | | X | | | | |
| Hematology, Serum<br>Chemistries, and Urine<br>Analysis | X | X | | X | X | |
| Vital signs, height <sup>b</sup> , weight <sup>b</sup> | X | X | X | X | X | X |
| S-IGA <sup>c</sup> , B-IGA <sup>c</sup> , PSSI <sup>c</sup> ,<br>BSA <sup>c</sup> , PASI/mPASI | X | X | X | X | X | X |
| Scalp Itch NRS, WI-NRS<br>pruritus, DLQI, CDLQI,<br>PSD <sup>d</sup> | X | X | X | X | X | |
| Application Site Reaction<br>Assessment/Local<br>tolerability <sup>e</sup> | | X | | X | X | |
| C-SSRS, PHQ-8/PHQ-Af | X | X | | X | X | |
| Medical Photography <sup>g</sup> | | X | X | X | X | |
| Pregnancy test <sup>h</sup> | X | X | | X | X | |
| PK draws <sup>i</sup> | | X | | X | X | |
| IP/vehicle application in clinic <sup>j</sup> | | X | X | X | | |
| Dispense IP kit <sup>k</sup> | | X | X | X | | |
| Dispense/review diary | | X | X | X | X | |
| Weigh IP kit <sup>l</sup> | | X | X | X | X | |
| Compliance calculation <sup>m</sup> | | X | X | X | X | |
| Adverse event assessment <sup>n</sup> | X | X | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X |

#### Footnote:

- <sup>a</sup> Limited physical examination: skin, lungs, and heart only
- b Height will be collected at Baseline and Week 8. Weight will be collected at all study visits. Subject to void prior to weight being taken. Remove any jackets, outerwear and shoes. Remove any objects of significant weight (i.e. cell phones, wallet, key chains). A 5% unintentional weight loss should be reported to the medical monitor.
- c S-IGA will be a 5-point scale ranging from clear (0) to severe (4) and is evaluated for the scalp only. B-IGA will use the same scale as S-IGA, but will evaluate the entire body (except the scalp, palms, and soles). PSSI is scored on a 0-72 scale and evaluates the scalp only. Total BSA and scalp BSA affected by psoriasis will be determined (except the palms and soles). PASI/mPASI assessment should exclude palms and soles. S-IGA and B-IGA should be completed prior to other physician assessments.
- d. Subjects will complete the WI-NRS pruritus, Scalp Itch-NRS, DLQI, CDLQI (for adolescents) and PSD questionnaires.
- <sup>e.</sup> Local Tolerability Assessments: the Investigator local tolerability assessment of skin irritation (Berger and Bowman skin irritation score) should be performed prior to the investigational product application at Day 0, Weeks 4 and 8. **Note for**





investigator tolerability assessments: reactions at the site of product application, which may occur post-Baseline, should be differentiated from the preexisting inflammation associated with the subject's psoriasis. Subjects will perform the local tolerability 10-15 minutes post-IP application at Day 0 and Week 4, and recall assessment at Week 8 for the subject's '0-3' burning/stinging assessment.

- f Adolescents and adults will complete the C-SSRS. Adults will complete the PHQ-8. Adolescents will complete a modified version of the PHQ-A (PHQ-9 modified for Adolescents).
- g At selected sites, medical photography will be obtained for target lesions. All efforts will be made to de-identify the subjects. Subjects who are unwilling to participate in the medical photography will be allowed to opt out of this procedure.
- h A pregnancy test will be administered to all females of child-bearing potential. A serum pregnancy test will be performed at the Screening visit only. A urine pregnancy test will be performed at Day 0, Week 4, and Week 8. A negative result is required for continued participation in the study, and results must be available prior to dispensing of the IP at each visit.
- <sup>1</sup> PK draws will be collected at Days 0, Weeks 4 and 8 pre-dose (within 1 hour) for all subjects. Serial PK will be obtained in a subset of approximately 15 subjects on Days 0 and 28 at 1, 2, 4, 6 (all + 20 min), and 24 hours (+ 2 hours) post-dose
- <sup>j</sup> Subjects to apply assigned IP in clinic at Day 0, Weeks 2 and 4.
- <sup>k</sup> Kits will be dispensed based on %BSA affected. See IP Handling Manual for details.
- <sup>1</sup> The entire kit should be weighed and recorded at every visit. See IP Handling Manual for details.
- <sup>m</sup> Compliance calculation is described in the IP Handling Manual
- <sup>n</sup> Any emergent AEs will be followed in the clinic for up to one month at the Investigator's discretion until resolved or otherwise judged as clinically stable.

## 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations, will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted for analyses conducted by Premier Research, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with nonmissing values, mean, standard deviation (SD), median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment group, unless otherwise specified.

Unless otherwise indicated, all statistical tests will be conducted at the familywise  $\alpha$ =0.05 significance level using 2-tailed tests, and P values will be reported. Corresponding 95% confidence intervals (CIs) will be presented for statistical tests. Details for splitting the familywise  $\alpha$  to control for multiple comparisons will be discussed in Section 6.1.3.

#### 4.2. Interim Analysis and Data Monitoring

No interim efficacy analyses are planned.



#### 5. Analysis Populations

The following analysis populations are planned for this study:

- Safety Population (SAF): The Safety population will include all subjects who are enrolled and received at least 1 confirmed dose of investigational product (IP). This population will be used for all safety analyses.
- Intent-To-Treat Population (ITT): The ITT population will include all randomized subjects. This population will be the primary analysis population for the analysis of efficacy endpoints, along with subject disposition.
- Modified Intent-To-Treat Population (mITT): The mITT population includes all randomized subjects with the exception of subjects who missed the Week 8 S-IGA assessment specifically due to novel coronavirus disease-19 (COVID-19) disruptions. This population will be the sensitivity analysis population for the analysis of primary and secondary efficacy endpoints.
- Scalp Pruritus ITT Population (SPRU4-ITT): The SPRU4-ITT population is a subset of the ITT population and includes subjects with SI-NRS score ≥4 at baseline. This population will be used for the analysis of achievement of a 4-point reduction in SI-NRS score as compared to baseline for this subset of ITT subjects.
- Scalp Pruritus mITT Population (SPRU4-mITT): The SPRU4-mITT population is a subset of the mITT population and includes subjects with SI-NRS score ≥4 at baseline. This population will be used for the analysis of achievement of a 4-point reduction in SI-NRS score as compared to baseline for this subset of mITT subjects.
- **Pruritus ITT Population (PRU4-ITT):** The PRU4-ITT population is a subset of the ITT population and includes subjects with WI-NRS score ≥4 at baseline. This population will be used for the analysis of achievement of a 4-point reduction in WI-NRS score as compared to baseline for this subset of ITT subjects.
- **Pruritus mITT Population (PRU4-mITT):** The PRU4-mITT population is a subset of the mITT population and includes subjects with WI-NRS score ≥4 at baseline. This population will be used for the analysis of achievement of a 4-point reduction in WI-NRS score as compared to baseline for this subset of mITT subjects.
- **Pharmacokinetic Population (PK):** The PK population will include all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist. This population will be used for analyses of PK parameters.

#### 6. General Issues for Statistical Analysis

## **6.1.** Statistical Definitions and Algorithms

#### 6.1.1. Baseline

For most efficacy assessments (i.e., S-IGA, B-IGA, PSSI, PASI/mPASI, and % BSA) and all safety assessments except PHQ-8/PHQ-A, the last observation recorded before the first application of study drug will be used as the baseline observation for all calculations of change





from baseline. For other efficacy and safety assessments with a 24-hour or greater recall period (i.e., SI-NRS, WI-NRS, PSD, DLQI/CDLQI, and PHQ-8/PHQ-A), for the previously-named assessments where time is missing (and therefore we are assuming that the assessment was collected before first dose of study drug as per the protocol), or for subject local tolerability (which is expected to be post-dose), the last observation recorded on or before the day of first application of study drug will be used as the baseline observation for all calculations of change from baseline.

For assessments that are collected both before and after application of study drug at the Baseline Day 0 visit, the last observation recorded before the first dose of study will be used as the baseline observation. For assessments collected only after application of study drug, no baseline will be defined (except for subject local tolerability). If the tolerability assessments are not done as per protocol Section 5.1.8, those records will be excluded from the analysis.

## **6.1.2.** Adjustments for Covariates

Subgroup analyses may be generated for the baseline covariates.

#### **6.1.3.** Multiple Comparisons

To control for multiple comparisons among the secondary endpoints, the following testing plan will be used, as outlined in Figure 1.

Upon demonstration of statistical significance for S-IGA Success at Week 8, the secondary endpoint of B-IGA Success at Week 8 will be tested hierarchically at the 5% significance level.

If the test for B-IGA Success at Week 8 is significant, the  $\alpha$  of 0.05 will be split to test 2 families of secondary endpoints. The first family comprise the PSSI-75, which will be tested at the  $\alpha$  = 0.03 level. If the test of PSSI-75 is statistically significant, then  $\alpha$  = 0.03 will be used with a Holm testing procedure to test the 4 endpoints of time to success in PSSI-50, change from baseline in Total PSD score at Week 8, change from baseline in Total PSD score at Week 4, and PSSI-90 at Week 8. The remaining  $\alpha$  = 0.02 will be used to test the second family, comprising the SI-NRS at Week 8, the SI-NRS at Week 4, and the SI-NRS at Week 2. The tests within this second family will be hierarchical, beginning with the endpoint at Week 8, followed by Week 4 and Week 2.



## Figure 1: Primary and Secondary Endpoint Testing



Achievement of IGA success is a score of "clear" or "almost clear" plus a 2-grade improvement from baseline. SI-WRS Success is a 4-point reduction in SI-NRS among subjects with SI-NRS  $\geq$  4 at baseline. B-IGA = Body-Investigator Global Assessment; EP = endpoint; CFB = change from baseline; PSSI = Psoriasis Scalp Severity Index; S-IGA = Scalp-Investigator Global Assessment; SI-NRS = Scalp Itch - Numeric Rating Scale.



## 6.1.4. Handling of Dropouts or Missing Data

## 6.1.4.1. Imputation of Missing Data

Any subject who prematurely withdraws from the study will have their last available data assigned to an analysis window as described in Section 6.1.5.

For the primary efficacy endpoint of S-IGA score, the primary analysis will impute missing values using a regression-based multiple imputation model. This is a three step process.

- 1. The first step is to understand the pattern of missingness. In order to perform the multiple imputation, a monotone missing pattern has to be achieved. For example, if there exists values for baseline and Week 8 visits, but missing values for the Week 2 or 4 visits, Markov-Chain Monte-Carlo (MCMC) method will be used to impute the small amount of missing data that may be missing at the intermediate visits that is required to make the missing data pattern monotone before applying the multiple imputation algorithm. This method uses a non-informative Jeffreys prior to derive the posterior mode from the expectation-maximization (EM) algorithm as the starting values for the MCMC method. MCMC method will use seed of 34978264. The S-IGA score will be treated as a continuous variable for this step. To avoid values that could not be observed in practice, imputed values will be constrained to be integers in the range of 0 to 4.
  - a. The table below will determine the number of datasets to be imputed in this step. Determine the proportion of datapoints with non-monotone pattern across all visits and subjects which could be derived as a percentage of number of nonmonotone data points/total number of expected data points.

This can be determined as  $\frac{number\ of\ non\ montone\ visits}{total\ number\ of\ visits\ across\ all\ subjects}*100$ 

| Non-monotone<br>Missing Data | Number of Imputed Datasets |
|------------------------------|----------------------------|
| ≤ 2% | 1 |
| $> 2\%$ to $\le 5\%$ | 3 |
| > 5% | 10 |

2. Once the monotone pattern is achieved, the next step is to implement the imputation algorithm. For this, the Predictive Mean Matching method (PMM) will be used. This method is particularly helpful if the normality assumption is violated. For subjects with complete data up to a particular visit, a PMM model will be fit that includes the outcome at that visit as the dependent variable and as independent variables, S-IGA score outcomes at previous visits, treatment group, and country using a seed of 51192215. This process will be repeated 25 times, resulting in a total of 25 to 250 complete analysis



datasets, depending on the number of imputed monotone datasets that are required. The seed may be changed after unblinding in case of any issues with the imputation process, and it will be documented in the CSR if any change is required.

3. For each completed dataset, compute the necessary derived variables. The dichotomous success rate (clear or almost clear with at least a 2-point change from baseline) will be derived. The results obtained will be analyzed using the Cochran-Mantel-Haenszel (CMH) analysis for each of the complete analysis data sets stratified by baseline S-IGA score category, baseline B-IGA score category, and country. The results will be combined into one multiple imputation inference (odds ratio, associated CI, and *P* value) using PROC MIANALYZE as illustrated<sup>4</sup>.

This approach to imputation should be superior to other strategies such as carrying forward the last available observation, which may yield unrealistic imputed values. Also, the use of multiple imputation avoids the problem of artificially increasing power through data imputation associated with single-imputation methods because it accounts for the uncertainty associated with the imputation. Other missing data will not be imputed, with the exception of incomplete dates as described in Section 6.1.8. For responder analyses, missing data will be treated as a nonresponse with the exception of S-IGA. Only observed data will be summarized using descriptive statistics.

The SAS pseudo code for the multiple imputation process is listed below:

#### Step 1:

```
proc mi data=example seed=34978264 nimpute=XX round=1 out=example_1;
    mcmc impute=monotone;
    var <baseline score> ............ <visit8 score>;
run;

Step 2:

proc mi data=example_1 seed=51192215 nimpute=XX out=example_2;
    class <treatment> <country>;
    monotone regpmm(<baseline score> ............ <visit8 score>);
    var <treatment> <country> <baseline score> ........... <visit8 score>;
run;

XX will be the determined based on the proportion of missing data across visits.
```

Step 3: This step involves running CMH test stratified by baseline S-IGA score category, baseline B-IGA score category, and country on each completed dataset and combining the results using PROC MIANALYZE.



In order to apply PROC MIANALYZE, normalizing transformations have to be applied to odds ratio. *P* values are obtained using Wilson Hilferty transformation as illustrated<sup>4</sup>.

#### 6.1.4.2. Tipping Point Analysis

As a sensitivity analysis to the multiple imputation analysis as described in Section 6.1.4.1 for the S-IGA primary endpoint, a tipping point analysis will be performed in order to determine the inflection point at which the inference under the MNAR assumption changes substantially. This will be used to check the robustness of the imputation.

The sensitivity analysis will be performed by using a specified sequence of shift parameters, which will adjust the imputed values for observations in the active treatment group. The range of shift parameters to be included in this analysis are -1.5 to 1.5 by 0.2. Once the likely point of the shift is determined, the analysis will be rerun using an expanded range around the suspected tipping point, with greater precision (i.e., to 2 decimal places, by 0.01). Thus, the value at which the results of the analysis are shifted from significant (i.e.,  $\alpha \le 0.05$ ) to non-significant (i.e.,  $\alpha > 0.05$ ) will be determined.

Step 1 of the analysis will be the same as for the multiple imputation analysis as described in Section 6.1.4.1. However, Step 2 of the analysis is where the shift parameters will be applied. Step 3 will be similar to the multiple imputation analysis described in Section 6.1.4.1, however, the BY statement in PROC FREQ will also include the shift parameter (i.e., by <shift parameter> <imputation number> <shift parameter> <visit>); this will also be included in the PROC MIANALYZE steps. Pseudo-code for Step 2 is as follows:

```
proc mi data=example_1 seed=51192215 nimpute=XX   out=example_2;
   class <treatment> <country> ;
   monotone regpmm(<baseline score> ............ <visit8 score>);
   var <treatment> <country> <baseline score> ........... <visit8 score>;
   mnar adjust( <visit2 score> / shift=YY adjustobs=(treatment = 'Vehicle') );
   mnar adjust( <visit4 score> / shift=YY adjustobs=(treatment = 'Vehicle') );
   mnar adjust( <visit8 score> / shift=YY adjustobs=(treatment = 'Vehicle') );
   run;
```

XX will be the determined based on the proportion of missing data across visits. YY will encompass the range of shift parameters as pre-specified above.

#### **6.1.5.** Analysis Visit Windows

Visits will be analyzed as scheduled. Unscheduled, early termination, and/or repeated measurements will only be included if a scheduled measurement is not available and the unscheduled, early termination, or repeated measurement falls within the analysis visit windows as described in Table 2. The windows follow the Schedule of Events in Table 1. Unscheduled/repeated measurements will be listed.

**Table 2: Analysis Visit Windows** 

| Visit Name | Visit Number | <b>Target Start Day</b> | <b>Lower Limit</b> | <b>Upper Limit</b> |
|---|---|---|---|---|
| Week 2 | 3 | 14 | 2 | 22 |
| Week 4 | 4 | 28 | 23 | 42 |





| Visit Name | Visit Number | <b>Target Start Day</b> | <b>Lower Limit</b> | <b>Upper Limit</b> |
|---|---|---|---|---|
| Week 8 | 5 | 56 | 43 | 61 |
| Week 9 | 6 | 63 | 62 | |

#### 6.1.6. Pooling of Sites

Not applicable.

#### 6.1.7. Derived Variables

- **S-IGA success** = S-IGA of "Clear" or "Almost Clear" plus a 2-grade improvement from baseline.
- **B-IGA success** = B-IGA of "Clear" or "Almost Clear" plus a 2-grade improvement from baseline.
- SI-NRS 4-point reduction = achievement of a 4-point reduction in SI-NRS pruritus score at Weeks 2, 4, and 8 compared to baseline, calculated only for subjects with an SI-NRS pruritus score of ≥ 4 at baseline.
- WI-NRS 4-point reduction = achievement of a 4-point reduction in WI-NRS pruritus score at Weeks 2, 4, and 8 compared to baseline, calculated only for subjects with a WI-NRS pruritus score of ≥ 4 at baseline.
- **PSSI** = (erythema score + induration + desquamation)  $\times$  extent of scalp affected (range 0 to 72). Erythema, induration, and desquamation are scored on a scale of 0 to 4, where 0 = absent and 4 = severest possible; extent of scale affected is scored on a scale of 0 to 6, where 0 = 0% of involved area and 6 = 90-100% of involved area.
- **PSSI-50** = achievement of a 50% reduction in PSSI from baseline
- PSSI-75 = achievement of a 75% reduction in PSSI from baseline
- **PSSI-90** = achievement of a 90% reduction in PSSI from baseline
- **PSSI-100** = achievement of a 100% reduction in PSSI from baseline
- Time to PSSI-50 (days) = date of first PSSI-50 achievement Day 1 date + 1. Subjects not achieving PSSI-50 will be censored at day of study discontinuation or date lost to follow-up, whichever is later. Due COVID-19-related site closures, some discontinuation visits occurred much later than Week 9, so time to PSSI-50 may be after Week 9.
- Time to PSSI-75 (days) = date of first PSSI-75 achievement Day 1 date + 1. Subjects not achieving PSSI-75 will be censored at day of study discontinuation or date lost to follow-up, whichever is later. Due COVID-19-related site closures, some discontinuation visits occurred much later than Week 9, so time to PSSI-75 may be after Week 9.



- Time to PSSI-90 (days) = date of first PSSI-90 achievement Day 1 date + 1. Subjects not achieving PSSI-90 will be censored at day of study discontinuation or date lost to follow-up, whichever is later. Due COVID-19-related site closures, some discontinuation visits occurred much later than Week 9, so time to PSSI-90 may be after Week 9.
- **PASI** =  $(0.1 \times [E_h + T_h + S_h] \times A_h) + (0.2 \times [E_a + T_a + S_a] \times A_a) + (0.3 \times [E_t + T_t + S_t] \times A_t) + (0.4 \times [E_l + T_l + S_l] \times A_l)$

where E, T, and S are erythema, thickness, and scaling, respectively, scored on a scale of 0 to 4, A is estimated area of skin involved, graded on a scale of 0 to 6, and h, a, t, and l are head, arms, trunk, and legs, respectively (range for total score 0 to 72). If any of the component scores are missing, the PASI cannot be calculated.

- PASI-50 = achievement of a 50% reduction in PASI from baseline
- PASI-75 = achievement of a 75% reduction in PASI from baseline
- PASI-90 = achievement of a 90% reduction in PASI from baseline
- Time to PASI-50 = date of first PASI-50 achievement Day 1 date + 1. Subjects not achieving PASI-50 will be censored at day of study discontinuation or date lost to follow-up, whichever is later. Due COVID-19-related site closures, some discontinuation visits occurred much later than Week 9, so for purposes of this calculation, the upper limit for time to PASI-50 will be capped at Day 68 (Week 9).
- **mPASI** =  $(0.1 \times [E_h + T_h + S_h] \times pA_h) + (0.2 \times [E_a + T_a + S_a] \times pA_a) + (0.3 \times [E_t + T_t + S_t] \times pA_t) + (0.4 \times [E_l + T_l + S_l] \times pA_l)$

where E, T, and S are erythema, thickness, and scaling, respectively, scored on a scale of 0 to 4, pA is estimated area of skin involved as an actual percentage (i.e., percentage in the eCRF/10) if the percent involvement is <10% OR as graded on a scale of 0 to 6, and h, a, t, and l are head, arms, trunk, and legs, respectively (range for total score 0 to 72). If any of the component scores are missing, the mPASI cannot be calculated.

- **DLQI Score** = sum of the 10 questions (individual questions scored as Very much=3, A lot=2, A little=1, Not at all=0, with Not relevant recoded to 0; Question 7: Yes=3, No=0, with Not relevant recoded to 0; range for score 0 to 30). If 1 item is missing, that item is scored as 0. If 2 or more items are missing, the score should not be calculated.
- **CDLQI Score** = sum of the 10 questions (individual questions scored as Very much=3, Quite a lot=2, Only a little=1, Not at all=0; Question 7: if the last week was school time, the question was scored as Very much=3, Quite a lot=2, Only a little=1, Not at all=0, with Prevented school recoded to 3, and if the last week was vacation, the standard responses apply; range for score 0 to 30). If 1 item is missing, that item is scored as 0. If 2 or more items are missing, the score should not be calculated.



- **PSD Total score** = sum of the 16 questions (individual questions scored 0 to 10, where higher scores indicate more severe symptoms; range for total score 0 to 160). If 1 or more items are missing, the score is not calculated.
- **Compliance** = number of applications divided by the expected number of IP applications for each subject. Compliance will be calculated using drug accountability data over the entire treatment period for each subject, up to treatment completion or discontinuation.
  - Number of expected IP applications = 56 for subjects who complete the study or number of days between first and last application of IP (last treatment date first treatment date + 1) for subjects who discontinue early from the study.
  - **Number of IP applications** = number of expected IP applications missed IP applications as collected in the electronic case report form (eCRF).
- Weight of IP (g) = returned can weight dispensed can weight.
- Body mass index (BMI)  $(kg/m^2) = [weight (kg) / height (cm) / height (cm)] \times 10,000.$
- BMI Categories
  - Underweight: BMI < 18.5
  - Normal:  $18.5 \le BMI \le 24.9$
  - Overweight:  $25.0 \le BMI \le 29.9$
  - Obese: BMI  $\geq$  30.0
- Change from baseline = value at current time point value at baseline.
- Treatment emergent AE (TEAE) = any AE with an onset date/time after the first application of IP.
- **PHQ-8** = sum of the 8 questions (individual questions scored as Not at all=0, Several days=1, More than half the days=2, and Nearly every day=3; range for score 0 to 24). If more than 1 item is missing, the score should not be calculated. If 1 item is missing, the score is calculated as (sum of answered items\*8)/number of answered items.
- **PHQ-A** = sum of the 8 questions (individual questions scored as Not at all=0, Several days=1, More than half the days=2, and Nearly every day=3, (range for score 0 to 24). If 1 item is missing, the score should not be calculated. If 1 item is missing, the score is calculated as (sum of answered items\*8)/number of answered items.
- C-SSRS Suicidal Ideation = A "yes" answer at any time during treatment to any 1 of the 5 suicidal ideation questions (Categories 1-5: Wish to be Dead, Nonspecific Active Suicidal Thoughts, Active Suicidal Ideation with Any Methods (Not Plan) without Intent





to Act, Active Suicidal Ideation with Some Intent to Act, without Specific Plan, and Active Suicidal Ideation with Specific Plan and Intent).

- C-SSRS Suicidal Behavior = A "yes" answer at any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 6-10: Preparatory Acts or Behavior, Aborted Attempt, Interrupted Attempt, Actual Attempt (nonfatal), Completed Suicide).
- C-SSRS Suicidal Ideation or Behavior = A "yes" answer at any time during treatment to any 1 of the 10 suicidal ideation and behavior questions (Categories 1-10) on the C-SSRS.
- Completion of Study = Completion of the primary efficacy assessment (S-IGA) at Week 8. This may differ than what was recorded in the eCRF.

## 6.1.8. Data Adjustments/Handling/Conventions

All collected data will be presented in Clinical Data Interchange Standards Consortium (CDISC) datasets. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the CDISC datasets.

All P values will be displayed in 4 decimals and rounded using standard scientific notation (e.g., 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as <0.0001; similarly, if a P value greater than 0.9999 occurs it will be shown in tables as >0.9999.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 23.0 thesaurus.

A treatment-related AE is any AE with a relationship to the study drug of possibly, probably, likely, or missing.

For partial AE and medication start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of first dose date and the end date (if present) is after first dose date, then impute as the month and day of the first dose date.
  - o Otherwise, assign 01 January.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the first dose date, then impute as the day of the first dose date.
  - o Otherwise, assign 01.

For partial AE and medication end dates:

- If the year is unknown, then do not impute the date but assign as missing value.
- If the year is known, but the month or month and day is unknown, then:



- o If the year matches the year of the last date of the study (date of last contact if subject lost to follow-up; date of completion or early termination otherwise), then impute as the month and day of the last date of the study.
- o Otherwise, assign 31 December.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the last date of the study, then impute as the day of the last date of the study.
  - Otherwise, assign the last day of the month.

These conventions will be applied to AE and medication onset dates and times with the following precaution: if the missing date and time reflect the date and time of onset of an AE, the modified date and time will be constructed to match the first documented date/time post drug administration while preserving the order in which the AE was reported in the eCRF.

In cases where variables for questionnaires were derived in the eCRF (e.g., total scores) and a derivation is indicated in Section 6.1.7, the results as derived by statistics (as opposed to the results derived in the eCRF) will be used in analysis.

## 6.2. Special Handling for COVID-19 Disruptions

In some cases, study visits will have to be delayed/not performed as a result of COVID-19 disruptions (e.g., sites were closed or subjects were under stay-at-home orders). Where possible, study sites may collect post-baseline data from subjects remotely by telephone, traditional mail, and/or email; this will be clearly documented in the source. If possible, sites should adhere to the protocol visit window for remote data collection.

Investigator assessments and subject questionnaires normally completed directly in the electronic patient reported outcomes (ePRO) tablet during on-site visits should be completed on the appropriate paper source documents. The following assessments/questionnaires are approved to be collected via telemedicine/remotely:

- WI-NRS/SI-NRS
- DLQI/CDLQI
- C-SSRS
- PHQ-8/PHQ-A
- Subject Local Tolerability
- PSD

The following assessments cannot be completed via telemedicine/remotely:

- S-IGA/B-IGA
- BSA
- Investigator Local Tolerability
- PASI/mPASI
- PSSI
- Subject Weight





Study visits and procedures must be followed per protocol whenever possible. Any specific changes in study conduct that deviate from the protocol should be communicated to the institutional review board and Sponsor. All protocol deviations which occurred as a result of COVID-19 disruptions (e.g., visits out of window, missed assessments, etc.) will be differentiated from other protocol deviations.

Subjects who were affected by COVID-19 disruptions by either missing their Week 8 visit or being discontinued before having a Week 8 visit due to COVID-19 related disruptions will be excluded from the mITT population, as described in Section 5.

#### 7. Study Subjects and Demographics

#### 7.1. Disposition of Subjects and Withdrawals

Disposition will include tabulations of the number of subjects randomized into each treatment group, the number of subjects who received treatment, subjects completing study, tabulated reasons for discontinuation from the study, including whether or not the subject did not complete the study due to COVID-19 disruption and reasons, and number of subjects in each analysis population. Disposition will be summarized for all subjects who were entered into database by treatment group and overall.

#### 7.2. Protocol Deviations

The number of subjects with major protocol deviations and/or eligibility deviations will be summarized in categories by treatment group and overall for subjects in Safety population.

#### 7.3. Demographics and Other Baseline Characteristics

Summary statistics for age, age category (12-17, ≥18), gender (including child-bearing potential), race, ethnicity, height, weight, percent BSA, BMI, and baseline disease characteristics (S-IGA, B-IGA, PSSI, SI-NRS, PSD total score, PASI, mPASI, WI-NRS, DLQI, and CDLQI) will be presented by treatment group and overall.

A summary of treatment history, including history of response, intolerance, or contraindication to topical corticosteroids and/or topical vitamin D derivatives, and psoriasis involvement on knees and/or elbows and genitalia will be provided.

For the continuous variables, the number of nonmissing values and the mean, SD, minimum, median and maximum will be tabulated.

For ordinal variables such as the S-IGA, B-IGA, SI-NRS, and WI-NRS, summary statistics including the mean, median, and range of the ordinal variable will be presented, as well as frequency counts of each level of the ordinal variable.

For the categorical variables, the counts and proportions of each value will be tabulated.

These analyses will be conducted for the ITT, mITT, and Safety populations, except for treatment history summary, which will only be summarized on the Safety population.



#### 7.4. Exposure and Compliance

The number of IP applications by each subject based on diary data will be summarized using descriptive statistics appropriate for continuous variables.

The amount of IP each subject used based on can weight will be summarized descriptively by treatment group using continuous methods.

A subject will be considered compliant with the dosing regimen if the subject applies at least 80% of the expected applications during the IP application period and does not miss more than 3 consecutive doses.

Investigational product application compliance will be calculated based on number of applications divided by the expected number of IP applications. Compliance will be summarized descriptively by treatment group using the following categories:

#### 8. Efficacy Analysis

The order of testing for the primary and secondary endpoints is discussed in Section 6.1.3. Exploratory endpoints are not included in the testing strategy.

## 8.1. Primary Efficacy Analysis

#### 8.1.1. Scalp Investigator Global Assessment (S-IGA)

The S-IGA is an ordinal scale with 5 severity grades which is reported only in integers. Table 3 illustrates the description of each severity grade.

Table 3: S-IGA

| Score | Grade | Description |
|---|---|---|
| 0 | Clear | Plaque thickening = no elevation or thickening over normal skin |
| | | Scaling = no evidence of scaling |
| | | Erythema = none (no residual red coloration but post-inflammatory |
| | | hyperpigmentation may be present) |
| 1 | Almost | Plaque thickening = none or possible thickening but difficult to ascertain |
| | Clear | if there is a slight elevation above normal skin level |
| | | Scaling = none or residual surface drying and scaling |
| | | Erythema = light pink coloration |
| 2 | Mild | Plaque thickening = slight but definite elevation |
| | | Scaling = fine scales partially or mostly covering the lesions |
| | | Erythema = light red coloration |





| Score | Grade | Description |
|---|---|---|
| 3 | Moderate | Plaque thickening = moderate elevation with rounded or sloped edges |
| | | Scaling = most lesions at least partially covered |
| | | Erythema = definite red coloration |
| 4 | Severe | Plaque thickening = marked or very marked elevation typically with |
| | | hard or sharp edges |
| | | Scaling = non-tenacious or thick tenacious scale, covering most or all of |
| | | lesions |
| | | Erythema = very bright red coloration; extreme red coloration; deep red |
| | | coloration |

For this study, the primary estimand is the odds of achieving S-IGA success at 8 weeks; that is, the ratio of the odds of achieving S-IGA success at 8 weeks roflumilast foam 0.3% relative to the odds of success at 8 weeks of using a matching vehicle cream. In the course of the 8-week randomized treatment period, subjects may be exposed to possible known or unknown intercurrent events that could possibly impact the estimand, such as treatment discontinuation due to a specific adverse effect or perhaps a lack of effect. The "Treatment Policy Strategy" has been adopted for handling all known or unknown intercurrent events in this study. To this end, the ITT principle will serve as the analytical basis for interpreting the estimand. In other words, the odds ratio of achieving S-IGA success for roflumilast foam 0.3% relative to vehicle at 8 weeks will be evaluated regardless of the occurrence of any such intercurrent event. This estimand shall be estimated using the CMH approach. This approach produces an estimate that is the combined odds ratio resulting from adjusting for the possible effects of 3 classification factors: country, baseline S-IGA category (2 vs.  $\geq$ 3) and baseline B-IGA category (2 vs.  $\geq$ 3).

## Categorical Data Analysis

The primary efficacy endpoint is success in S-IGA of disease severity, defined as an S-IGA of "Clear" or "Almost Clear" plus a 2-grade improvement from baseline at Week 8.

The primary endpoint will be analyzed using a CMH test stratified by country, baseline S-IGA category, and baseline B-IGA category. Statistical significance will be concluded at the 5% significance level (2-sided) or less, as discussed in Section 6.1.3. Odds ratios and 95% CIs for the odds ratios will be provided. Additionally, the 95% Wilson CIs for proportion of successes in each treatment group will be presented.

For the primary analysis, missing S-IGA scores will be imputed using multiple imputation as described in Section 6.1.4.1. These imputations will result in a minimum of 25 to a maximum of 250 complete analysis datasets, depending on the number of imputed monotone datasets required. The CMH analyses will be performed separately for each of the complete analysis data sets, and the results will be combined into one multiple imputation inference (estimated treatment effect and associated CI and *P* value). As a sensitivity analysis, the above described CMH test will be performed on the nonimputed data.

Sensitivity analyses of the primary endpoint will also be performed using the original (nonimputed) dataset. These will include a repeated measures logistic regression model (GEE) with S-IGA success as the dependent variable and treatment, country, visit, and baseline S-IGA score as the independent variables.





Achievement of a score of clear will also be analyzed using the CMH test, on nonimputed data.

A tipping point analysis will be performed as described in Section 6.1.4.2. For the tipping point analysis, a figure will be provided that displays the P values in the analysis plotted against the range of shift parameters; included in this figure will be the shift parameters and P values for the range of shift parameters to provide information on where the analysis tips from significant to non-significant.

## Subgroup Analyses – Observed Data

For the primary endpoint of IGA success (S-IGA of "Clear" or "Almost Clear" plus a 2-grade improvement from baseline at Week 8), the CMH analysis will be performed on the following subgroups, using observed data:

- Topical Corticosteroids Naïve Subjects
- Topical Vitamin D Derivatives Naïve Subjects
- Psoriasis involvement on the knee and/or elbow
- Subjects who achieved both S-IGA and B-IGA success at Week 8
- By Study Site

#### <u>Subgroup Analyses – Multiple Imputation Data</u>

For the primary endpoint of IGA success (S-IGA of "Clear" or "Almost Clear" plus a 2-grade improvement from baseline at Week 8), the CMH analysis will be performed on the following subgroups, using multiple imputation data:

- Baseline S-IGA = 3
- Baseline S-IGA = 4
- Age Category = 12-17 years
- Age Category =  $\ge 18$  years
- Subjects who achieved both S-IGA and B-IGA success at Week 8

#### Continuous Data Analysis

Analysis of change from baseline in S-IGA scores at Weeks 2, 4, 8, and 9 will be performed using descriptive summaries (mean, median, inter-quartile range) by treatment group and study visit. These descriptive statistics will also be presented based on the multiple imputation data.

#### All Analyses

All other missing data for all other analyses and summaries will remain missing and will not be imputed. All weeks will be included in these analyses, although only Week 8 using the ITT population will be included in the testing strategy.

The primary efficacy analysis will be based on ITT population, and all of the above analyses will be repeated for the mITT population.

#### 8.2. Secondary Efficacy Analysis

All secondary efficacy analyses will be performed using the ITT and mITT populations, unless otherwise specified.





## 8.2.1. Body Investigator Global Assessment (B-IGA)

The scale, grade, and description for the B-IGA is identical to the S-IGA, as discussed in Section 8.1.

Achievement of a B-IGA score of "clear" or "almost clear" PLUS a 2-grade improvement from baseline at Weeks 2, 4, 8, and 9 will be analyzed similar to the primary efficacy endpoint using CMH test stratified by country, baseline S-IGA category, and baseline B-IGA category, with the exception that missing data will not be replaced (i.e., observed data). Odds ratios and 95% CIs of the odds ratios will be provided. Additionally, the 95% Wilson CIs for proportion of successes in each treatment group will be presented. In addition, the number and percentage of subjects in each category will be summarized by treatment and visit. Only the Week 8 results using the ITT population will be included in the testing strategy.

Analysis of change from baseline in B-IGA scores at Weeks 2, 4, 8, and 9 will be performed using descriptive summaries (mean, median, inter-quartile range) by treatment group and study visit.

#### 8.2.2. Psoriasis Scalp Severity Index (PSSI)

The PSSI is used to measure the severity of psoriasis, combining the assessment of the severity of scalp lesions and the area of scalp affected into a single score ranging from 0 (no disease) to 72 (maximal disease). The PSSI score will be analyzed as follows:

- Change and percent change from baseline to Weeks 2, 4, 8, and 9 in the PSSI will be analyzed using descriptive summaries and an analysis of covariance (ANCOVA) with terms for country, baseline S-IGA category, and baseline B-IGA category, and baseline PSSI score as a covariate. Statistical comparisons between the treatment groups will be obtained using contrasts. The least-squares (LS) means, standard errors, 95% CIs, and P values will be presented.
- Frequencies and percentages of subjects achieving PSSI-50, PSSI-75, PSSI-90, and PSSI-100 will be presented by study week and treatment group. Additionally, these endpoints will be analyzed similar to the primary efficacy endpoint using a CMH test stratified by country, baseline S-IGA category, and baseline B-IGA category, on observed data. Only the PSSI-75 and PSSI-90 at Week 8 using the ITT population will be included in the testing strategy. Odds ratios and 95% CIs of the odds ratios will be provided. Additionally, the 95% Wilson CIs for proportion of successes in each treatment group will be presented.
- Time to achieving PSSI-50, PSSI-75, and PSSI-90 will be summarized using Kaplan-Meier methods and the difference between treatment groups evaluated using the log-rank statistic, and 95% CIs of the median for each treatment group will be presented. In addition, a Cox proportional hazards model that includes the stratification factors will be run and the hazard ratio and associated 95% Wald CIs will be presented. Time to achieving PSSI-50 using the ITT population will also be included in the testing strategy. Time to achieving PSSI-75 or PSSI-90 using the ITT population will not be included in the testing strategy, but will be considered as a supportive analysis.





#### 8.2.3. Scalp Itch – Numeric Rating Scale (SI-NRS)

The SI-NRS scale ranges from 0 to 10 with 0 being "no scalp itch" and 10 equaling "worst scalp itch imaginable." This will be determined by asking the subject's assessment of worst scalp itch over the past 24 hours. The SI-NRS will be analyzed as follows:

- Change and percent change from baseline to Weeks 2, 4, and 8 in SI-NRS will be analyzed using descriptive summaries and an ANCOVA with terms for country, baseline S-IGA category, and baseline B-IGA category, and baseline SI-NRS score as a covariate. Statistical comparisons between the treatment groups will be obtained using contrasts. The LS means, standard errors, 95% CIs, and *P* values will be presented.
- In subjects with a baseline SI-NRS score ≥4, achievement of a ≥4-point improvement from baseline in SI-NRS score at Weeks 2, 4, and 8 will be analyzed using CMH tests stratified by country, baseline S-IGA category, and baseline B-IGA similar to the primary analysis above, with the exception that missing data will not be replaced. Odds ratios and 95% CIs of the odds ratios will be provided. Additionally, the 95% Wilson CIs for proportion of successes in each treatment group will be presented. This will be summarized using SPRU-ITT and SPRU-mITT populations.

## 8.2.4. Psoriasis Symptoms Diary (PSD)

The PSD assesses the severity of symptoms or how bothersome are the symptoms of psoriasis. The PSD will be analyzed as follows:

• Change and percent change from baseline to Weeks 2, 4, and 8 in the PSD individual item and total scores will be analyzed using descriptive statistics and an ANCOVA (total score only) with terms for country, baseline S-IGA category, and baseline B-IGA category, and baseline PSD score as a covariate. Statistical comparisons between the treatment groups will be obtained using contrasts. The LS means, standard errors, 95% CIs, and *P* values will be presented. Only change from baseline in PSD total score at Weeks 4 and 8 using the ITT population will be included in the testing strategy.

#### 8.3. Exploratory Efficacy Analysis

Exploratory efficacy analysis will be performed for subjects belonging to ITT and mITT populations.

The exploratory endpoints include:

- Achievement of success in PASI-90, PASI-75, and PASI-50 at Weeks 2, 4, 8, and 9
- Time to success in PASI-50
- Change and percent change from baseline in PASI/mPASI at Weeks 2, 4, 8, and 9
- Change and percent change from baseline in WI-NRS at Weeks 2, 4, and 8
- For subjects with baseline WI-NRS score ≥4, achievement of ≥4-point improvement from baseline in WI-NRS at Weeks 2, 4, and 8 (summarized on the PRU4-ITT and PRU4-mITT populations)





- Change and percent change from baseline in DLQI/CDLQI total scores at Weeks 2, 4, and 8
- Change and percent change from baseline in % BSA affected by disease at Weeks 2, 4, 8, and 9

Time to success in PASI-50 and change and percent change from baseline for all relevant exploratory endpoints will be summarized descriptively; additionally, all endpoints will be analyzed using an ANCOVA with terms for country, baseline S-IGA category, and baseline B-IGA category, and baseline assessment score as a covariate. Statistical comparisons between the treatment groups will be obtained using contrasts. The LS means, standard errors, 95% CIs, and *P* values will be presented. Achievement of success in PASI-50, PASI-75, and PASI-90; achievement of success in mPASI-50, mPASI-75, and mPASI-90; and improvement in WI-NRS will be presented using proportions. Odds ratios and 95% CIs of the odds ratios will be provided. Additionally, the 95% Wilson CIs for proportion of successes in each treatment group will be presented.

For efficacy analysis purposes, the data that is collected by the ePRO will be used for % BSA affected by disease summarization.

## 9. Safety and Tolerability Analysis

Safety will be evaluated from reported AEs, physical examinations, local tolerability assessments, changes in clinical laboratory values, changes in vital signs/weight, C-SSRS, PHQ-8, and modified PHQ-A results. No inferential statistical tests will be performed.

All safety analyses will be performed on the Safety population.

#### 9.1. Adverse Events

All AEs, TEAEs, and SAEs will be coded using the MedDRA dictionary version 23.0.

A TEAE is defined as an AE that started post application of IP at the Baseline visit through study completion. An overall summary of TEAEs will be provided; this will present number and percent of subjects who reported at least 1 of the following: TEAE (including all TEAEs, TEAEs by maximum severity, and TEAEs by greatest relationship), SAE, discontinued the study due to a TEAE, or a TEAE resulting in death.

The number and percent of subjects reporting TEAEs, grouped by MedDRA system organ class (SOC) and preferred term, will be tabulated by severity or greatest relationship to study IP and treatment group. In the case of multiple occurrences of the same TEAE within the same subject, each subject will only be counted once for each preferred term. Additionally, the number and percent of subjects reporting related TEAEs will be summarized by MedDRA preferred term and treatment group.

In the summaries showing severity and relationship to study medication the event with the maximum severity (mild < moderate < severe) or strongest relationship (not related < related) will be reported. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = likely).





In the AE data listings, all AEs will be displayed. Any AEs that are treatment emergent will be flagged.

#### 9.1.1. Adverse Events Leading to Withdrawal

A summary of incidence rates (frequencies and percentages) of TEAEs leading to withdrawal of study drug by treatment group, SOC, and preferred term will be prepared for the Safety population. Additionally, this table will be repeated for TEAEs leading to withdrawal from the study. No inferential statistical tests will be performed.

A data listing of AEs leading to withdrawal of study drug will also be provided, displaying details of the event(s) captured on the eCRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study will be listed.

Serious adverse events (SAEs) will be listed and tabulated by SOC and preferred term and presented by treatment group, severity, and relationship to study treatment.

#### 9.2. Local Tolerability Assessments

The investigator's assessment of the application site reaction will be summarized by study visit using both categorical methods (number and percentage of subjects with each score) as well as continuous methods (e.g., mean, median). Categorical summaries will be provided for dermal response as well as other effects. No inferential statistical tests will be performed.

The subject's assessment of the application site reaction will be summarized similarly.

## 9.3. Clinical Laboratory Evaluations

Laboratory test results will be summarized descriptively by treatment and study visit as both observed values and change from baseline values for continuous hematology, chemistry, and urinalysis results. Categorical urinalysis results will be summarized using frequencies by study visit and treatment.

The number of subjects with clinical laboratory values below, within, or above the normal range by study visit and in relation to baseline will be tabulated for each clinical laboratory analyte by treatment group (shift table).

Abnormal results will be flagged in the listings. In addition, pregnancy test results and hormonal laboratory results will be listed.

#### 9.4. Vital Signs

Descriptive summaries of observed values and changes from baseline will be calculated for systolic blood pressure, diastolic blood pressure, heart rate, height, weight, BMI, and oral body temperature by treatment group and visit.





The number of subjects who gain or lose  $\geq 5\%$  of their baseline body weight during the course of the study, as well as subjects who gain or lose  $\geq 10\%$  of their baseline body weight over the course of the study, will be summarized by treatment group. This summary will be repeated by intentionality of weight loss (intentional or unintentional, as captured on the eCRF).

Shift tables for subjects who shift from their baseline BMI category as defined in Section 6.1.7 (underweight, normal, overweight, obese) to a different BMI category throughout the course of the study will be provided by treatment group and visit. This summary will be repeated by intentionality of weight loss (intentional or unintentional, as captured on the eCRF).

## 9.5. PHQ-8 and Modified PHQ-A

Data for PHQ-8 and modified PHQ-A will be classified using each subject's total score at a time point into a category based on the following scoring system:

- None Minimal depression (0 to 4)
- Mild depression (5 to 9)
- Moderate depression (10 to 14)
- Moderately severe depression (15 to 19)
- Severe depression (20 to 24)

Shift tables showing the category of severity at each visit by treatment group will be presented.

#### 9.6. **C-SSRS**

The C-SSRS is a questionnaire that prospectively assesses Suicidal Ideation and Suicidal Behavior. At the Screening study visit, "Baseline/Screening" version of the C-SSRS will be used. This version assesses Suicidal Ideation and Suicidal Behavior during the subject's lifetime and during the past 6 months. For the Screening visit, "lifetime" experience of the subject with Suicidal Ideation and Suicidal Behavior will be summarized. From Baseline visit, the "Since Last Visit" version will be used.

Suicidality data collected on the C-SSRS will be listed for all subjects. Tables will include results from the Suicidal Ideation and Suicidal Behavior sections of the C-SSRS. Frequencies and percentages of subjects with a response of "Yes" at any point on the Suicidal Ideation and Suicidal Behavior items will be summarized by study visit and treatment group.

#### 9.7. Physical Examination

The number and percentage of subjects with normal and abnormal findings in the physical examination will be displayed at each study visit and treatment group.

#### 9.8. Concomitant Medication

Prior and concomitant medications will be summarized descriptively by treatment, Anatomical Therapeutic Chemical (ATC) Class Level 4, and Preferred Term using counts and percentages.





Prior medications will be presented separately from concomitant medications. Medications that started before the first application of IP will be considered prior medications whether or not they were stopped prior to the first application of study drug. Any medications continuing or starting after the first application of study drug will be considered to be concomitant. If a medication starts before the first application of study drug and continues after the first application of study drug it will be considered both prior and concomitant.

Medications will be coded using World Health Organization (WHO) Drug Global B3, version September 2019.

#### 10. Changes from Planned Analysis

The following analysis populations have been added:

- The mITT population has been added to handle situations where a subject was unable to attend the Week 8 visit or discontinued from the study before the Week 8 visit due to COVID-19 disruptions;
- The SPRU4-ITT and SPRU4-mITT populations have been added to facilitate SI-NRS analysis on the ITT and mITT populations, respectively; and
- The PRU4-ITT and PRU4-mITT populations have been added to facilitate WI-NRS analysis on the ITT and mITT populations, respectively.

These populations are not included in the protocol.

The PP population and associated analyses have been removed at the request of the Sponsor, as they were considered to be uninformative.

Additional exploratory endpoints have been added in the SAP which are not specified in the protocol. They are:

- Change and percent change from baseline in SI-NRS at Weeks 2, 4, and 8
- Change and percent change from baseline in PASI at Weeks 2, 4, 8, and 9
- Change and percent change from baseline in WI-NRS at Weeks 2, 4, and 8

Additionally, odds ratios and 95% CIs of odds ratios for comparisons between treatment groups, and 95% Wilson CIs for proportion of successes in each treatment group for binary outcomes will be provided.

Additional efficacy analyses have been added in the SAP which are not specified in the protocol, as requested by the Sponsor. They are:

- Analysis of S-IGA success based on the following subgroups (both ITT and mITT populations, observed data only):
  - o Topical corticosteroids naïve subjects
  - o Topical vitamin D derivatives naïve subjects
  - Subjects with psoriasis involvement on the knee and/or elbow
  - Subjects who achieved S-IGA and B-IGA success at Week 8
  - o By study site
- Analysis of S-IGA score of clear (included in the fixed-sequence testing strategy)
- Analysis of S-IGA success based on the following subgroups (both ITT and mITT)





populations, multiple imputation data only):

- $\circ$  Baseline S-IGA = 3
- $\circ$  Baseline S-IGA = 4
- o Age Category: 12-17 years
- o Age Category: ≥18 years
- o Subjects who achieved S-IGA and B-IGA success at Week 8
- Achievement of success in PSSI-100
- Time to achievement of PSSI-75 and PSSI-90
- Achievement of success in mPASI-50, mPASI-75, and mPASI-90

Additional safety analyses have been added in the SAP which are not specified in the protocol, as requested by the Sponsor. They are:

- Incidence of TEAEs leading to study discontinuation by SOC and preferred term
- Incidence of related TEAEs by preferred term
- Summarization of weight loss categories by intentionality of weight lose
- Shift tables for BMI categories

#### 11. Other Planned Analysis

## 11.1. Pharmacokinetic Analysis

All PK collection information from the eCRF will be presented in a listing. Concentration data and PK parameters will be summarized by timepoint (concentrations data) and treatment group using summary statistics. In addition, PK concentration and parameter listings will be presented.

#### 12. References

- 1. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 2. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 4. Ratitch, B., Lipkovich, I., & O'Kelly, M. (2013). Combining Analysis Results from Multiply Imputed Categorical Data.
  - PharmaSUG. <a href="https://www.pharmasug.org/proceedings/2013/SP/PharmaSUG-2013-SP03.pdf">https://www.pharmasug.org/proceedings/2013/SP/PharmaSUG-2013-SP03.pdf</a>



## 13. Tables, Listings, and Figures

All TLFs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (e.g., listing number).

## 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number ARQ-154-204. The table numbers and page numbers are place holders only and will be determined when the tables are produced.

## 13.1.1. Demographic Data

**Table 4: Demographic Data Summary Tables** 

| Number | Population | Title |
|---|---|---|
| Table 14.1.1 | All<br>Randomized | Summary of Subject Disposition |
| Table 14.1.2.1 | Safety | Summary of Demographics and Baseline Characteristics |
| Table 14.1.2.2 | ITT | Summary of Demographics and Baseline Characteristics |
| Table 14.1.2.3 | mITT | Summary of Demographics and Baseline Characteristics |
| Table 14.1.3 | Safety | Previous Treatment History of Scalp and Body Psoriasis |
| Table 14.1.4 | Safety | Summary of Protocol Deviations |
| Table 14.1.5 | Safety | Summary of Prior Medications by ATC Class Level 4 and Preferred Term |
| Table 14.1.6 | Safety | Summary of Study Drug Exposure and Compliance |

## 13.1.2. Efficacy Data

**Table 5: Efficacy Data Summary Tables** 

| Number | Population | Title |
|---|---|---|
| Table 14.2.1.1 | ITT | Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit – Observed Data |
| Table 14.2.1.2 | mITT | Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit – Observed Data |
| Table 14.2.1.3 | ITT | Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit – Multiple Imputation |
| Table 14.2.1.4 | mITT | Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit – Multiple Imputation |



| Number | Population | Title |
|---|---|---|
| Table 14.2.1.5.1 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results |
| Table 14.2.1.5.2 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Topical Corticosteroids – Naïve Subjects |
| Table 14.2.1.5.3 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Topical Vitamin D Derivatives – Naïve Subjects |
| Table 14.2.1.5.4 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Subjects with Psoriasis Involvement on the Knee and/or Elbow |
| Table 14.2.1.5.5 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Subjects who Achieved S-IGA and B-IGA Success at Week 8 |
| Table 14.2.1.5.6 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit and Study Site – Observed Data Categorical Results |
| Table 14.2.1.6.1 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results |
| Table 14.2.1.6.2 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Topical Corticosteroids – Naïve Subjects |
| Table 14.2.1.6.3 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Topical Vitamin D Derivatives – Naïve Subjects |
| Table 14.2.1.6.4 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Subjects with Psoriasis Involvement on the Knee and/or Elbow |



| Number | Population | Title |
|---|---|---|
| Table 14.2.1.6.5 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results Subjects who Achieved S-IGA and B-IGA Success at Week 8 |
| Table 14.2.1.6.6 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit and Study Site – Observed Data Categorical Results |
| Table 14.2.1.7.1 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results |
| Table 14.2.1.7.2 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Baseline S-IGA = 3 |
| Table 14.2.1.7.3 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Baseline S-IGA = 4 |
| Table 14.2.1.7.4 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Age Category = 12-17 Years |
| Table 14.2.1.7.5 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Age Category = ≥18 Years |
| Table 14.2.1.7.6 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Subjects who Achieved S-IGA and B-IGA Success at Week 8 |
| Table 14.2.1.8.1 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results |
| Table 14.2.1.8.2 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Baseline S-IGA = 3 |


| Number | Population | Title |
|---|---|---|
| Table 14.2.1.8.3 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Baseline S-IGA = 4 |
| Table 14.2.1.8.4 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Age Category = 12-17 Years |
| Table 14.2.1.8.5 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Age Category = ≥18 Years |
| Table 14.2.1.8.6 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results Subjects who Achieved S-IGA and B-IGA Success at Week 8 |
| Table 14.2.1.9 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Tabulation of Fitted Point Estimates from Generalized Estimating Equations for Binary Response |
| Table 14.2.1.10 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Tabulation of Fitted Point Estimates from Generalized Estimating Equations for Binary Response |
| Table 14.2.1.11 | ITT | Summary of Scalp Investigator Global Assessment (S-IGA) – Score of Clear – Observed Data |
| Table 14.2.1.12 | mITT | Summary of Scalp Investigator Global Assessment (S-IGA) – Score of Clear – Observed Data |
| Figure 14.2.1.11 | ITT | Plot of Scalp Investigator Global Assessment (S-IGA) Tipping Point Analysis P Values vs Shift Parameters |
| Figure 14.2.1.12 | mITT | Plot of Scalp Investigator Global Assessment (S-IGA) Tipping Point Analysis P Values vs Shift Parameters |
| Table 14.2.2.1 | ITT | Summary and Change from Baseline in Body Investigator Global Assessment (B-IGA) Grades by Study Visit |
| Table 14.2.2.2 | mITT | Summary and Change from Baseline in Body Investigator Global Assessment (B-IGA) Grades by Study Visit |
| Table 14.2.2.3 | ITT | Summary of Body Investigator Global Assessment (B-IGA) Grades and Success by Study Visit Categorical Results |



| Number | Population | Title |
|---|---|---|
| Table 14.2.2.4 | mITT | Summary of Body Investigator Global Assessment (B-IGA) Grades and Success by Study Visit |
| | | Categorical Results |
| Table 14.2.3.1 | ITT | Summary and Change from Baseline in PSSI Scores by Study Visit |
| Table 14.2.3.2 | mITT | Summary and Change from Baseline in PSSI Scores by Study Visit |
| Table 14.2.3.3 | ITT | Summary of Achievement of PSSI-50, PSSI-75, PSSI-90, and PSSI-100 by Study Visit |
| Table 14.2.3.4 | mITT | Summary of Achievement of PSSI-50, PSSI-75, PSSI-90, and PSSI-100 by Study Visit |
| Table 14.2.3.5 | ITT | Time to Achievement of PSSI-50, PSSI-75, and PSSI-90 |
| Table 14.2.3.6 | mITT | Time to Achievement of PSSI-50, PSSI-75, and PSSI-90 |
| Table 14.2.3.7 | ITT | Summary of PSSI Scores by Study Visit – ANCOVA |
| Table 14.2.3.8 | mITT | Summary of PSSI Scores by Study Visit – ANCOVA |
| Table 14.2.4.1 | ITT | Summary and Change from Baseline in Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit |
| Table 14.2.4.2 | mITT | Summary and Change from Baseline in Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit |
| Table 14.2.4.3 | SPRU4-ITT | Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score Success by Study<br>Visit |
| Table 14.2.4.4 | SPRU4-mITT | Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score Success by Study<br>Visit |
| Table 14.2.4.5 | ITT | Summary of Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit – ANCOVA |
| Table 14.2.4.6 | mITT | Summary of Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit – ANCOVA |
| Table 14.2.5.1 | ITT | Summary and Change from Baseline in Psoriasis Symptom Diary (PSD) Total and Individual Item Scores by Study Visit |
| Table 14.2.5.2 | mITT | Summary and Change from Baseline in Psoriasis Symptom Diary (PSD) Total and Individual Item Scores by Study Visit |
| Table 14.2.5.3 | ITT | Summary of Psoriasis Symptom Diary (PSD) Total Scores by Study Visit – ANCOVA |
| Table 14.2.5.4 | mITT | Summary of Psoriasis Symptom Diary (PSD) Total Scores by Study Visit – ANCOVA |
| Table 14.2.6.1 | ITT | Summary and Change from Baseline in PASI/mPASI by Study Visit |
| Table 14.2.6.2 | mITT | Summary and Change from Baseline in PASI/mPASI by Study Visit |
| Table 14.2.6.3 | ITT | Summary of PASI/mPASI by Study Visit – ANCOVA |
| Table 14.2.6.4 | mITT | Summary of PASI/mPASI by Study Visit – ANCOVA |
| 1 | • | 1 |



| Number | Population | Title |
|---|---|---|
| Table 14.2.6.5 | ITT | Summary of Achievement of PASI-50, PASI-75, and PASI-90 by Study Visit |
| Table 14.2.6.6 | mITT | Summary of Achievement of PASI-50, PASI-75, and PASI-90 by Study Visit |
| Table 14.2.6.7 | ITT | Time to Achievement of PASI-50 |
| Table 14.2.6.8 | mITT | Time to Achievement of PASI-50 |
| Table 14.2.6.9 | ITT | Summary of Achievement of mPASI-50, mPASI-75, and mPASI-90 by Study Visit |
| Table 14.2.6.10 | mITT | Summary of Achievement of mPASI-50, mPASI-75, and mPASI-90 by Study Visit |
| Table 14.2.7.1 | ITT | Summary and Change from Baseline in Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit |
| Table 14.2.7.2 | mITT | Summary and Change from Baseline in Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit |
| Table 14.2.7.3 | ITT | Summary of Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit – ANCOVA |
| Table 14.2.7.4 | mITT | Summary of Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit – ANCOVA |
| Table 14.2.7.5 | PRU4-ITT | Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit |
| Table 14.2.7.6 | PRU4-mITT | Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit |
| Table 14.2.8.1 | ITT | Summary and Change from Baseline in Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit |
| Table 14.2.8.2 | mITT | Summary and Change from Baseline in Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit |
| Table 14.2.8.3 | ITT | Summary of Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit – ANCOVA |
| Table 14.2.8.4 | mITT | Summary of Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit – ANCOVA |
| Table 14.2.9.1 | ITT | Summary and Change from Baseline in % Body Surface Area (BSA) Affected by Disease by Study Visit |
| Table 14.2.9.2 | mITT | Summary and Change from Baseline in % Body Surface Area (BSA) Affected by Disease by Study Visit |
| Table 14.2.9.3 | ITT | Summary of % Body Surface Area (BSA) Affected by Disease by Study Visit – ANCOVA |
| Table 14.2.9.4 | mITT | Summary of % Body Surface Area (BSA) Affected by Disease by Study Visit – ANCOVA |



## 13.1.3. Safety Data

# **Table 6: Safety Data Summary Tables**

| Number | Population | Title |
|---|---|---|
| 14.3.1 Displays | of Adverse I | Events |
| Table 14.3.1.1 | Safety | Summary of Treatment Emergent Adverse Events |
| Table 14.3.1.2 | Safety | Incidence of Treatment Emergent Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.1.3 | Safety | Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity |
| Table 14.3.1.4 | Safety | Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug |
| Table 14.3.1.5 | Safety | Incidence of Treatment Emergent Adverse Events Leading to Study Drug<br>Discontinuation by System Organ Class and Preferred Term |
| Table 14.3.1.6 | Safety | Incidence of Treatment Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term |
| Table 14.3.1.7 | Safety | Incidence of Related Treatment Emergent Adverse Events by Preferred Term |
| 14.3.2 Summar | ry of Deaths, | Other Serious and Significant Adverse Events |
| Table 14.3.2.1 | Safety | Incidence of Serious Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.2.2 | Safety | Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug |
| Table 14.3.2.3 | Safety | Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Maximum Severity |
| 14.3.3 Narrativ | ves of Deaths, | Other Serious and Certain Other Significant Adverse Events |
| Table 14.3.3.1 | Safety | Listing of Adverse Events Leading to Study Drug Discontinuation |
| Table 14.3.3.2 | Safety | Listing of Serious Adverse Events |
| Table 14.3.3.3 | Safety | Listing of Deaths |
| 14.3.4 Abnorm | al Laborator | y Value |
| NA | | |
| 14.3.5 Laborat | ory Data Sun | nmary Tables |
| Table 14.3.5.1.1 | Safety | Summary of Serum Chemistry Laboratory Results by Study Visit |
| Table 14.3.5.1.2 | Safety | Shift from Baseline in Clinical Chemistry Laboratory Results by Study Visit |
| Table 14.3.5.2.1 | Safety | Summary of Hematology Laboratory Results by Study Visit |
| Table 14.3.5.2.2 | Safety | Shift from Baseline in Hematology Laboratory Results by Study Visit |



| Number | Population | Title |
|---|---|---|
| Table 14.3.5.3.1 | Safety | Summary of Quantitative Urinalysis Laboratory Results by Study Visit |
| Table 14.3.5.3.2 | Safety | Shift from Baseline in Quantitative and Qualitative Urinalysis Laboratory Results by Study Visit |
| Table 14.3.5.3.3 | Safety | Summary of Qualitative Urinalysis Laboratory Results by Study Visit |
| 14.3.6 Other Sa | afety Data Su | ımmary Tables |
| Table 14.3.6.1 | Safety | Shift from Baseline in Patient Health Questionnaire (PHQ-8)/Modified PHQ-Adolescents by Study Visit |
| Table 14.3.6.2.1 | Safety | Summary of Investigator Local Tolerability Assessment by Study Visit |
| Table 14.3.6.2.2 | Safety | Summary of Investigator Local Tolerability Assessment (Dermal Response) by Study Visit Categorical Results |
| Table 14.3.6.2.3 | Safety | Summary of Investigator Local Tolerability Assessment (Other Effects) by Study Visit Categorical Results |
| Table 14.3.6.3.1 | Safety | Summary of Subject Local Tolerability Assessment by Study Visit |
| Table 14.3.6.3.2 | Safety | Summary of Subject Local Tolerability Assessment by Study Visit Categorical Results |
| Table 14.3.6.4.1 | Safety | Summary of Vital Signs by Study Visit |
| Table 14.3.6.4.2 | Safety | Shift from Baseline in Weight by Study Visit |
| Table 14.3.6.4.3 | Safety | Shift from Baseline in Weight by Study Visit and Weight Loss Intentional/Non-Intentional Categories |
| Table 14.3.6.4.4 | Safety | Shift from Baseline in BMI Categories by Study Visit |
| Table 14.3.6.4.5 | Safety | Shift from Baseline in BMI Categories by Study Visit and Weight Loss<br>Intentional/Non-Intentional Categories |
| Table 14.3.6.5 | Safety | Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and Suicidal Behavior by Study Visit |
| Table 14.3.6.6 | Safety | Summary of Physical Examination by Study Visit |
| Table 14.3.6.7 | Safety | Summary of Concomitant Medications by ATC Class Level 4 and Preferred Term |
| 14.4 Pharmaco | kinetic and I | Pharmacodynamic Summary Tables |
| 14.4.1.1 | PK | Summary of Pharmacokinetic Results by Study Visit and Time Point |
| 14.4.1.2 | PK | Summary of Pharmacokinetic Parameters by Study Visit |





### 13.2. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number ARQ-154-204.

In general, one listing will be produced per eCRF domain. All listings will be sorted by treatment, site, and subject number. All calculated variables will be included in the listings. Screen failures will only be presented in Listing 16.2.2.1.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 7: Planned Listings** 

| NT 1 | D 1.4 | mu. |
|---|---|---|
| Number | Population | Title |
| 16.2.1 Subject Disco | ontinuations/Comp | letions |
| Listing 16.2.1.1 | All Subjects | Subject Disposition |
| Listing 16.2.1.2 | All Subjects | Subject Visits |
| 16.2.2 Protocol Dev | iations | |
| Listing 16.2.2.1 | All Subjects | Inclusion and Exclusion Criteria Not Met |
| Listing 16.2.2.2 | All Subjects | Protocol Deviations |
| 16.2.3 Subjects Exc | luded from the Effi | cacy Analyses |
| Listing 16.2.3.1 | All Subjects | Subject Randomization |
| Listing 16.2.3.2 | All Subjects | Analysis Populations |
| 16.2.4 Demographic | Data and Other B | aseline Characteristics |
| Listing 16.2.4.1.1 | All Subjects | Subject Demographics |
| Listing 16.2.4.1.2 | All Subjects | Baseline Characteristics |
| Listing 16.2.4.2 | All Subjects | Medical History |
| 16.2.5 Compliance | and/or Drug Conce | ntration Data |
| Listing 16.2.5.1 | All Subjects | Study Drug Application at the Study Site |
| Listing 16.2.5.2 | All Subjects | Cans |
| Listing 16.2.5.3 | All Subjects | Diary Dispensation |
| Listing 16.2.5.4 | All Subjects | Compliance (CRF) |
| Listing 16.2.5.5 | All Subjects | Missed Doses |
| Listing 16.2.5.6 | PK | Pharmacokinetic Blood Collection |
| Listing 16.2.5.7 | PK | Pharmacokinetic Calculated Parameters |



| Number | Population | Title |
|---|---|---|
| 16.2.6 Individual Et | fficacy Response Da | ita |
| Listing 16.2.6.1 | All Subjects | Scalp Investigator Global Assessment (S-IGA) |
| Listing 16.2.6.2 | All Subjects | Body Investigator Global Assessment (B-IGA) |
| Listing 16.2.6.3 | All Subjects | Psoriasis Scalp Severity Index (PSSI) |
| Listing 16.2.6.4 | All Subjects | Scalp Itch – Numeric Rating Scale (SI-NRS) |
| Listing 16.2.6.5 | All Subjects | Psoriasis Symptoms Diary (PSD) |
| Listing 16.2.6.6 | All Subjects | Psoriasis Area Severity Index (PASI)/Modified PASI (mPASI) |
| Listing 16.2.6.7 | All Subjects | Worst Itch – Numeric Rating Scale (WI-NRS) |
| Listing 16.2.6.8 | All Subjects | Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) |
| Listing 16.2.6.9 | All Subjects | Body Surface Area (BSA) (excluding Palms and Soles) |
| 16.2.7 Adverse Ever | nt Listings (by Subj | ect) |
| Listing 16.2.7.1 | All Subjects | Adverse Events |
| 16.2.8 Laboratory V | Values (by Subject) | |
| Listing 16.2.8.1.1 | All Subjects | Clinical Laboratory Data: Clinical Chemistry |
| Listing 16.2.8.1.2 | All Subjects | Clinical Laboratory Data: Hematology |
| Listing 16.2.8.1.3 | All Subjects | Clinical Laboratory Data: Urinalysis |
| Listing 16.2.8.1.4 | All Subjects | Clinical Laboratory Data: Serum and Urine Pregnancy Test |
| 16.2.9 Other Clinica | al Observations and | Measurements (by Subject) |
| Listing 16.2.9.1 | All Subjects | Investigator Local Tolerability Assessments |
| Listing 16.2.9.2 | All Subjects | Subject Local Tolerability Assessments |
| Listing 16.2.9.3.1 | All Subjects | Vital Signs |
| Listing 16.2.9.3.2 | All Subjects | Vital Signs - Weight |
| Listing 16.2.9.4 | All Subjects | Physical Examination |
| Listing 16.2.9.5 | All Subjects | Medical Photography |
| Listing 16.2.9.6 | All Subjects | Prior and Concomitant Medications |
| Listing 16.2.9.7 | All Subjects | Patient Health Questionnaire (PHQ-8)/Modified PHQ-Adolescents (PHQ-A) |
| Listing 16.2.9.8 | All Subjects | Columbia-Suicide Severity Rating Scale (C-SSRS) |





### 14. Table, Listing, and Figure Shells

## 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all TLFs in support of this study. Note that programming notes may be added if appropriate after each TLF shell.



# Figure 2: Standardized Layout

| Arcutis Biotherapeutics, Inc. Protocol: ARQ-154-204 | Page X of Y |
|---|---|
| <table, figure="" listing,=""> xx.x.x.x <title figure="" listing="" of="" or="" table=""> &lt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;pre&gt;&lt;Note: If directly Applicable&gt; Footnote 1 &lt;if applicable&gt; Recommendation is to keep footnotes to a minimum Footnote 2 &lt;if applicable&gt; Footnote n &lt;if applicable&gt; Footnote n &lt;if applicable&gt; Footnote n+1 &lt;pre&gt;/papplicable&gt;&lt;/pre&gt; Footnote n+1 &lt;/pre&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title></table,> | |



**premier** research



See Figure 3 below.





Figure 3: Planned Table Shells

Summary of Subject Disposition All Randomized Subjects Table 14.1.1

premier research

| | Roflumilast Foam 0.3% | Vehicle | Overall |
|---|---|---|---|
| Status | (X=XX) | (N=XX) | (N=XX) |
| Study Populations: | | | |
| ITT Population [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Safety Population [2] | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) |
| mITT Population [3] | XX (XX.X%) | XX (XX.X%) | XX (XX: X%) |
| SPRU4-ITT Population [4] | XX (XX.X%) | XX (XX. X%) | XX (XX.X%) |
| SPRU4-mITT Population [4] | XX (XX.X%) | XX (XX. X%) | XX (XX.X%) |
| PRU4-ITT Population [5] | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) |
| PRU4-mITT Population [5] | XX (XX.X%) | XX (XX. X%) | XX (XX.X%) |
| PK Population [6] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: COVID-19 = novel coronavirus disease-19; eCRF = electronic case report form; ITT = Intent-to-treat; IP = investigational product; mITT = modified intent-to-treat; IP = principal investigator; PK = pharmacokinetic; PRU4 = Subjects with WI-NRS Pruritus Score ≥4 at Baseline; S-IGA = scalp investigator global assessment; SI-NRS = Scalp Itch – Numeric Rating Scale; SPRU4 = Subjects with SI-NRS Pruritus Score ≥4 at Baseline; WI-NRS = Worst Itch - Numeric Rating Scale.

Note: Percentages are n/Number of subjects randomized within planned treatment and overall\*100.

The ITT population includes all randomized subjects.

[2] The Safety population includes all subjects who are enrolled and received at least 1 confirmed dose of IP.
[3] The mITT population includes all randomized subjects with the exception of subjects who missed the Week 8 disease assessment specifically due to COVID-19 disruptions. [4] The SPRU4-ITT and SPRU4-mITT populations are subsets of the ITT and mITT populations, respectively, and include subjects with SI-NRS pruritus score ≥ 4 at Baseline. These populations will be used for the analyses of achievement of a 4-point reduction in SI-NRS pruritus score as compared to Baseline.

[5] The PRU4-ITT and PRU4-mITT populations are subsets of the ITT and mITT populations, respectively, and include subjects with WI-NRS pruritus score as compared to Baseline. A at Baseline. These populations will be used for the analyses of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline. [6] The PK population includes all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist.

[7] Based on completion of the S-IGA assessment at the Week 8 visit; if a subject is marked as not completing the study in the eCRF but completed the S-IGA assessment at the Week 8 visit before discontinuation, that subject will be considered as a completer for purposes of this summary, and reason for discontinuation is not summarized

Reference Listings: 16.2.1.1, 16.2.3



premier research

| | Roflumilast Foam 0.3% | Vehicle | Overall |
|---|---|---|---|
| Status | (N=XX) | (N=XX) | (N=XX) |
| Completed Study [7] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ongoing in Study | XX (XX.X%) | XX (XX.X%) | (%X.XX) XX |
| Prematurely Discontinued from Study [7] | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX |
| Reason for Discontinuation: | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| Withdrawal by Subject | XX (XX.X%) | (%X:X%) | XX (XX.X%) |
| Sponsor's Decision | XX (XX.X%) | XX (XX. X%) | XX (XX.X%) |
| Pi's Decision | XX (XX.X%) | XX (XX.X%) | XX (XX: X%) |
| Non-Compliance | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| Protocol Violation | XX (XX.X%) | XX (XX.X%) | (%X.XX) XX |
| Lost to Follow-up | XX (XX.X%) | (%X:X%) | XX (XX.X%) |
| Adverse Event | XX (XX.X%) | XX (XX. X%) | XX (XX.X%) |
| Death | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX |
| Pregnancy | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| Other | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX |

Programming note: only display reason for discontinuation if COMPLFL=N, regardless of ADSL.DCREAS.

Abbreviations: COVID-19 = novel coronavirus disease-19; eCRF = electronic case report form; ITT = Intent-to-treat; IP = investigational product; mITT = modified intent-to-treat; PI = principal investigator; PK = pharmacokinetic; PRU4 = Subjects with WI-NRS Pruritus Score ≥4 at Baseline; S-IGA = scalp investigator global assessment; SI-NRS = Scalp Itch – Numeric Rating Scale; SPRU4 = Subjects with SI-NRS Pruritus Score ≥4 at Baseline; WI-NRS = Worst Itch - Numeric Rating Scale.

Note: Percentages are n/Number of subjects randomized within planned treatment and overall\*100.

(1) The ITT population includes all randomized subjects.

[2] The Safety population includes all subjects who are enrolled and received at least 1 confirmed dose of IP.
[3] The mITT population includes all randomized subjects with the exception of subjects who missed the Week 8 disease assessment specifically due to COVID-19 disruptions. [4] The SPRU4-ITT and SPRU4-mITT populations are subsets of the ITT and mITT populations, respectively, and include subjects with SI-NRS pruritus score ≥ 4 at Baseline. These populations will be used for the analyses of achievement of a 4-point reduction in SI-NRS pruritus score as compared to Baseline.

[5] The PRU4-ITT and PRU4-mITT populations are subsets of the ITT and mITT populations, respectively, and include subjects with WI-NRS pruritus score ≥ 4 at Baseline. These populations will be used for the analyses of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline.
[6] The PK population includes all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist.

[7] Based on completion of the S-IGA assessment at the Week 8 visit; if a subject is marked as not completing the study in the eCRF but completed the S-IGA assessment at the Week 8 visit before discontinuation, that subject will be considered as a completer for purposes of this summary, and reason for discontinuation is not summarized.

Reference Listings: 16.2.1.1, 16.2.3



| Status | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Prematurely Discontinued from the Study Due to COVID-19 Disruption | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Reason for Discontinuation: | | | |
| XXXXXXXX | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| XXXXXXXX | XX (XX.X%) | (%X:X%) XX | (%X:X%) |
| XXXXXXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXXXXX | XX (XX.X%) | (%X:X%)<br>XX | (%X:X%) |

Abbreviations: COVID-19 = novel coronavirus disease-19; eCRF = electronic case report form; ITT = Intent-to-treat; IP = investigational product; mITT = modified intent-to-treat; PI = principal investigator; PK = Pharmacokinetic; PRU4 = Subjects with WI-NRS Pruritus Score ≥4 at Baseline; S-IGA = scalp investigator global assessment; SI-NRS = Scalp Itch – Numeric Rating Scale; SPRU4 = Subjects with SI-NRS Pruritus Score ≥4 at Baseline; WI-NRS = Norst Itch - Numeric Rating Scale.

Note: Percentages are n/Number of subjects randomized within planned treatment and overall\*100

1] The ITT population includes all randomized subjects.

COVID-19 disruptions.[4] The SPRU4-ITT and SPRU4-mITT populations are subsets of the ITT and mITT populations, respectively, and include subjects with SI-NRS pruritus score ≥ 4 at Baseline. These populations will be used for the analyses of achievement of a 4-point reduction in SI-NRS pruritus score as [2] The Safety population includes all subjects who are enrolled and received at least 1 confirmed dose of IP.
[3] The mITT population includes all randomized subjects with the exception of subjects who missed the Week 8 disease assessment specifically due to compared to Baseline.

[5] The PRU4-ITT and PRU4-mITT populations are subsets of the ITT and mITT populations, respectively, and include subjects with WI-NRS pruritus score ≥ 4 at Baseline. These populations will be used for the analyses of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline.
[6] The PK population includes all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist.

[7] Based on completion of the S-IGA assessment at the Week 8 visit; if a subject is marked as not completing the study in the eCRF but completed the S-IGA assessment at the Week 8 visit before discontinuation, that subject will be considered as a completer for purposes of this summary, and reason for discontinuation is not summarized.

Reference Listings: 16.2.1.1, 16.2.3

Programming note: "Ongoing in Study" row will be removed once the database has hardlocked and all subjects have completed the study. For COVID-19 Disruption, list only the reasons for discontinuation as populated in the database.

Table 14.1.2.1 Summary of Demographics and Baseline Characteristics Safety Population

**premier** research

| Age (years) Nean (SD) Median Min, Max Age Category 12-17 years ≥18 years | XX | × | |
|---|---|---|---|
| ean (SD) edian in, Max in, Max Category 2-17 years 18 years | XX | | × |
| n, Max<br>Category<br>-17 years<br>8 years | (% X X X X X X X X X X X X X X X X X X X | XX.X (XX.XX) | XX.X (XX.XX) |
| Category<br>2-17 years<br>18 years | (%X XX) XX | XX, XX | XX, XX |
| | XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| ender<br>Male<br>Female | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Child-Bearing Potential? [1]<br>Yes<br>No | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Ethnicity<br>Hispanic or Latino<br>Not Hispanic or Latino | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Race<br>American-Indian or Alaska Native<br>Asian<br>Black or African-American | X (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X:XX)<br>XX (XX:X%)<br>XX (XX:X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Native Hawaiian or Other Pacific Islander<br>White | (%X XX) XX<br>XX (%X XX) XX | (%X:XX)<br>XX (XX:X%) | (%X:XX)<br>XX (XX:X%) |
| Other<br>More than One Race | XX (XX.X%)<br>XX (XX.X%) | (%X:X%)<br>XX (XX:X%) | (%X:X%)<br>XX (XX:X%) |

Index; SI-NRS = Scalp Itch – Numeric Rating Scale; PSD = Psoriasis Symptoms Diary; PASI = Psoriasis Area Severity Index; mPASI = modified PASI; WI-NRS = Worst Itch – Numeric Rating Scale; DLQI = Dermatology Life Quality Index; CDLQI = Children's DLQI.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Abbreviations: S-IGA = scalp investigator global assessment; B-IGA = body investigator global assessment; PSSI = Psoriasis Scalp Severity

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population. [2] The SI-NRS was determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10,

Which ranges from "no scalp itch" to "worst scalp itch imaginable".
[3] The WI-NRS was determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".
Reference Listings: 16.2.4.1.1, 16.2.4.1.2, 16.2.6.1, 16.2.6.2, 16.2.6.3, 16.2.6.5, 16.2.6.5, 16.2.6.7, 16.2.9.4.1, 16.2.9.4.2



Table 14.1.2 (cont.)
Demographics and Baseline Characteristics
Safety Population

| Variable<br>Statistic or Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Height (cm)<br>n<br>Mean (SD)<br>Median<br>Min, Max | ()<br>XX XX<br>XX XX<br>XX XX<br>XX XX | × | ×××××××××××××××××××××××××××××××××××××× |
| Weight (kg)<br>n<br>Mean (SD)<br>Median<br>Min, Max | XX | XX | XX XX (XX.XX) XX |
| Body Mass Index (kg/m²)<br>n<br>Mean (SD)<br>Median<br>Min, Max | XX | (XX XX | XX |
| Body Surface Area (%) Affected by Disease<br>n<br>Mean (SD)<br>Median<br>Min, Max | (X | (X; X; X | (X |

Abbreviations: S-IGA = scalp investigator global assessment; B-IGA = body investigator global assessment; PSSI = Psoriasis Scalp Severity Index; SI-NRS = Scalp Itch – Numeric Rating Scale; PSD = Psoriasis Symptoms Diary; PASI = Psoriasis Area Severity Index; mPASI = modified PASI; WI-NRS = Worst Itch – Numeric Rating Scale; DLQI = Dermatology Life Quality Index; CDLQI = Children's DLQI.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population. Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100.

<sup>[2]</sup> The SI-NRS was determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10, which ranges from "no scalp itch" to "worst scalp itch imaginable".
[3] The WI-NRS was determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".



Table 14.1.2.1 (cont.) Demographics and Baseline Characteristics Safety Population

| Variable<br>Statistic or Category | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline S-IGA<br>Clear | (%X XX) XX | XX (XX.X%) | (%X:XX) XX |
| Almost Clear | XX (XX X%) | XX (XX.X%) | (%X:XX) XX |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX: X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Baseline S-IGA - Numeric | | | |
| n | × | × | × |
| Mean (SD) | XX:X (XX:XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | ××× | ××× | ××× |
| Min, Max | XX | XX, XX | X, XX |
| Baseline B-IGA | | | |
| Clear | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| Almost Clear | XX (XX.X%) | (%X:X%) XX | (%X:X%) XX |
| Mild | (%X:X%) XX | (%X:XX) XX | (%X:XX) XX |
| Moderate | (%X:X%) XX | (%X:XX) XX | (%X:XX) XX |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Baseline B-IGA - Numeric | | | |
| n | × | × | × |
| Mean (SD) | XX:X (XX:XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | ××× | ×.×× | XXX |
| Min, Max | ××,×× | ×××× | ×××× |

Abbreviations: S-IGA = scalp investigator global assessment; B-IGA = body investigator global assessment; PSSI = Psoriasis Scalp Severity Index; SI-NRS = Scalp Itch – Numeric Rating Scale; PSD = Psoriasis Symptoms Diary; PASI = Psoriasis Area Severity Index; mPASI = modified PASI; WI-NRS = Worst Itch – Numeric Rating Scale; DLQI = Dermatology Life Quality Index; CDLQI = Children's DLQI.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. [1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population.

[2] The SI-NRS was determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10, which

ranges from "no scalp itch" to "worst scalp itch imaginable".
[3] The WI-NRS was determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".
Reference Listings: 16.2.4.1.1, 16.2.4.1.2, 16.2.6.1, 16.2.6.3, 16.2.6.3, 16.2.6.5, 16.2.6.6, 16.2.6.7, 16.2.6.8, 16.2.9.3.1, 16.2.9.3.2



Table 14.1.2.1 (cont.)
Demographics and Baseline Characteristics Safety Population

| Variable | Roflumilast Foam 0.3% | Vehicle | Overall |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Baseline PSSI - Numeric | | | |
| 2 | × | × | × |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XXX | ××× | ××× |
| Min, Max | X, X | XX, XX | XX, XX |
| Baseline SI-NRS - Numeric [2] | | | |
| | × | × | × |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XXX | ××× | ××× |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Baseline SI-NRS [2] | | | |
| 0 | XX (XX.X%) | XX (XX: X%) | XX (XX:X%) |
| _ | XX (XX.X%) | XX (XX: X%) | XX (XX:X%) |
| 2 | XX (XX.X%) | XX (XX: X%) | XX (XX:X%) |
| 8 | XX (XX. X%) | XX (XX: X%) | XX (XX:X%) |
| 4 | XX (XX.X%) | (%X:X%) | XX (XX:X%) |
| 2 | XX (XX: X%) | XX (XX.X%) | (%X:XX) |
| 9 | XX (XX: X%) | XX (XX.X%) | (%X:XX) |
| 7 | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| 8 | XX (XX.X%) | (%X:X%) | XX (XX:X%) |
| 0 | XX (XX.X%) | XX (XX: X%) | XX (XX:X%) |
| 10 | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) |

Abbreviations: S-IGA = scalp investigator global assessment; B-IGA = body investigator global assessment; PSSI = Psoriasis Scalp Severity Index; SI-NRS = Scalp Itch – Numeric Rating Scale; PSD = Psoriasis Symptoms Diary; PASI = Psoriasis Area Severity Index; mPASI = modified PASI; WI-NRS = Worst Itch – Numeric Rating Scale; DLQI = Dermatology Life Quality Index; CDLQI = Children's DLQI.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population.
[2] The SI-NRS was determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10, which

ranges from "no scalp itch" to "worst scalp itch imaginable".

[3] The WI-NRS was determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch". Reference Listings: 16.2.4.1.1, 16.2.4.1.2, 16.2.6.1, 16.2.6.3, 16.2.6.4, 16.2.6.5, 16.2.6.6, 16.2.6.7, 16.2.6.8, 16.2.9.3.1, 16.2.9.3.2



| Overall (N=XX) | XX | XX | XX.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|
| Vehicle<br>(N=XX) | XX.X(XX.XX)<br>XX.X.XX<br>XX.XX | XX | (XX.XX)<br>XX.XX<br>XX.XX |
| Roflumilast Foam 0.3% (N=XX) | XX | XX.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX XX (XX.XX) XX.X XX XX XX |
| Variable<br>Statistic or Category | Baseline PSD Total Score<br>n<br>Mean (SD)<br>Median<br>Min, Max | Baseline PASI<br>n<br>Mean (SD)<br>Median<br>Min, Max | Baseline mPASI<br>n<br>Mean (SD)<br>Median<br>Min, Max |

Abbreviations: S-IGA = scalp investigator global assessment; B-IGA = body investigator global assessment; PSSI = Psoriasis Scalp Severity Index; SI-NRS = Scalp Itch – Numeric Rating Scale; PSD = Psoriasis Symptoms Diary; PASI = Psoriasis Area Severity Index; mPASI = modified PASI; WI-NRS = Worst Itch – Numeric Rating Scale; DLQI = Dermatology Life Quality Index; CDLQI = Children's DLQI.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population. [2] The SI-NRS was determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10,

which ranges from "no scalp itch" to "worst scalp itch imaginable".
[3] The WI-NRS was determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".



Table 14.1.2.1 (cont.)
Demographics and Baseline Characteristics Safety Population

| Overall (N=XX) | XX | (%X:X%)<br>(%X:X%)<br>(%X:X%)<br>(%X:X%)<br>(XX:X%)<br>(XX:X% |
|---|---|---|
| Vehicle<br>(N=XX) | XX.X(XX.XX) XX.X XX.X XX.X | (%(%(%(%(%(%(%(%(%(%(%(%(%(%(%(%(%(%(% |
| Roflumilast Foam 0.3% (N=XX) | XX.X (XX.XX)<br>XX.X<br>XX, XX | (%(%(%(%)(%)(%)(%)(%)(%)(%)(%)(%)(%)(%)( |
| Variable<br>Statistic or Category | Baseline WI-NRS - Numeric [3]<br>n<br>Mean (SD)<br>Median<br>Min, Max | Baseline WI-NRS [3] 0 1 2 3 4 5 6 7 10 |

Abbreviations: S-IGA = scalp investigator global assessment; B-IGA = body investigator global assessment; PSSI = Psoriasis Scalp Severity Index; SI-NRS = Scalp Itch – Numeric Rating Scale; PSD = Psoriasis Symptoms Diary; PASI = Psoriasis Area Severity Index; mPASI = modified PASI; WI-NRS = Worst Itch – Numeric Rating Scale; DLQI = Dermatology Life Quality Index; CDLQI = Children's DLQI. Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population.
[2] The SI-NRS was determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10, which ranges from "no scalp itch" to "worst scalp itch imaginable".
[3] The WI-NRS was determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch".



Table 14.1.2.1 (cont.)
Demographics and Baseline Characteristics Safety Population

| Variable | Roflumilast Foam 0.3% | Vehicle | Overall |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Baseline DLQI | | | |
| u | × | × | × |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | ××× | ××× | ××× |
| Min, Max | ××,×× | ××× | ××× |
| | | 3 | } |
| C | × | × | × |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | ××× | ××× | ××× |
| Min, Max | X, X | XX, XX | XX XX |

Abbreviations: S-IGA = scalp investigator global assessment; B-IGA = body investigator global assessment; PSSI = Psoriasis Scalp Severity Index; SI-NRS = Scalp Itch – Numeric Rating Scale; PSD = Psoriasis Symptoms Diary; PASI = Psoriasis Area Severity Index; mPASI = modified PASI; WI-NRS = Worst Itch – Numeric Rating Scale; DLQI = Dermatology Life Quality Index; CDLQI = Children's DLQI.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety population.
[2] The SI-NRS was determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10, which ranges from "no scalp itch" to "worst scalp itch imaginable".
[3] The WI-NRS was determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges

from "no itch" to "worst imaginable itch".



(Same shell as Table 14.1.2.1; subjects are summarized by planned treatment, not treatment received; Update Note: footnote as Percentages are n/Number of subjects in the ITT population within planned treatment and overall\*100.)

Table 14.1.2.3
Summary of Demographics and Baseline Characteristics
mITT Population

(Same shell as Table 14.1.2.1; subjects are summarized by planned treatment, not treatment received; Update Note: footnote as Percentages are n/Number of subjects in the mITT population within planned treatment and overall\*100.)

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



Table 14.1.3
Previous Treatment History of Scalp and Body Psoriasis
Safety Population

| Category | Roflumilast Foam 0.3%<br>(N=XX) | Vehide<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Inadequate Response, Intolerance or<br>Contraindication to<br>Topical Corticosteroids<br>Topical Vitamin D Derivatives<br>Missing | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Subject has Psoriasis Involvement on<br>Knees and/or Elbow<br>Genitalia<br>Missing | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%X`XX) XX<br>(%X`XX) XX<br>(%X`XX) XX |

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Subjects with a response of "Yes" are summarized.

Reference Listing: 16.2.4.2

Programming note: Only display Missing rows if a subject does not have an answer to the questions on the CRF regarding previous treatment and/or psoriasis involvement.



**premier** research

| Category | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with Any Protocol Deviations | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with Major Protocol Deviations | XX (XX.X%) | (%X:XX) | XX (XX:X%) |
| XXXXXXXXXXXXX | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) |
| XXXXXXXXXXXXX | XX (XX:X%) | XX (XX.X%) | XX (XX: X%) |
| XXXXXXXXXX | XX (XX:X%) | XX (XX.X%) | XX (XX: X%) |

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Only major protocol deviations are presented. Subjects with any protocol deviations row can include counts from major and minor deviations. Subjects with one or more deviations within a type of protocol deviation were counted only once. Protocol Deviations were collected throughout the

Reference Listing: 16.2.2.2

Programming note: the structure of this table may change depending on the information in the protocol deviations file.



| ATC Class Level 4<br>Preferred Term | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with at least 1 Prior Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX X%) | XX (XX.X%) | XX (XX. X%) |
| Preferred Term 3 | XX (XX X%) | XX (XX.X%) | XX (XX. X%) |
| ATC Class 2 | (%X:X%) | (XX:X%) | (%X:X%) |
| Preferred Term 1 | XX (XX:X%) | XX (XX:X%) | XX (XX:X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX. X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX. X%) |

Abbreviations: ATC = Anatomic Therapeutic Chemical; PT = preferred term; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Medications were coded using WHO-DDE Global B3 version September 2019. Prior medications are all medications that were started before the application of study drug. Medications are displayed by alphabetical order of ATC Level 4 classification, then descending frequency of PT within ATC, and then alphabetically by PT. Subjects were counted only once for each ATC and PT.

Reference Listing: 16.2.9.6

Programming note: ATC & PT text should be presented as is from the dataset.



Table 14.1.6 Summary of Study Drug Exposure and Compliance Safety Population

| Variable<br>Statistic / Category | Roflumilast Foam 0.3% (N=XX) | Vehicle (N=XX) |
|---|---|---|
| Total Number of IP Applications<br>n<br>Mean (SD)<br>Median<br>Min, Max | XX.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX |
| Total Weight of IP Applied (g) [1] n Mean (SD) Median Min, Max | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ××××<br>××××<br>×××× |
| Compliance [2]<br>>100%<br>≥ 80% - ≤100%<br>< 80% | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| > 3 Consecutive Missed Doses<br>Compliant [3] | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |

Abbreviation: IP = investigational product. Note: n is the number of subjects in the Safety Note: n is the number of subjects in the Safety Population within treatment received\*100.

[1] Total weight of IP is determined by subtracting returned can weight from the dispensed can weight. [2] Compliance is calculated based on number of applications divided by the expected number of IP applications for each subject\*100.

[3] A subject is considered compliant if the subject applies at least 80% of the expected applications during the IP application period and does not miss more than 3 consecutive doses.

Reference Listings: 16.2.5.1, 16.2.5.2, 16.2.5.4

Table 14.2.1.1 Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit – Observed Data ITT Population

| | Roflumilast | Roflumilast Foam 0.3% | Vehicle | icle |
|---|---|---|---|---|
| Study Visit | (XX=N) | (XX | XX=N) | (X |
| Statistic | Observed | Change | Observed | Change |
| Baseline | | | | |
| n | × | | × | |
| Mean (SD) | XX.X (X.XX) | | XX.X (X.XX) | |
| Median | XXX | | XXX | |
| Min, Max | ×××× | | ××× | |
| Q1, Q3 | XXX | | XXX | |
| Week 2 | | | | |
| _ | × | × | × | × |
| Mean (SD) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) |
| Median | ××× | ××× | XX.Xs | ××× |
| Min, Max | ××× | ×××× | ××× | ××× |
| Q1, Q3 | ××× | ××× | ××× | ××× |

Repeat for Week 4, Week 8, Week 9.

Abbreviation: S-IGA = scalp investigator global assessment.

Note: Subjects are summarized by planned treatment. S-IGA is a static qualitative evaluation of overall psoriasis severity involving an ordinal scale with 5 severity grades (reported only in integers of 0 to 4) where 0 = Clear; 1 = Almost Clear; 2 = Mild; 3 = Moderate; 4 = Severe. Baseline is the last non-missing measurement taken before the first application of study drug. Change from baseline is calculated as result – baseline result.

Reference Listing: 16.2.6.1



Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit - Observed Data mITT Population Table 14.2.1.2

(Same shell as Table 14.2.1.1)

Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit – Multiple Imputation Table 14.2.1.3

ITT Population

pattern, a predictive mean matching model was used to impute missing value for a subject at particular visit having baseline S-IGA score, treatment group, and country as independent variables and study visit as dependent variable. For non-monotone missing IGA values, Markov-Chain Monte Carlo (MCMC) method was used to impute the data at intermediate visits (Same shell as Table 14.2.1.1; add "B-IGA = body investigator global assessment" to abbreviations in alphabetical order; Programming note: update "Note:" portion of footnote to add in the following text just after "Note:": Separate multiple imputation steps were used for monotone and non-monotone missing data. For monotone missing to make the missing data pattern into monotone before applying the predictive mean matching multiple imputation algorithm. )

Summary and Change from Baseline in Scalp Investigator Global Assessment (S-IGA) Grades by Study Visit – Multiple Imputation mITT Population Table 14.2.1.4

pattern, a predictive mean matching model was used to impute missing value for a subject at particular visit having baseline S-IGA score, treatment group, and country as independent variables. For non-monotone missing IGA values, Markov-Chain Monte Carlo (MCMC) method was used to impute the data at intermediate visits Same shell as Table 14.2.1.1; add "B-IGA = body investigator global assessment" to abbreviations in alphabetical order; Programming note: update "Note:" portion of footnote to add in the following text just after "Note:": Separate multiple imputation steps were used for monotone and non-monotone missing data. For monotone missing to make the missing data pattern into monotone before applying the predictive mean matching multiple imputation algorithm.)

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results
ITT Population Table 14.2.1.5.1

| Study Visit | Roflumilast Foam 0.3% | Vehicle |
|---|---|---|
| Category/Statistic | (YY=NI) | (XX=NI) |
| Baseline | × | × |
| O = Clear | (%X XX) XX | (%x xx) xx |
| 1 = Almost Clear | (%X:XX) XX | (%X:XX) XX |
| 2 = Mild | (%X:XX) XX | (%X:XX) XX |
| 3 = Moderate | (%X:XX) XX | (%X:XX) |
| 4 = Severe | xx (xx.x%) | XX (XX.X%) |
| Week 2 | × | × |
| 0 = Clear | XX (XX:X%) | XX (XX.X%) |
| 1 = Almost Clear | XX (XX:X%) | XX (XX.X%) |
| 2 = Mild | XX (XX.X%) | XX (XX.X%) |
| 3 = Moderate | XX (XX:X%) | (%X:X%) |
| 4 = Severe | XX (XX.X%) | XX (XX.X%) |
| S-IGA Success [1] | | |
| Yes | XX (XX.X%) | XX (XX.X%) |
| 95% CI [2] | (X.XX, X.XX) | (XXX, XXX) |
| No | XX (XX.X%) | XX (XX.X%) |
| Odds Ratio (95% CI) [3]<br>P value [3] | X.XX (X.XX, X.XX)<br>X.XXXX | |

# Repeat for all Week 4, Week 8, and Week 9.

Abbreviations: B-IGA = body investigator global assessment; CI = confidence interval; S-IGA = scalp investigator global assessment.

Note: Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100. Baseline is the last non-missing measurement taken before the first application of study drug. [1] S-IGA Success ("Yes") is defined as an S-IGA score of "Clear" or "Almost Clear" plus a ≥2-grade improvement from baseline; "No" otherwise.

[2] 95% Cls for "Yes" are obtained using Wilson method.
[3] The odds ratio, 95% Cl, and P value are obtained from Cochran Mantel Haenszel test (stratified by country, baseline S-IGA category, and baseline B-IGA category) comparing roflumilast foam 0.3% to vehicle. Reference Listings: 16.2.6.1, 16.2.6.2





Table 14.2.1.5.2 Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results

ITT Population - Topical Corticosteroids - Naïve Subjects

(Same shell as Table 14.2.1.5.1; add 16.2.4.2 to reference listings; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that are topical corticosteroids – naïve subjects within planned treatment at each visit\*100.")

Table 14.2.1.5.3 Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data

Categorical Results

ITT Population - Topical Vitamin D Derivative - Naïve Subjects

(Same shell as Table 14.2.1.5.1; add 16.2.4.2 to reference listings; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that are topical vitamin D derivative - naive subjects within planned treatment at each visit\*100.")

Table 14.2.1.5.4

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results

ITT Population - Subjects with Psoriasis Involvement on the Knee and/or Elbow

(Same shell as Table 14.2.1.5.1; add 16.2.4.2 to reference listings; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that have psoriasis involvement on the knee and/or elbow within planned treatment at each visit\*100.")

Table 14.2.1.5.5

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Observed Data

Categorical Results

ITT Population - Subjects who Achieved S-IGA and B-IGA Success at Week 8

(Same shell as Table 14.2.1.5.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that achieved both S-IGA and B-IGA suclass at Week 8 within planned treatment at each visit\*100.")




Table 14.2.1.5.6 Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results

ITT Population - by Study Site

| Study Site: SITENAM (Site SITEID) | | | |
|---|---|---|---|
| Study Visit | Roflumilast Foam 0.3% | Vehicle | |
| Category/Statistic | (N=XX) | (N=XX) | - 1 |
| : | | | |
| Baseline | × | × | |
| 0 = Clear | XX (XX.X%) | XX (XX:X%) | |
| 1 = Almost Clear | (%X:XX) | (%X:XX) XX | |
| 2 = Mild | XX XXX XX | (%X:XX)<br>XX | |
| 3 = Moderate | XX (XX.X%) | (%X:XX) XX | |
| 4 = Severe | XX (XX.X%) | xx (xx.x%) | |
| Week 2 | × | × | |
| 0 = Clear | XX (XX.X%) | XX (XX.X%) | |
| 1 = Almost Clear | XX (XX.X%) | XX (XX: X%) | |
| 2 = Mild | XX (XX.X%) | XX (XX: X%) | |
| 3 = Moderate | XX (XX:X%) | XX (XX: X%) | |
| 4 = Severe | XX (XX.X%) | xx (xx.x%) | |
| S-IGA Success [1] | | | |
| Yes | XX (XX.X%) | (%X:XX) | |
| 95% CI [2] | (X.XX, X.XX) | (X.XX, X.XX) | |
| No | XX (XX.X%) | XX (XX.X%) | |
| Odds Ratio (95% CI) [3]<br>P value [3] | X.XX (X.XX, X.XX)<br>X.XXXX | | |

# Repeat for all Week 4, Week 8, and Week 9.

Abbreviations: B-IGA = body investigator global assessment; CI = confidence interval; S-IGA = scalp investigator global assessment.

Note: Percentages are n/Number of subjects in the ITT population within planned treatment and study site at each visit\*100. Baseline is the last non-missing measurement taken before the first application of study drug.

[1] S-IGA Success ("Yes") is defined as an S-IGA score of "Clear" or "Almost Clear" plus a ≥2-grade improvement from baseline; "No"

otherwise.

[2] 95% CIs for "Yes" are obtained using Wilson method.
[3] The odds ratio, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by country, baseline S-IGA category, and baseline B-IGA category) comparing roflumilast foam 0.3% to vehicle.
Reference Listings: 16.2.6.1, 16.2.6.2

Programming note: sort by ADSL.SITEID. Format study site as shown (e.g., "Study Site Name (Site 01)").



Table 14.2.1.6.1 Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results mITT Population

(Same shell as Table 14.2.1.5)

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Observed Data Categorical Results Table 14.2.1.6.2

mITT Population - Topical Corticosteroids - Naïve Subjects

(Same shell as Table 14.2.1.5.2; add 16.2.4.2 to reference listings; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that are topical corticosteroids – naïve subjects within planned treatment at each visit\*100.")

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Observed Data Table 14.2.1.6.3

mITT Population - Topical Vitamin D Derivative - Naïve Subjects Categorical Results

(Same shell as Table 14.2.1.5.3; add 16.2.4.2 to reference listings; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that are topical vitamin D derivative – naïve subjects within planned treatment at each visit\*100.")

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Observed Data Categorical Results Table 14.2.1.6.4

mITT Population - Subjects with Psoriasis Involvement on the Knee and/or Elbow

(Same shell as Table 14.2.1.5.4; add 16.2.4.2 to reference listings; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT that have psoriasis involvement on the knee and/or elbow within planned treatment at each visit\*100.")




**premier** research

Table 14.2.1.6.5 Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data Categorical Results

mITT Population - Subjects who Achieved S-IGA and B-IGA Success at Week 8

(Same shell as Table 14.2.1.5.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that achieved both S-IGA and B-IGA success at Week 8 within planned treatment at each visit\*100.")

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Observed Data Categorical Results mITT Population – by Study Site Table 14.2.1.6.6

(Same shell as Table 14.2.1.5.6; )





Table 14.2.1.7.1

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation Categorical Results

ITT Population

(Same shell as Table 14.2.1.5.1; add "B-IGA = body investigator global assessment" to abbreviations in alphabetical order; update "Note:" portion of footnote to add in the matching model was used to impute missing value for a subject at particular visit having baseline S-IGA score, treatment group, and country as independent variables and study visit following text just after "Note:". Separate multiple imputation steps were used for monotone and non-monotone missing data. For monotone missing pattern, a predictive mean as dependent variable. For non-monotone missing IGA values, Markov-Chain Monte Carlo (MCMC) method was used to impute the data at intermediate visits to make the missing data pattern into monotone before applying the predictive mean matching multiple imputation algorithm.)

Table 14.2.1.7.2

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results

ITT Population – Baseline S-IGA = 3

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that have a baseline S-IGA score of 3 within planned treatment at each visit\*100.")

Table 14.2.1.7.3

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results

ITT Population – Baseline S-IGA = 4

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that have a baseline S-IGA score of 4 within planned treatment at each visit\*100.")



Table 14.2.1.7.4

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation Categorical Results

ITT Population – Age Category = 12-17 Years

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that are between 12 and 17 years of age, inclusive, within planned treatment at each visit\*100.")

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation Table 14.2.1.7.5

Categorical Results
ITT Population – Age Category = ≥18 Years

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that are aged 18 years or older within planned treatment at each visit\*100.")

Table 14.2.1.7.6

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation

Categorical Results
ITT Population – Subjects who Achieved S-IGA and B-IGA Success at Week 8

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the ITT population that achieved both S-IGA and B-IGA subjects in the ITT population that achieved both S-IGA and B-IGA and B-IGA and Italian success at Week 8 within planned treatment at each visit\*100.")




Table 14.2.1.8.1 Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation

Categorical Results mITT Population

(Same shell as Table 14.2.1.7.1)

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation Table 14.2.1.8.2

Categorical Results mITT Population – Baseline S-IGA = 3

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that have a baseline S-IGA score of 3 within planned treatment at each visit\*100.")

Table 14.2.1.8.3

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation

Categorical Results

mITT Population – Baseline S-IGA = 4

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that have a baseline S-IGA score of 4 within planned treatment at each visit\*100.")




Table 14.2.1.8.4 Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Multiple Imputation Categorical Results

mITT Population - Age Category = 12-17 Years

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that are between 12 and 17 years of age, inclusive, within planned treatment at each visit\*100.")

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation Categorical Results Table 14.2.1.8.5

mITT Population – Age Category = ≥18 Years

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that are aged 18 years or older within planned treatment at each visit\*100.")

Table 14.2.1.8.6

Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit - Multiple Imputation

mITT Population – Subjects who Achieved S-IGA and B-IGA Success at Week 8 Categorical Results

(Same shell as Table 14.2.1.7.1; change "Percentages" footnote to be "Percentages are n/Number of subjects in the mITT population that achieved both S-IGA and B-IGA success at Week 8 within planned treatment at each visit\*100.")






| | | Roflumik<br>( | Roflumilast Foam 0.3% (N=XX) | | Vehicle<br>(N=XX) | (Roflum | Treatment Difference (Roflumilast Foam 0.3% vs Vehicle) [3] | 3] |
|---|---|---|---|---|---|---|---|---|
| XXX | Study Visit | n [1] | Responder [2] | n [1] | Responder [2] | Odds Ratio | 95% CI for OR | P value |
| XX.X | Week 2 | × | | × | %X:X% | ××× | (XX.XX, XX.XX) | X.XXXX |
| XX.X | Week 4 | × | | × | %X:X% | ××× | (XX.XX, XX.XX) | XXXXX |
| XX.X | Week 8 | × | | × | %X:X% | ××× | (XX.XX, XX.XX) | X.XXXX |
| | Week 9 | × | | × | %X:X% | XX.X | (XX.XX, XX.XX) | X.XXXX |

Abbreviations: CI = Confidence interval; OR = odds ratio; S-IGA = scalp investigator global assessment.

Note: Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100. Baseline is the last non-missing measurement taken before the first application of study drug.

[1] Number of subjects at each visit.

subject correlation. In case of convergence issues, other covariance structures will be used including Toeplitz, compound symmetry or Autoregressive (1) (AR[1]) covariance structure will be used, following this sequence until convergence is achieved. The odds ratio is the estimate of the odds of having S-IGA response for subjects treated with dependent variable and treatment, country, visit, and baseline S-IGA score as the independent variables. An unstructured correlation matrix was used to model the within [2] Number of subjects with an S-IGA score of "Clear" or "Almost Clear" plus a ≥2-grade improvement from baseline.
[3] Estimates for odds ratio, 95% CI for odds ratio, and P value are from a generalized estimating equations for binary response model, with S-IGA success as the roflumilast foam 0.3% relative to that for subjects treated with vehicle. Reference Listing: 16.2.6.1

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



**premier** research

Table 14.2.1.10
Summary of Scalp Investigator Global Assessment (S-IGA) Grades and Success by Study Visit – Observed Data
Tabulation of Fitted Point Estimates from Generalized Estimating Equations for Binary Response
mITT Population

(Programming note: Same as table shell 14.2.1.9)

Table 14.2.1.11 Summary of Scalp Investigator Global Assessment (S-IGA) – Score of Clear – Observed Data ITT Population

**premier** research

| Study Visit | Roflumilast Foam 0.3% | Vehicle |
|---|---|---|
| Categoly/Statistic | (VV=NI) | (V-N) |
| Week 2 | × | × |
| S-IGA Clear [1] | | |
| Yes | XX (XX.X%) | (%X:XX) XX |
| 95% CI [2] | (X.XX, X.XX) | (X X X XX) |
| No | XX (XX.X%) | XX (XX.X%) |
| Odds Ratio (95% CI) [3]<br>P value [3] | X.XX (X.XX, X.XX)<br>X.XXXX | |

Repeat for all Week 4, Week 8, and Week 9.

Abbreviations: CI = confidence interval; S-IGA = scalp investigator global assessment.

Note: Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100. Baseline is the last non-missing measurement taken before the first application of study drug.

[1] S-IGA Clear ("Yes") is defined as an S-IGA score of "Clear"; "No" otherwise.

[2] 95% CIs for "Yes" are obtained using Wilson method.

[3] The odds ratio, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by country, baseline S-IGA category, and baseline B-IGA category) comparing roflumilast foam 0.3% to vehicle. Reference Listing: 16.2.6.1





Table 14.2.1.12 Summary of Scalp Investigator Global Assessment (S-IGA) – Score of Clear – Observed Data mITT Population

(Same as table shell 14.2.1.11)

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



Figure 14.2.1.13
Plot of Scalp Investigator Global Assessment (S-IGA) Tipping Point Analysis
P Values vs Shift Parameters
ITT Population



Abbreviation: MNAR = missing not at random.

changes substantially and is used to check the robustness of the imputation. Shift parameters from -1.5 to 1.5 by 0.2 were initially used to determine approximately where results of the analysis are shifted from significant (i.e., P ≤ 0.05) to non-significant (i.e., P > 0.05). Once this was determined, the range around the approximate inflection point was expanded to include values with greater precision (i.e., to 2 decimal places, by 0.01); this expanded range of shift parameters and P Note: A tipping point analysis was performed in order to determine the inflection point at which the inference under the MNAR assumption for multiple imputation values are presented here. If this tipping point value is considered clinically implausible, then there is evidence of efficacy with respect to the primary endpoint despite missing data.



Figure 14.2.1.14
Plot of Scalp Investigator Global Assessment (S-IGA) Tipping Point Analysis
P Values vs Shift Parameters
mITT Population

(Programming note: Same as figure shell 14.2.1.13)

Table 14.2.2.1
Summary and Change from Baseline in Body Investigator Global Assessment (B-IGA) Grades by Study Visit
ITT Population

(Programming note: Same as table shell 14.2.1.1; update reference listing to Reference Listing: 16.2.6.2; Update any instances of S-IGA to B-IGA)

Table 14.2.2.2 Summary and Change from Baseline in Body Investigator Global Assessment (B-IGA) Grades by Study Visit mITT Population (Programming note: Same as table shell 14.2.1.1; update reference listing to Reference Listing: 16.2.6.2; Update any instances of S-IGA to B-IGA)

Table 14.2.2.3
Summary of Body Investigator Global Assessment (B-IGA) Grades and Success by Study Visit
Categorical Results

ITT Population

(Programming note: Same as table 14.2.1.5; update reference listing to Reference Listings: 16.2.6.1, 16.2.6.2; Update any instances of S-IGA to B-IGA)

Table 14.2.2.4
Summary of Body Investigator Global Assessment (B-IGA) Grades and Success by Study Visit
Categorical Results
mITT Population

(Programming note: Same as table 14.2.1.5; update reference listing to Reference Listing: 16.2.6.2; Update any instances of S-IGA to B-IGA)



Table 14.2.3.1 Summary and Change from Baseline in PSSI Scores by Study Visit ITT Population

| 8^ |
|----------------|
| XX, XX<br>XX.X |
| ××××× |

Repeat for Week 4, Week 8, Week 9.

Abbreviation: PSSI = Psoriasis Scalp Severity Index.

Note: Subjects are summarized by planned treatment. PSSI total score is calculated as (erythema score + induration + desquamation) × extent of scale affected. The score ranges from 0 to 72. Erythema, induration, and desquamation are scored on a scale of 0 to 4, where 0 = absent and 4 = severest possible; extent of scale affected is scored on a scale of 0 to 6, where 0 = 0% of involved area and 6 = 90-100% of involved area. Baseline is the last non-missing measurement taken before the first application of study drug. Change from baseline is calculated as result – baseline result. Percent change from baseline is calculated as (change from baseline)\*100. Reference Listing: 16.2.6.3



Table 14.2.3.2 Summary and Change from Baseline in PSSI Scores by Study Visit mITT Population

(Programming note: Same as table 14.2.3.1)



ITT Population

| Study Visit<br>Category/Statistic | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
|---|---|---|
| Week 2 | X | × |
| 700-50 [1]<br>768<br>569 745 | XX (XX. X%) | XX (XX.X%) |
| 95% CI [5]<br>No | (X.X.X%)<br>XX (XX.X%) | XX (XX.X%) |
| Odds Ratio (95% CI) [6]<br>P value [6] | X.XX (X.XX, X.XX)<br>X.XXXX | |
| PSSI-75 [2]<br>Yes | XX (XX.X%) | XX (XX.X%) |
| 93% CI [3]<br>No | (X.X.X%)<br>XX (XX.X%) | (%.X., %.%%)<br>XX (XX.X%) |
| Odds Ratio (95% CI) [6]<br>P value [6] | X.XX (X.XX, X.XX)<br>X.XXXX | X.XX (X.XX, X.XX) |

## Continue for PSSI-90 [3] and PSSI-100 [4]; Repeat for Week 4, Week 8, and Week 9.

Abbreviations: B-IGA = body investigator global assessment; CI = confidence interval; S-IGA = scalp investigator global assessment; PSSI = Psoriasis Scalp Severity Index

Note: Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100. Baseline is the last non-

missing measurement taken before the first application of study drug.

[1] PSSI-50 is populated with "Yes" when there is an achievement of a 50% reduction in PSSI total score from baseline; "No" otherwise.

[2] PSSI-75 is populated with "Yes" when there is an achievement of a 75% reduction in PSSI total score from baseline; "No" otherwise.

[3] PSSI-90 is populated with "Yes" when there is an achievement of a 90% reduction in PSSI total score from baseline; "No" otherwise.

[4] PSSI-100 is populated with "Yes" when there is an achievement of a 100% reduction in PSSI total score from baseline; "No" otherwise.

[5] 95% CI for "Yes" are obtained using Wilson method.

[6] The odds ratio, 95% CI, and P value are obtained from Cochran Mantel Haenszel test (stratified by country, baseline S-IGA score category) comparing roflumilast foam 0.3% to vehicle.

Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.3





Table 14.2.3.4 Summary of Achievement of PSSI-50, PSSI-75, PSSI-90, and PSSI-100 by Study Visit mITT Population

(Programming note: Same as table 14.2.3.3.)

Table 14.2.3.5 Time to Achievement of PSSI-50, PSSI-75, and PSSI-90 ITT Population

**premier** research

| Variable<br>Statistic | Roflumilast Foam 0.3% (N=XXX) | Vehicle<br>(N=XXX) |
|---|---|---|
| Time to Achieve PSSI-50 (Days) [1]<br>n | ×× | × |
| Events/Censors [2]<br>Mean (SD) | XX/XX<br>XXXX X | XX/XX<br>XXXX XXX |
| Median<br>Min, Max | ××× | ××× |
| Kaplan-Meier Estimate of Time to Achieve PSSI-50 (Days)<br>Median (95% CI)<br>P value [3] | X X X X X X X X X X X X X X X X X X X | X X (X X X X X X X X X X X X X X X X X |
| Cox Proportional Hazards Model [4]<br>Hazard Ratio<br>(95% Wald CI for Hazard Ratio) | XXXX<br>(X.XXX, XXXX) | |

## Repeat for "Time to Achieve PSSI-75 (Days) [5]" and "Time to Achieve PSSI-90 (Days) [6]"

Abbreviations: CI = confidence interval; NE = not estimable; PSSI = Psoriasis Scalp Severity Index; SD = standard deviation.

Note: Subjects are summarized by planned treatment. Censored values are not included in the descriptive statistics. Only subjects who achieved PSSI-50, PSSI-75, or PSSI-90 are included in the relevant descriptive statistics. [1] PSSI-50 is achievement of 50% reduction in PSSI from baseline. Time to PSSI-50 is calculated as date of PSSI-50

achievement - Day 1 date + 1.

[2] Subjects who did not achieve PSSI-50, PSSI-75, or PSSI-90 were censored at day of discontinuation or date lost to follow-úp, whichever is earlier.

[3] P value was obtained from the log rank test where roflumilast foam 0.3% was compared to vehicle. [4] The hazard ratio and 95% Wald CI are obtained from a Cox Proportional Hazards model with country, baseline S-IGA score category, and baseline B-IGA score category as factors in the model, comparing roflumilast foam 0.3% to vehicle. [5] PSSI-75 is achievement of 75% reduction in PSSI from baseline. Time to PSSI-75 is calculated as date of PSSI-75

[6] PSSI-90 is achievement of 90% reduction in PSSI from baseline. Time to PSSI-90 is calculated as date of PSSI-90 achievement - Day 1 date + 1.

achievement - Day 1 date + 1. Reference Listing: 16.2.6.3



**premier** research

Table 14.2.3.6 Time to Achievement of PSSI-50, PSSI-75, and PSSI-90 mITT Population

(Programming note: Same as table 14.2.3.6.)

premier



| Study Visit<br>Category<br>Statistic [1] | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
|---|---|---|
| Week 2 | | |
| Change from Baseline | | |
| u | × | × |
| LS Mean Change from Baseline (SE) | X.XX (X.XXX) | X.XX (X.XXX) |
| (95% CI for LS Mean Change from Baseline) | (X.XX, X.XX) | (X.XX, X.XX) |
| P value for LS Mean Change from Baseline) [2] | X.XXXX | |
| LS Mean Difference from Vehicle (SE)<br>(95% Cl for Difference from Vehicle)<br>P value for Difference from Vehicle [3] | (XXX, XXX)<br>XXX (XXXX)<br>XXXXX | |

Continue for Percent Change from Baseline. Repeat for Week 4, Week 8, Week 9.

Abbreviations: ANCOVA = analysis of covariance; B-IGA = body investigator global assessment; CI = confidence interval; LS = least-squares;

scalp affected. The score ranges from 0 to 72. Erythema, induration, and desquamation are scored on a scale of 0 to 4, where 0 = absent and 4 = PSSI = Psoriasis Scalp Severity Index; S-IGA = scalp investigator global assessment; SE = standard error.

Note: Subjects are summarized by planned treatment. PSSI total score is calculated as (erythema score + induration + desquamation) × extent of missing measurement taken before the first application of study drug. Percent change from baseline is calculated as (result – baseline result)\*100. [1] Estimates for LS means (change/percent change from baseline and difference from vehicle [i.e., change/percent change from baseline for roflumilast foam 0.3% minus change from baseline for vehicle]) and accompanying 95% Cls, and P values are from an ANCOVA with country, baseline B-IGA score category, baseline B-IGA score category, and baseline PSSI score as independent variables. Baseline is the last nonseverest possible; extent of scale affected is scored on a scale of 0 to 6, where 0 = 0% of involved area and 6 = 90-100% of involved area.

[2] P value for testing change/percent change from baseline is zero. [3] P value for testing difference (roflumilast foam 0.3% minus vehicle) in change/percent change from baseline from is zero. Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.5

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101 Table 14.2.3.8
Summary of PSSI Scores by Study Visit – ANCOVA
mITT Population

**premier** research

(Programming note: Same as table 14.2.3.7.)

Summary and Change from Baseline in Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit ITT Population Table 14.2.4.1

(Programming note: Same as table 14.2.3.1. Update abbreviation row to display "SI-NRS = Scalp Itch – Numeric Rating Scale". Change reference listing to Reference Listing: 16.2.6.4. Update the footnotes as "Note: Subjects are summarized by planned treatment. The SI-NRS will be determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10, which ranges from "no scalp itch" to "worst scalp itch imaginable". Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result – baseline result. Percent change from baseline is calculated as (change from baseline/baseline)\*100.")

Summary and Change from Baseline in Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit mITT Population Table 14.2.4.2

(Programming note: Same as table 14.2.4.1.)



Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score Success by Study Visit ITT Population, Subjects with SI-NRS Pruritus Score ≥4 at Baseline (SPRU4-ITT Population) Table 14.2.4.3

| Study Visit/ | Roflumilast Foam 0.3% | Vehicle |
|---|---|---|
| Category/Statistic | (N=XX) | (N=XX) |
| Week 2 | × | × |
| SI-NRS Success [1] | | |
| Yes | XX (XX.X%) | XX (XX.X%) |
| 95% CI [2] | (X.XX, X.XX) | (x.xx, x.xx) |
| ON | XX (XX.X%) | XX (XX X%) |
| Odds Ratio (95% CI) [3]<br>P value [3] | X.XX (X.XX, X.XX)<br>X.XXXX | |

## Repeat for all Week 4, Week 8, and Week 9.

Abbreviations: B-IGA = body investigator global assessment; CI = confidence interval; S-IGA = scalp investigator global assessment; SI-NRS = Scalp Itch – Numeric Rating Scale.

Note: Percentages are n/Number of subjects in the SPRU4-ITT population within planned treatment at each visit\*100. Baseline is the last non-missing measurement taken on or before the day first application of study drug.

[1] SI-NRS success ("Yes") is defined as an achievement of a ≥4-point improvement from baseline score of ≥4; "No" otherwise. [2] 95% Cls for "Yes" are obtained using Wilson method. [3] The odds ratio, 95% Cl, and P value are obtained from Cochran Mantel Haenszel test (stratified by country, baseline S-IGA score category) comparing roflumilast foam 0.3% to vehicle. Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.4



Table 14.2.4.4

Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score Success by Study Visit mITT Population, Subjects with SI-NRS Pruritus Score ≥4 at Baseline (SPRU4-mITT Population)

(Programming note: Same as table 14.2.4.3. Change "Note: Percentages are n/Number of subjects in the SPRU4-mITT population within planned treatment at each visit\*100.")

Table 14.2.4.5
Summary of Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit – ANCOVA ITT Population

Numeric Rating Scale" Change reference listing to Reference Listings: 16.2.6.1, 16.2.6.4. Update the Note as "Note: Subjects are summarized by planned treatment. The SI-NRS will be determined by asking the subject's assessment of worst itch of scalp over the past 24 hours. The scale is from 0 to 10, which ranges from "no scalp itch" to "worst scalp itch imaginable". Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Percent change from baseline is calculated as (result – (Programming note: Same as table 14.2.3.7. Update [1] as to use "SI-NRS score" instead of "PSSI score". Update abbreviation row to display "SI-NRS = Scalp ltch – baseline result)\*100.")

Table 14.2.4.6 Summary of Scalp Itch – Numeric Rating Scale (SI-NRS) Pruritus Score by Study Visit – ANCOVA mITT Population

(Programming note: Same as table 14.2.4.5.)

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



Summary and Change from Baseline in Psoriasis Symptom Diary (PSD) Total and Individual Item Scores by Study Visit ITT Population

(Programming note: Same as table 14.2.3.1, except add header rows at the top for

"Item: Total Score"

"Item: How severe was your psoriasis-related itching?",
"Item: How bothered were you by your psoriasis-related itching?",
"Item: How severe was your psoriasis-related stinging?",
"Item: How bothered were you by your psoriasis-related stinging?",
"Item: How severe was your psoriasis-related burning?",

"Item: How bothered were you by your psoriasis-related burning?",
"Item: How severe was your psoriasis-affected skin cracking?",
form: How bothered were you by your psoriasis-affected skin cracking?"

"Item: How bothered were you by your psoriasis-affected skin cracking?",
 "Item: How severe was your psoriasis-related pain?",
 "Item: How bothered were you by your psoriasis-related pain?",
 "Item: How severe was your psoriasis scaling?",

"Item: How bothered were you by your psoriasis scaling?",
"Item: How noticeable did you think the color of your psoriasis-affected skin was?",
"Item: How much did you try to hide your psoriasis affected skin?",
"Item: How much did your psoriasis cause you to avoid activities with other people?",

calculated as sum of the 16 questions (individual questions scored 0 to 10, where higher scores indicate more severe symptoms). The total score ranges from 0 to 160. If 1 or more items are missing, the total score was not calculated. Baseline is the last non-missing measurement taken on or before the day first application of study drug. Change from baseline is Change abbreviation from PSSI to PSD = Psoriasis Symptom Diary. Change reference listings to Reference Listing: 16.2.6.5. Update footnoteas "The PSD total score is calculated as result – baseline result. Percent change from baseline is calculated as (change from baseline/baseline)\*100.") "Item: How embarrassed were you because of your psoriasis?"





Table 14.2.5.2 Summary and Change from Baseline in Psoriasis Symptom Diary (PSD) Total and Individual Item Scores by Study Visit mITT Population

(Programming note: Same as table 14.2.5.1.)

Summary of Psoriasis Symptom Diary (PSD) Total Scores by Study Visit – ANCOVA ITT Population Table 14.2.5.3

(Programming note: Same as table 14.2.3.7. Update [1] as to use "PSD total score" instead of "PSSI score". Change abbreviation from PSSI to PSD = Psoriasis Symptom Diary. Change reference listings to Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.5. Update the Note as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken before the first application of study drug. PSD total score is calculated as sum of the 16 questions (individual questions scored 0 to 10, where higher scores indicate more severe symptoms). The score ranges from 0 to 160. If 1 or more items are missing, the score is not calculated.")






Table 14.2.5.4
Summary of Psoriasis Symptom Diary (PSD) Total Scores by Study Visit – ANCOVA mITT Population

(Programming note: Same as table 14.2.5.3.)

Table 14.2.6.1 Summary and Change from Baseline in PASI/mPASI by Study Visit ITT Population

Index" and "mPASI = modified PASI" in alphabetical order. Change reference listing to Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.6. Update [1] as "PASI is calculated as (0.1×[Eh + Th + Sh]×Ah) + (0.2×[Et + Tt + St]×At) + (0.4×[El + Tl + Sl]×Ah), where E, T, and S are erythema, thickness, and scaling, respectively, scored on a scale of 0 to 6, and h, e, t, and I are head, arms, trunk, and legs respectively. The total score ranges from 0 to 72. (Programming note: Same as table 14.2.3.1, except add header rows at the top for "Scale: PASI" or "Scale: mPASI". Add Abbreviations "PASI = Psoriasis Area Severity mPASI is calculated similar to PASI except that for subjects with < 10% of any particular involved anatomic area, the mPASI will be calculated using the actual percentage of the anatomical area involved rather than the 0 to 6 estimated area score (e.g., 0.1 for 1%, 0.2 for 2%, 0.3 for 3%, ... 0.9 for 9%). Lower scores indicate improvement. Change from baseline is calculated as result – baseline result. Percent change from baseline is calculated as result – baseline result.

Table 14.2.6.2 Summary and Change from Baseline in PASI/mPASI by Study Visit mITT Population

(Programming note: Same as table 14.2.6.1)



Table 14.2.6.3
Summary of PASI/mPASI by Study Visit – ANCOVA
ITT Population

following to Abbreviations "PASI = Psoriasis Area Severity Index" and "mPASI = modified Psoriasis Area Severity Index" in alphabetical order. Change reference listings to Abbreviations "PASI = Psoriasis Area Severity Index" in alphabetical order. Change reference listings to Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.6. Replace PSD Total Score text in the note footnote with "PASI is calculated as (0.1x[E<sub>n</sub> + T<sub>n</sub> + S<sub>n</sub>]xA<sub>n</sub>) + (0.2x[E<sub>a</sub> + T<sub>a</sub> + S<sub>a</sub>]xA<sub>a</sub>) + graded on a scale of 0 to 6, and h, e, t, and I are head, arms, trunk, and legs respectively. The total score ranges from 0 to 72. mPASI is calculated similar to PASI except that for subjects with < 10% of any particular involved anatomic area, the mPASI will be calculated using the actual percentage of the anatomical area involved rather than the 0 to 6 estimated area score (e.g., 0.1 for 1%, 0.2 for 2%, 0.3 for 3%, ..., 0.9 for 9%). Lower scores indicate improvement.") (Programming note: Same as table 14.2.5.3, except add header rows at the top for "Scale: PASI" or "Scale: mPASI". Replace instances of PSD with PASI/mPASI. Add the (0.3×[E<sub>1</sub> + T<sub>1</sub> + S<sub>1</sub>]×A<sub>1</sub>) + (0.4×[E<sub>1</sub> + T<sub>1</sub> + S<sub>1</sub>]×A<sub>2</sub>), where E, T, and S are erythema, thickness, and scaling, respectively, scored on a scale of 0 to 4, A is estimated area of skin involved,

Table 14.2.6.4 Summary of PASI/mPASI by Study Visit – ANCOVA mITT Population (Programming note: Same as table 14.2.6.3.)

Table 14.2.6.5 Summary of Achievement of PASI-50, PASI-75, and PASI-90 by Study Visit ITT Population

| Study Visit<br>Category/Statistic | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) |
|---|---|---|
| Week 2 | × | × |
| Yes<br>Yes<br>95% CI [4] | XX (XX.X%)<br>(X.X, X.XX) | XX (XX.X%) |
| No | XX (XX.X%) | (%X:X%) |
| Odds Ratio (95% CI) [5]<br>P value [5] | X.XX (X.XX, X.XX)<br>X.XXXX | |
| PASI-75 [2]<br>Yes<br>95% CI [4]<br>No | XX (XX.X%)<br>(X.XX, X.XX)<br>XX (XX.X%) | XX (XX.X%)<br>(X.XX, X.XX)<br>XX (XX.X%) |
| Odds Ratio (95% CI) [5]<br>P value [5] | X.XX (X.XX, X.XX)<br>X.XXXX | X.XX (X.XX, X.XX) |
| PASI-90 [3]<br>Yes<br>95% CI [4]<br>No | XX (XX.X%)<br>(X.XX, X.XX)<br>XX (XX.X%) | XX (XX.X%)<br>(X.XX, X.XX)<br>XX (XX.X%) |
| Odds Ratio (95% CI) [5]<br>P value [5] | X.XX (X.XX, X.XX)<br>X.XXXX | X.XX (X.XX, X.XX) |

Repeat for Week 4, Week 8, and Week 9.

Abbreviations: B-IGA = body investigator global assessment; CI = confidence interval; S-IGA = scalp investigator global assessment; PASI = Psoriasis Area Severity Index.

Note: Percentages are n/Number of subjects in the ITT population within planned treatment at each visit\*100. Baseline is the last non-missing measurement taken before the first application of study drug.

Institute and baseline; "No" otherwise.

[2] PASI-56 is populated with "Yes" when there is an achievement of a 50% reduction in PASI total score from baseline; "No" otherwise.

[3] PASI-56 is populated with "Yes" when there is an achievement of a 75% reduction in PASI total score from baseline; "No" otherwise.

[3] PASI-90 is populated with "Yes" when there is an achievement of a 90% reduction in PASI total score from baseline; "No" otherwise.

[4] 95% Cls for "Yes" are obtained using Wilson method.

[5] The odds ratio, 95% Cl, and P value are obtained from Cochran Mantel Haenszel test (stratified by country, baseline S-IGA score category) comparing roflumilast foam 0.3% to vehicle.

Reference Listings: 16.2.6.1, 16.2.6.6



Table 14.2.6.6 Summary of Achievement of PASI-50, PASI-75, and PASI-90 by Study Visit mITT Population

(Programming note: Same as table 14.2.6.5)

Time to Achievement of PASI-50 ITT Population Table 14.2.6.7

(Programming note: Same as table 14.2.3.5. Replace instances of PSSI-50 with PASI-50 and update the abbreviations accordingly. Change the reference listings to 16.2.6.1, 16.2.6.5, 16.2.6.6)

Time to Achievement of PASI-50 mITT Population Table 14.2.6.8

(Programming note: Same as table 14.2.3.5. Replace instances of PSSI-50 with PASI-50 and update the abbreviations accordingly. Change the reference listings to 16.2.6.1, 16.2.6.5, 16.2.6.6)

Table 14.2.6.9 Summary of Achievement of mPASI-50, mPASI-75, and mPASI-90 by Study Visit ITT Population

(Same shell as Table 14.2.6.5; change all instances of PASI to mPASI)

Table 14.2.6.10 Summary of Achievement of mPASI-50, mPASI-75, and mPASI-90 by Study Visit mITT Population

(Same shell as Table 14.2.6.5; change all instances of PASI to mPASI)




Table 14.2.7.1 Summary and Change from Baseline in Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit ITT Population (Programming note: Same as table 14.2.3.1. Change reference listing to Reference Listing: 16.2.6.7. Update abbreviation row to display "WI-NRS = Worst Itch – Numeric Rating Scale". Update footnote as follows: "Note: Subjects are summarized by planned treatment. The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch". Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result — baseline result. Percent change from baseline is calculated as (change from baseline)\*100.")

Table 14.2.7.2 Summary and Change from Baseline in Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit mITT Population

(Programming note: Same as table 14.2.7.1)

Table 14.2.7.3
Summary of Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit – ANCOVA ITT Population

Update abbreviation row to display "WI-NRS = Worst Itch - Numeric Rating Scale". Update the baseline definition to read, "Baseline is the last non-missing measurement (Programming note: Same as table 14.2.3.7; Replace instances of PSD with WI-NRS in [1]. Change reference listings to Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.7. taken on or before the day first application of study drug." Replace PSD Total Score text in the note footnote with "The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from 0 to 10, which ranges from "no itch" to "worst imaginable itch". Lower scores indicate improvement.")

Table 14.2.7.4
Summary of Worst Itch – Numeric Rating Scale (WI-NRS) by Study Visit – ANCOVA mITT Population

(Programming note: Same as table 14.2.7.3)



Table 14.2.7.5

Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit
ITT Population, Subjects with WI-NRS Pruritus Score ≥4 at Baseline (PRU4-ITT Population)

(Programming note: Same as table 14.2.4.3, except replace all instances of SI-NRS with WI-NRS. Update abbreviation row to display "WI-NRS = Worst Itch – Numeric Rating Scale". Change reference listings to Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.7.)

Table 14.2.7.6
Worst Itch – Numeric Rating Scale (WI-NRS) Pruritus Score Success by Study Visit mITT Population, Subjects with WI-NRS Pruritus Score ≥4 at Baseline (PRU4-mITT Population)

(Programming note: Same as table 14.2.7.5.)



Summary and Change from Baseline in Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit Table 14.2.8.1 ITT Population

summarized by planned treatment. The DLQI/CDLQI score is calculated as sum of all the 10 questions at each visit and ranges between 0-30. The individual questions are scored as (Programming note: Same as table 14.2.3.1, except add header rows at the top for "Scale: DLQ!" and "Scale: "CDLQ!". Add "DLQ! = Dermatology Life Quality Index" and "CDLQ! = Children's DLQ!" to abbreviations in alphabetical order. Change reference listing to Reference Listing: 16.2.6.8. Update footnotes as "Note: Subjects are "Very much" or "Yes"= 3, "A lot" = 2, "A Little" = 1, "Not at all" or "Not Relevant" = 0. If 1 item is missing, it is scored as 0 for that item. If 2 or more items are missing, the score should not be calculated. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as result – baseline result. Percent change from baseline is calculated as (change from baseline)\*100.")

Table 14.2.8.2 Summary and Change from Baseline in Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit mITT Population

(Programming note: Same as table 14.2.8.1)

Table 14.2.8.3 Summary of Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit – ANCOVA ITT Population

item. If 2 or more items are missing, the score should not be calculated. Lower scores indicate improvement. Baseline is the last non-missing measurement taken on or before the day first application of study drug. Change from baseline is calculated as result – baseline result. Percent change from baseline is calculated as (change from baseline)\*100.") 0-30. The individual questions are scored as "Very much" or "Yes" = 3, "A lot" = 2, "A Little" = 1, "Not at all" or "Not Relevant" = 0. If 1 item is missing, it is scored as 0 for that Programming note: Same as table 14.2.3.7, except add header rows at the top for "Scale: DLQ!" and "Scale: "CDLQ!". Add "DLQ! = Dermatology Life Quality Index" and "CDLQI = Children's DLQI" to abbreviations in alphabetical order. Change reference listings to Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.8. Replace instances of PSD with DLQI/CDLQI score is calculated as sum of all the 10 questions at each visit and ranges

Table 14.2.8.4
Summary of Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI) by Study Visit – ANCOVA mITT Population

(Programming note: Same as table 14.2.8.4)



Table 14.2.9.1 Summary and Change from Baseline in % Body Surface Area (BSA) Affected by Disease by Study Visit ITT Population (Programming note: Same as table 14.2.3.1. Add "BSA = body surface area" to abbreviations in alphabetical order. Change reference listing to Reference Listing: 16.2.6.9. Update footnotes as "Note: Subjects are summarized by planned treatment. Baseline is the last non-missing measurement taken before the first application of study drug. Change from baseline is calculated as result – baseline result. Percent change from baseline is calculated as (change from baseline/baseline)\*100.")

Table 14.2.9.2
Summary and Change from Baseline in % Body Surface Area (BSA) Affected by Disease by Study Visit
mITT Population

(Programming note: Same as table 14.2.9.2)

Table 14.2.9.3 Summary of % Body Surface Area (BSA) Affected by Disease by Study Visit – ANCOVA ITT Population (Programming note: Same as table 14.2.3.7. Add "BSA = body surface area" and "ePRO = electronic patient reported outcomes" to abbreviations in alphabetical order. Change reference listings to Reference Listings: 16.2.6.1, 16.2.6.2, 16.2.6.9. Replace instances of PSD with BSA in [1]. Replace PSD Total Score text in the note footnote with "BSA collected on the ePRO tablet will be used for summarization.")

Table 14.2.9.4
Summary of % Body Surface Area (BSA) Affected by Disease by Study Visit – ANCOVA mITT Population

(Programming note: Same as table 14.2.9.3)





Table 14.3.1.1 Summary of Treatment Emergent Adverse Events Safety Population

| Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Maximum Severity of TEAE [1]<br>Grade 1 (Mild) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Grade 2 (Moderate) | XX (XX. X%) | XX (XX: X%) | XX (XX:X%) |
| Grade 3 (Severe)<br>Grade 4 (Life-threatening consequences) | (%X:XX)<br>XX (XX:X%) | (%X:XX)<br>XX (XX:X%) | (%X:XX)<br>XX (XX:X%) |
| Grade 5 (Death related to AE) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a Related TEAE [2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a TEAE Leading to Discontinuation of Study Drug | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with an SAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a Grade 5 TEAE [3] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event, CTCAE = Common Terminology Criteria for Adverse Events; IP = investigational product; SAE = serious adverse event; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety population within treatment received\*100. A TEAE is defined as an AE that started post

application of IP at the baseline visit through study completion.
[1] Severity grades are reported according to the CTCAE version 4.0. Subjects are counted only once at the worst severity. If a severity designation is

missing, it will be considered as severe.
[2] AEs with a relationship of possibly, probably, likely, or missing were considered related.
[3] A Grade 5 TEAE is a TEAE leading to death.
Reference Listing: 16.2.7.1



Table 14.3.1.2 Incidence of Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| System Organ Class | Roflumilast Foam 0.3% | Vehicle | Overall (N=XX) |
|---|---|---|---|
| Preferred Term | (N=XX) | (N=XX) | |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX. X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX. X%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 Preferred Term 3 | XX (XX: X%) | XX (XX.X%) | (%XXX) |
| | XX (XX: X%) | XX (XX.X%) | XX (XXXX) |
| | XX (XX: X%) | XX (XX.X%) | XX (XXXX) |
| | XX (XX: X%) | XX (XX.X%) | XX (XXXX) |

Abbreviations: AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. AEs were coded using MedDRA version 23.0. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT). AEs are displayed alphabetically by SOC, then by descending frequency of PT within SOC, and then alphabetically by PT.

Programming note: SOC & PT text should be presented as is from the dataset.

Table 14.3.1.3 Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Safety Population

**premier** research

| System Organ Class<br>Preferred Term<br>Maximum Severity [1] | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with at least 1 TEAE Grade 1 (Mild) Grade 2 (Moderate) Grade 3 (Severe) Grade 4 (Life-threatening consequences) Grade 5 (Death related to AE) | XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%) | (%X.XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX) | (%X.XX)<br>(%X.XX)<br>(%X.XX)<br>(XX.XX)<br>(XX.XX |
| System Organ Class 1 Any Event (Total) Grade 1 (Mild) Grade 2 (Moderate) Grade 3 (Severe) Grade 4 (Life-threatening consequences) Grade 5 (Death related to AE) | XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%)<br>XX (XX. X%) | (%X XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX)<br>(XX) | (%X:XX)<br>(%X:XX)<br>(%X:XX)<br>(X:XX) |
| Preferred Term 1 Grade 1 (Mild) Grade 2 (Moderate) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |

Abbreviations: AE = adverse event; CTCAE = Common Terminology Criteria for Adverse Events; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. AEs were coded using MedDRA

once for each system organ class (SOC) and once for each preferred term (PT) at the maximum severity.

[1] Severity grades are reported according to the CTCAE version 4.0. The severity shown is the greatest severity reported for a particular subject (Grade 5 [Death related to AE] > Grade 4 [Life-threatening consequences] > Grade 3 [Severe] > Grade 2 [Moderate] > Grade 1 [Mild]). AEs with a missing severity were counted as Severe. AEs are displayed alphabetically by SOC, then by descending frequency of PT within SOC, and then version 23.0. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion. Subjects are counted

alphabetically by PT.

Reference Listing: 16.2.7.1

Programming note: SOC & PT text should be presented as is from the dataset.

**premier** research Table 14.3.1.4 Incidence of Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug

Safety Population

| System Organ Class<br>Preferred Term<br>Relationship [1] | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Subjects with at least 1 TEAE<br>Related<br>Not Related | (%X.XX)<br>XX (XX.XX)<br>XX (XX.XX) | (%XXX)<br>XX (XXXX)<br>XX (XXXXX) | (%X:XX)<br>XX (XX:XX)<br>XX (XX:XX) |
| System Organ Class 1<br>Related<br>Not Related | (%XXX)<br>(XXX) | (%X:XX)<br>XX (XX:X%)<br>XX (XX:X%) | ( |
| Preferred Term 1<br>Related<br>Not Related | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |

Abbreviations: AE = adverse event; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. AEs were coded using Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT) at the greatest relationship category. The relationship shown is the greatest relationship reported for a particular subject (Related > Not Related). AEs with a missing relationship were counted as Related. AEs are displayed alphabetically by SOC, then by descending frequency of PT within SOC, and then alphabetically by PT. MedDRA version 23.0. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion.

[1] Related = Probably Related, Possibly Related, Likely Related, and Missing; Not Related = Unrelated and Unlikely Related. Reference Listing: 16.2.7.1

**Programming note:** SOC & PT text should be presented as is from the dataset.

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101

Table 14.3.1.5 Incidence of Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term Safety Population

**premier** research

(Same shell as Table 14.3.1.2)

Table 14.3.1.6 Incidence of Treatment Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term Safety Population

(Same shell as Table 14.3.1.2)



**premier** research

| | Roflumilast Foam 0.3% | Vehicle | Overall |
|---|---|---|---|
| Preferred Term | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 Related TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | XX (XX.X%) | (%X:X%) XX | (%X:X%) |
| Preferred Term 1 | XX (XX.X%) | (%X:XX) XX | (%X:X%)<br>XX |
| Preferred Term 2 | XX (XX.X%) | (%X:XX) XX | (%X:X%) |
| Preferred Term 3 | XX (XX.X%) | (%X:XX) XX | (%X:X%)<br>XX |
| Preferred Term 4 | XX (XX.X%) | (%X:X%) | XX (XX.X%) |
| Preferred Term 5 | XX (XX.X%) | (%X:XX) XX | (%X:X%) |
| Preferred Term 6 | XX (XX.X%) | (%X:X%) | XX (XX.X%) |
| Preferred Term 7 | XX (XX.X%) | (%X:X%) XX | (%X:X%) |
| Preferred Term 8 | XX (XX.X%) | (%X:X%) XX | (%X:X%) |
| Preferred Term 9 | XX (XX.X%) | (%X:X%) XX | (%X:X%) |
| Preferred Term 10 | XX (XX.X%) | (%X:XX) XX | (%X:X%)<br>XX |
| Preferred Term 11 | (%X:X%) | (%X:XX) XX | (%X:X%) XX |
| : | | | |

Abbreviations: AE = adverse event; CTCAE = Common Terminology Criteria for Adverse Events; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. AEs were coded using MedDRA version 23.0. A TEAE is defined as an AE that started post application of IP at the baseline visit through study completion. Related TEAEs are AE marked Probably Related, Possibly Related, Likely Related, or missing. Subjects are counted once for each once for each preferred term (PT). AEs are displayed by descending frequency of PT, and then alphabetically by PT in case of ties.

Programming note: PT text should be presented as is from the dataset.



**premier** research

(Same shell as Table 14.3.1.2; first-row text is "Subjects with at least 1 SAE"; add SAE = serious adverse event)

Table 14.3.2.2 Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Relationship to Study Drug Safety Population

(Same shell as Table 14.3.1.4; first-row text is "Subjects with at least 1 SAE"; add SAE = serious adverse event)

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



Table 14.3.2.3 Incidence of Serious Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Safety Population

(Same shell as Table 14.3.1.3; first-row text is "Subjects with at least 1 SAE"; add SAE = serious adverse event)





Table 14.3.3.1 Listing of Adverse Events Leading to Study Drug Discontinuation Safety Population

| 5 | Subject Treatment<br>ID Received | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Outcome/ Start Date/Time (Study Day)/ CTCAE Toxicity Grade/ Study Drug Action Taken/ End Date/Time (Study Day) Relationship Other Action Taken | CTCAE Toxicity Grade<br>Relationship | Outcome/<br>/ Study Drug Action Taken/<br>Other Action Taken | Serious?/<br>Criteria Met |
|---|---|---|---|---|---|---|
| XXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/hh:mm (X)/<br>DDMONYYYY/hh:mm (X) | XXXXXXXXXX | XXXXXXXXX<br>XXXXXXXXXXX | × |
| XXXX | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/hh:mm (X)/<br>DDMONYYYY/hh:mm (X) | XXXXXXXXXX | /XXXXXXXXX<br>/XXXXXXXXXXX | × |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY/hh:mm (X)/<br>DDMONYYYY/hh:mm (X) | XXXXXXXXX | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXX |

Note: Study day is calculated relative to the date of first application of study drug. AEs were coded using MedDRA version 23.0. Severity grades are reported according to the CTCAE Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; MedDRA = Medical Dictionary for Regulatory Activities.

Programming note: If time missing, display "--;--'." (Other Action Taken" will be either None, Concomitant Medication, Non-drug Therapy, Hospitalization or Prolongation of Hospitalization, Discontinued Study or Other; if specify text is needed, concatenate "Concomitant Medication:" or "Other:" with the text. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported." SOC & PT text should presented as is from the dataset. version 4.0.




Table 14.3.3.2 Listing of Serious Adverse Events Safety Population

(Same shell as Table 14.3.3.1)

Table 14.3.3.3 Listing of Deaths Safety Population

(Same shell as Table 14.3.3.1)



Table 14.3.5.1.1 Summary of Clinical Chemistry Laboratory Results by Study Visit Safety Population

Parameter: XXXXXXX (unit)

| | Roflumilast | last Foam 0.3% | Vehicle | je<br>je | Overall | rall |
|---|---|---|---|---|---|---|
| Study Visit | XX=N) | (X | XX=N) | $\widehat{x}$ | (XX=N) | 8 |
| Statistic | Observed | Change | Observed | Change | Observed | Change |
| Baseline | | | | | | |
| )<br>:::<br>::: | × | | × | | × | |
| Mean (SD) | XX:X (XX:XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | |
| Median | ××× | | ××× | | ×:×× | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | |
| Week 4 | | | | | | |
| _ | × | × | × | × | × | × |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | ××× | ××× | ××× | ××× | ××× | ××× |
| Min, Max | ××× | ××× | ×××× | ××× | ×,× | ×,× |

Repeat for Week 8. Continue for other parameters. Sort alphabetically by parameter.

Note: Subjects are summarized by treatment received and overall. Baseline is the last non-missing measurement taken before the first application of study drug. Reference Listing: 16.2.8.1.1



Table 14.3.5.1.2 Shift from Baseline in Clinical Chemistry Laboratory Results by Study Visit Safety Population

Parameter: XXXXXXX (unit)

| | | | | | | paselli | baseline Grade | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Post- | | Rc | Roflumilast Foam 0.3% | .3% | | | | Vehicle | | |
| | Baseline | | | (N=XX) | | | | | (N=XX) | | |
| Study Visit | Grade | Missing | Low | Normal | High | Total | Missing | Low | Normal | High | Total |
| Week 4 | Missing | (%X:X%) | (%X:X%) | XX (XX:X%) | (%X:X%)<br>XX | (%X:X%) | (%X:X%) | (%X:X%) | (%X:X%) | (%X:X%) | (%X:X%) XX |
| | Low | (%X.XX) XX | (%X:X%) XX | (%X:X%) XX | (%X:X%) XX | XX (XX:X%) | (%X:X%) XX | XX (XX:X%) | (%X:X%) | (%X:X%) XX | (%X:XX) XX |
| | Normal | (XX.XX) | (%X:X%) XX | (%X:XX) XX | XX (XX.X%) | XX (XX.X%) | (%X:X%) | XX (XX.X%) | (%X:X%) | (%X:X%) XX | (%X:XX) XX |
| | High | XX (XX.X%) | XX (XX:X%) | (%X:X%) XX | XX (XX.X%) | XX (XX:X%) | (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Total | (%X:X%) | XX (XX.X%) | XX (XX.X%) | (%X:X%)<br>XX | (%X:X%) XX | (XX:X%) | (%X:X%) XX | (%X:X%) XX | (%X:X%) | (%X:X%) XX |
| Week 8 | Missing | XX (XX.X%) | XX (XX.X%) | (%X:X%) | XX (XX.X%) | XX (XX:X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Low | XX (XX:X%) | (XX:X%) | (%X:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Normal | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX | XX (XX.X%) | XX (XX:X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX: X%) | XX (XX.X%) |
| | High | (%X.XX) XX | (%X:X%) XX | (%X:X%) XX | (%X:X%) XX | XX (XX:X%) | (%X:X%) | XX (XX.X%) | (%X:X%) | (%X:X%) XX | (%X:XX) XX |
| | Total | (%X:X%) | (%X:X%) | (%X:X%) | (%X:X%) | XX (XX:X%) | (%X:X%) | XX (XX:X%) | (%X:X%) | (%X:X%) | (%X:XX) XX |

Repeat for Overall. Repeat all for clinical chemistry parameters (excluding serum HCG results).

Note: Percentages are n/Number of subjects in the Safety population within treatment received\*100. Baseline is the last non-missing measurement taken before the first application of study

drug. Reference Listing: 16.2.8.1.1



Table 14.3.5.2.1 Summary of Hematology Laboratory Results by Study Visit Safety Population

**premier** research

(Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.8.1.2)

Shift from Baseline in Hematology Laboratory Results by Study Visit Safety Population Table 14.3.5.2.2

(Same shell as Table 14.3.5.1.2; Reference Listing: 16.2.8.1.2)

Table 14.3.5.3.1 Summary of Quantitative Urinalysis Laboratory Results by Study Visit Safety Population

(Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.8.1.3)

Table 14.3.5.3.2 Shift from Baseline in Quantitative and Qualitative Urinalysis Laboratory Results by Study Visit Safety Population

(Same shell as Table 14.3.5.1.2; Reference Listing: 16.2.8.1.3)



**premier** research

| Study Visit<br>Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX. X%) | (%X:X%)<br>(%X:X%) | XX (XX.X%) |
| XXXXXXXXX | XX (XX.X%) | XX (XX. X%) | XX (XX.X%) |
| Week 4 | | | |
| XXXXXXXX | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| XXXXXXXXXXXX | (%X:X%) | (%X:XX) XX | (%X:XX) |
| XXXXXXX | XX (XX: X%) | XX (XX.X%) | XX (XX.X%) |
| Week 8 | | | |
| XXXXXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXXXXXXXXX | (%X:X%) | XX (XX.X%) | (%X:X%) |
| XXXXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken before the first application of study drug.

Reference Listing: 16.2.8.1.3



Table 14.3.6.1 Shift from Baseline in Patient Health Questionnaire (PHQ-8)/Modified PHQ-Adolescents by Study Visit Safety Population

Scale: PHQ-8

| | | | | Baseline Category | | | |
|---|---|---|---|---|---|---|---|
| | | | Roflu | Roflumilast Foam 0.3% (N=XX) | =XX) | | |
| Study Visit | | | | | Moderately | | |
| Category [1] | Missing | None | Mild | Moderate | Severe | Severe | Total |
| Week 4 | | | | | | | |
| Missing | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | XX (XX: X%) | XX (XX.X%) | (%X:X%) |
| None | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | (%X:XX) XX |
| Mild | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | (%X:X%) XX |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) |
| Moderately Severe | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:X%) XX | XX (XX: X%) | XX (XX.X%) | XX (XX.X%) |
| Total | (%X:XX) XX | XX (XX.X%) | (%X XX) XX | (%X:XX) XX | XX (XX X%) | (%X:X%) | XX (XX.X%) |
| Week 8 | | | | | | | |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| None | (%X:XX) XX | XX (XX.X%) | (%X:XX) XX | (%X:X%) XX | (XX:X%) | (%X:X%) | XX (XX X%) |
| Mild | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) | (%X:X%) XX | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | (%X:XX) XX | XX (XX.X%) | (%X:XX) XX | (%X:X%) XX | (XX:X%) | (%X:X%) | XX (XX X%) |
| Moderately Severe | (%X:XX) | (%X:XX) XX | (%X:XX) XX | (%X:X%) XX | (XX:X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | (%X:XX) | (%X:XX) XX | (%X.XX) XX | (%X:XX) XX | (XX:X%) | (%X:X%) | (%X:XX) XX |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Repeat for Vehicle and Overall. Repeat for Scale: PHQ-A

Abbreviations: PHQ-8 = patient health questionnaire (8 questions); PHQ-A = patient health questionnaire - adolescents.

Note: Percentages are n/Number of subjects in the Safety population within scale (PHQ-A) and treatment received and overall\*100. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. The PHQ total score is calculated as sum of the 8 questions (individual questions scored as Not at all=0, Several days=1, More than half the days=2, and Nearly every day=3). The total score ranges from 0 to 24. If more than 1 item is missing the score was not calculated. If 1 item is missing the score is calculated as (sum of answered items\*8)/number of answered items. The PHQ-8 was filled out by adults and the modified PHQ-A was filled out

[i] If the total score ranges from 0 to 4, it is classified as None – Minimal Depression; 5 – 9 classified as Mild; 10 – 14 classified as Moderate; 15-19 classified as Moderately Severe; 20 – 24 classified as Severe Depression.
Reference Listing: 16.2.9.7 by adolescents.



(Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.9.1; Repeat for Week 8; Add this line at the end in note footnote – "Lower scores indicate no evidence of irritation while higher scores indicate worsening reaction. These assessments should be done prior to the IP application in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary.")

Table 14.3.6.2.2 Summary of Investigator Local Tolerability Assessment (Dermal Response) by Study Visit

| Categorical Results | Safety Population |
|---------------------|-------------------|
| ) | |
| • | |

| Study Visit<br>Category | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline | | | |
| 0 = No evidence of irritation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 1 = Minimal erythema | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 = Definite erythema | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| 3 = Erythema and papules | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| 4 = Definite edema | (%X:XX) | (%X:X%) XX | (%X:XX) XX |
| 5 = Erythema, edema and papules | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| 6 = Vesicular eruption | XX (XX.X%) | XX (XX.X%) | (%X:X%)<br>XX |
| 7 = Strong reaction spreading beyond application site | | | |
| Week 4 | | | |
| 0 = No evidence of irritation | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| 1 = Minimal erythema | (%X:XX) XX | (%X.XX) XX | (%X:XX) XX |
| 2 = Definite erythema | (%X:XX) | (%X:X%) XX | (%X:XX) XX |
| 3 = Erythema and papules | (%X:XX) XX | XX (XX.X%) | (%X:XX) XX |
| 4 = Definite edema | (%X:XX) XX | (%X:X%) XX | (%X:X%)<br>XX |
| 5 = Erythema, edema and papules | (%X:XX) XX | XX (XX:X%) | (%X:X%) |
| 6 = Vesicular eruption | (%X:XX) XX | (%X:X%) XX | (%X:XX) XX |
| 7 = Strong reaction spreading beyond application site | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

#### Repeat for Week 8

Abbreviation: IP = investigational product.

Note: Percentages are n/Number of subjects in the Safety Population within treatment received and overall\*100. Baseline is the last non-missing measurement taken before the first application of study drug. These assessments should be done prior to the IP application in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary. Reference Listing: 16.2.9.1



Table 14.3.6.2.3 Summary of Investigator Local Tolerability Assessment (Other Effects) by Study Visit Categorical Results Safety Population

| Study Visit<br>Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline | | | |
| A = Slight glazed appearance | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) |
| B = Marked glazing | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| C = Glazing with peeling and cracking | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX |
| D = Glazing with fissures | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| E = Film of dried serous exudates | XX (XX.X%) | (%X:XX) XX | (%X:XX) |
| F = Small petechial erosions and/or scabs | XX (XX.X%) | XX (XX.X%) | (%X:XX) XX |
| G = No other effects | (%X:X%) | XX (XX.X%) | XX (XX.X%) |
| Week 4 | | | |
| A = Slight glazed appearance | XX (XX.X%) | (%X:XX) XX | (%X:X%) |
| B = Marked glazing | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX |
| C = Glazing with peeling and cracking | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX |
| D = Glazing with fissures | (%X:X%) | (%X:XX) XX | (%X:XX) XX |
| E = Film of dried serous exudates | (%X:X%) | (%X:XX) XX | (%X:XX) XX |
| F = Small petechial erosions and/or scabs | (%X:X%) | (%X:XX) XX | (%X:XX) XX |
| G = No other effects | (%X:X%) XX | XX (XX.X%) | XX (XX.X%) |

#### Repeat for Week 8

Abbreviation: IP = investigational product.

Note: Percentages are n/Number of subjects in the Safety Population within treatment received and overall\*100. Baseline is the last non-missing measurement taken before the first application of study drug. These assessments should be done 10 - 15 minutes after the application of IP in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table

summary. Reference Listing: 16.2.9.1



### Table 14.3.6.3.1 Summary of Subject Local Tolerability Assessment by Study Visit Safety Population

(Same shell as Table 14.3.5.1.1; Reference Listing: 16.2.9.2; Repeat for Week 4, Week 8; add "IP = investigational product" to abbreviations; Add this line at the end in note footnote – "Lower scores indicate no sensation while higher scores indicate worsening/severe sensation. These assessments should be done 10 - 15 minutes after the application of IP in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary." Change baseline definition to "Baseline for subject local tolerability assessment is the last non-missing measurement taken on the day of first application of study drug.")

Table 14.3.6.3.2 Summary of Subject Local Tolerability Assessment by Study Visit Categorical Results Safety Population

**premier** research

| Study Visit<br>Category | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Baseline<br>0 = None (no sensation) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 1 = Mild (slight warm, tingling sensation) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 2 = Moderate (definite warm, tingling sensation) | (%X:XX) | XX (XX.X%) | XX (XX.X%) |
| 3 = Severe (hot, tingling/stinging sensation) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 4 | | | |
| 0 = None (no sensation) | (%X:XX) | (XX:X%) | (%X:X%)<br>XX |
| 1 = Mild (slight warm, tingling sensation) | XX (XX:X%) | XX (XX.X%) | (XX:X%) |
| 2 = Moderate (definite warm, tingling sensation) | (%X:XX) | XX (XX.X%) | (%X:X%) |
| 3 = Severe (hot, tingling/stinging sensation) | (%X:X%) | (%X.XX) XX | (%X.XX) XX |

#### Repeat for Week 8

Abbreviation: IP = investigational product.

Note: Percentages are n/Number of subjects in the Safety Population within treatment received and overall\*100. Baseline for subject local tolerability assessment is the last non-missing measurement taken on the day of first application of study drug. These assessments should be done 10 - 15 minutes after the application of IP in the study site. Subjects not meeting this condition on baseline visit are completely removed from the table summary. Reference Listing: 16.2.9.2





(Same shell as Table 14.3.5.1.1; visits include Baseline, Week 2, Week 8, Week 9; parameters include Temperature (°C), Heart Rate (bpm), Systolic Blood Pressure (mmHg), Height (cm), Weight (kg), and BMI (kg/m²) [11, where [1] goes to "[1] Body Mass Index (BMI) = weight (kg) / [height (m)]²."; Reference Listings: 16.2.9.3.1, 16.2.9.3.1)





Table 14.3.6.4.2 Shift from Baseline in Weight by Study Visit Safety Population

| Roflumilast Foam 0.3% Vehicle Overall (N=XX) (N=XX) | | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | | | XX (XX.X%) | (%X:X%) | XX (XX.X%) | XX (XX.X%) $XX (XX.X%)$ $XX (XX.X%)$ | | | XX (XX. X%) | XX (XX.X%) XX (XX.X%) XX (XX.X%) | (%X XX) XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit<br>Category | Week 2 | Weight Loss ≥ 10% | Weight Gain ≥ 10% | Weight Loss ≥ 5% | Weight Gain ≥ 5% | Week 4 | Weight Loss ≥ 10% | Weight Gain ≥ 10% | Weight Loss ≥ 5% | Weight Gain ≥ 5% | Week 8 | Weight Loss ≥ 10% | Weight Gain ≥ 10% | Weight Loss ≥ 5% | Weight Gain ≥ 5% |

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken before the first application of study drug.

Reference Listing: 16.2.9.3.2

Continue for Week 9



Table 14.3.6.4.3 Shift from Baseline in Weight by Study Visit and Weight Loss Intentional/Non-Intentional Categories Safety Population

(Same shell as Table 14.3.6.4.2, except will be presented by the following categories as headers in the by-line: "Weight Loss: Intentional" and "Weight Loss: Not Intentional or Missing").



Table 14.3.6.4.4 Shift from Baseline in BMI Categories by Study Visit Safety Population

| | | | | Baseline Category | Category | | |
|---|---|---|---|---|---|---|---|
| | Post-Baseline | | | Roflumilast Foam 0.3% (N=XX) | m 0.3% (N=XX) | | |
| Study Visit | Category [1] | Missing | Underweight | Normal | Overweight | Obese | Total |
| Week 2 | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Underweight | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Normal | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) | (XX.X%) | XX (XX:X%) |
| | Overweight | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Obese | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) | (%X:XX) XX | (XX.X%) | XX (XX.X%) |
| | Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 4 | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Underweight | (%X:X%) XX | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) | (%X.X%) XX | XX (XX.X%) |
| | Normal | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) | (%X:XX) XX | XX (XX.X%) | XX (XX.X%) |
| | Overweight | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X.X%) XX | XX (XX:X%) |
| | Obese | XX (XX.X%) | XX (XX.X%) | (XX.XX) | XX (XX.X%) | (XX.X%) | XX (XX.X%) |
| | Total | XX (XX.X%) | (XX:XX) | (%X.XX) XX | (%X:X%) | (%X.XX) XX | (%X:XX) XX |

# Repeat for Vehicle and Overall. Repeat all for Week 8.

Abbreviation: BMI = body mass index.

before the first application of study drug. BMI is derived as (weight in kg)/[(height in cm/100)²].

[1] If BMI is below 18.5 then it is categorized as underweight; if BMI ranges between 18.5 – 24.9 then it is categorized as overweight; if BMI is ≥ 30.0 then it is categorized as obese.

Reference Listings: 16.2.9.4.1, 16.2.9.4.2 Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken



Table 14.3.6.4.5 Shift from Baseline in Weight by Study Visit and Weight Loss Intentional/Non-Intentional Categories Safety Population

(Same shell as Table 14.3.6.4.5, except will be presented by the following categories as headers in the by-line: "Weight Loss: Intentional" and "Weight Loss: Not Intentional or Missing").



Table 14.3.6.5 Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation and Suicidal Behavior by Study Visit Safety Population

| Study Visit<br>C-SSRS Section<br>C-SSRS Item | Roflumilast Foam 0.3%<br>(N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Screening<br>Suicidal Ideation<br>Wish to be Dead | (%X.XX)<br>XX (XX.XX)<br>XX (XX.XX) | XX (XX. X%) | (%X XX) XX |
| Non-Specific Active Suicidal Thoughts Active Suicidal Ideation with Any Methods | (%X:X%)<br>XX (XX:X%)<br>XX (XX:X%) | (%X:XX)<br>XX<br>XX<br>XX<br>XX<br>XX | (%X;XX)<br>(%X;XX)<br>XX<br>XX<br>XX |
| Active Suicidal Ideation with Specific Plan | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Suicidal Behavior<br>Actual Attempt | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Interrupted Attempt<br>Aborted Attempt | XX (XX.X%)<br>XX (XX.X%) | XX (XX: X%)<br>XX (XX: X%) | XX (XX.X%)<br>XX (XX.X%) |
| Preparatory Acts or Behavior | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Suicidal Ideation or Behavior<br>Subject Engaged in Non-Suicidal Self-Injurious Behavior | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |

# Repeat for Baseline Day 0, Week 4, Week 8; Add Suicide row for all visits except Screening.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. The number and percent of subjects who experience the event at least once during treatment are summarized. Subjects are counted once for each C-SSRS section and once for each C-SSRS item answered "Yes" during treatment period. "Baseline/Screening" version was used for Screening visit and "Since Last Visit" was used for all other visits.

Reference Listing: 16.2.9.8



**premier** research

| Body System<br>Category | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Screening<br>Skin | | | |
| Normal | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| Abnormal (NCS) | (%X:X%) | XX (XX.X%) | (%X:XX) XX |
| Abnormal (CS) | XX (XX:X%) | XX (XX.X%) | (XX:X%)<br>XX |
| Missing | XX (XX.X%) | XX (XX.X%) | (%X:XX) |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Lungs | | | |
| Normal | XX (XX.X%) | XX (XX.X%) | (%X:X%) |
| Abnormal (NCS) | (XX.XX) | (%X:XX) | (%X:XX) |
| Abnormal (CS) | XX (XX:X%) | XX (XX.X%) | (%X:XX) |
| Missing | (XX.XX) | (%X:XX) XX | (%X:XX) |
| Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Heart | | | |
| Normal | XX (XX:X%) | XX (XX.X%) | (%X:X%) |
| Abnormal (NCS) | XX (XX.X%) | XX (XX.X%) | (%X:X%)<br>XX |
| Abnormal (CS) | (XX.XX) | (%X:XX) XX | (%X:XX) |
| Missing | XX (XX:X%) | XX (XX.X%) | (XX:X%)<br>XX |
| Total | (%X XX) XX | (%X XX) XX | (%X XX) XX |

Repeat for Baseline, Week 8

Abbreviations: CS = clinically significant; NCS = not clinically significant.

Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Baseline is the last non-missing measurement taken before the first application of study drug.

Reference Listing: 16.2.9.4



| ATC Class Level 4<br>Preferred Term | Roflumilast Foam 0.3% (N=XX) | Vehicle<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|
| Subjects with at least 1 Concomitant Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 Preferred Term 1 Preferred Term 2 Preferred Term 3 | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| ATC Class 2 Preferred Term 1 Preferred Term 2 Preferred Term 2 | (%XXX%)<br>XX (XXX%)<br>XX (XXXX%)<br>XX (XXXX%) | (%XXXX)<br>XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (%XXX)<br>XX (XXXX)<br>XX (XXXX)<br>XX (XXXXX)<br>XX (XXXXXXXXXX |

Abbreviations: ATC = Anatomic Therapeutic Chemical; PT = preferred term; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

first application of study drug. Medications are displayed by alphabetical order of ATC Level 4 classification, then descending frequency of PT within ATC, and then alphabetically by PT. Subjects were counted only once for each ATC and PT. Note: Percentages are n/Number of subjects in the Safety population within treatment received and overall\*100. Medications were coded using WHO-DDE Global B3 version September 2019. Concomitant medications are all medications that were continuing or starting after Reference Listing: 16.2.9.6

Programming note: ATC & PT text should be presented as is from dataset.

Table 14.4.1.1 Summary of Pharmacokinetic Concentration Results by Study Visit and Time Point PK Population

| Study Visit Time Point Statistic Baseline Day 0 Predose Nedian Min, Max Thour postdose NXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|
| sy 0 SD) ax stdose SD) ax stdose SD) ax stdose SD) SD) SD) |
| ay 0 SD) ax stdose SD) ax stdose SD) ax SD) SD) |
| sy 0 SD) ax stdose SD) ax stdose ax scostdose |
| sy 0 SD) ax stdose SD) ax stdose solo |
| sy 0 SD) ax stdose SD) ax stdose ostdose |
| SD) ax stdose SD) ax stdose stdose |
| ay 0 SD) ax stdose SD) ax |
| ay 0 SD) ax stdose SD) |
| sy 0<br>SD)<br>ax<br>stdose<br>SD) |
| ay 0<br>SD)<br>ax<br>stdose |
| ay 0<br>SD)<br>ax<br>stdose |
| ay 0<br>SD)<br>ax<br>stdose |
| ay 0<br>SD) |
| ay 0<br>SD) |
| ay 0<br>SD) |
| ay 0 |
| it<br>sy 0<br>SD) |
| nt<br>sy 0 |
| nt<br>sy 0 |
| nt<br>S<br>Sy O |
| <b>F</b> |
| ıt |
| tt. |

Programming note: Repeat for Baseline: 4 hours postdose, 6 hours postdose, and 24 hours postdose; Week 4: Predose, 1 hour postdose, 2 hours postdose, 4 hours postdose, 6 hours postdose, and 24 hours postdose; Week 8: Predose. Note: Subjects are summarized by treatment received. Results at the predose time point that occurred after dosing are excluded from this summary. Reference Listing: 16.2.5.6

Table 14.4.1.2 Summary of Pharmacokinetic Parameters by Study Visit PK Population

**premier** research

| Parameter: XXXXXXXX | |
|---------------------|-----------------------|
| Study Visit | Roflumilast Foam 0.3% |
| Statistic | (N=XX) |
| Baseline Day 0 | |
| L | × |
| Mean (SD) | XX.X (XX.XX) |
| Median | XXX |
| Min, Max | ×××× |
| Week 4 | |
| L | × |
| Mean (SD) | XX.X (XX.XX) |
| Median | XXX |
| Min, Max | ×××× |
| Week 8 | |
| C | × |
| Mean (SD) | XX.X (XX.XX) |
| Median | XXX |
| Min, Max | X, X |

Programming note: Continue for all parameters.

Note: Subjects are summarized by treatment received. Reference Listing: 16.2.5.7



## 14.3. Planned Listing Shells

Listing 16.2.1.1 Subject Disposition All Subjects

| Subject ID XXXXXX | Randomized | Did Subject Complete Study? [ eCRF Deriv Yes Yes | lbject<br>Study? [1]<br>Derived<br>Yes | Date of Completion/ Early Termination (Study Day) DDMMMYYYY | Date of Last Study Visit (Study Day) DDMMMYYYY (XX) | Reason for Early<br>Termination [2] | Cause of Death/<br>Date of Death | Early Termination Due<br>to COVID-19 Disruption |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | × × | × × | DDMMMYYYYY (XX) | DDMMMYYYY (XX) | | | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | S ON | √ es | (XX)<br>DDMMMYYYYY<br>(XX) | DDMIMINTTTT (XX) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | |
| XXXXX | XXXXXX | <u>8</u> | Yes | DDMMMYYYY<br>(XX) | DDMMMYYYY (XX) XXXXXX | XXXXX | XXXXX/<br>DDMMMYYYY | ×× |

Abbreviations: COVID-19 = novel coronavirus disease-19; eCRF = electronic case report form.

Note: Study day is calculated relative to the date of first application of study drug.

[1] The derived completion status is based on a subject completing the Week 8 visit; this is what is used in the subject disposition summary. The eCRF completion status is based on a subject completing the Week 8 visit; this is what is used in the eCRF.

[2] Based on the eCRF.

Programming Note: If reason for early termination is Other, concatenate the specify text as follow-up; "Other: XXXXXXXXXX". If reason for early termination is lost to follow-up, concatenate with date of last contact as follows-up; date of last contact: DDMMMYYYY?".



Listing 16.2.1.2 Subject Visits All Subjects

| Treatment<br>Received | Was Visit<br>Performed? | Visit | Visit Date<br>(Study Day) | If Visit not Performed,<br>COVID-19 Disruption<br>Contributed to Missed Visit |
|---|---|---|---|---|
| | Yes | XXXXXX | DDMMMYYYY (XX) | |
| | Yes | XXXXXX | DDMMMYYYY (XX) | |
| | Yes | XXXXXXXX | DDMMMYYYY (XX) | |
| | o<br>N | XXXXXXX | | Yes |
| | Yes | XXXXXX | DDMMMYYYY (XX) | |
| | Yes | XXXXXX | DDMMMYYYY (XX) | |

Abbreviation: COVID-19 = novel coronavirus disease-19. Note: Study day is calculated relative to the date of first application of study drug.



**premier** research

| | | Subject Screen | | _ | Date/Time (Study Day) of: | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Was Subject<br>Rescreened? | Failed<br>due to COVID-19<br>Disruption | Randomized<br>Treatment | Screening | Informed Consent | If Adolescent,<br>Date of Written<br>Assent | All Inclusion<br>Criteria Met?<br>[1] | Any Exclusion<br>Criteria Met?<br>[2] |
| XXXXX | × | | XXXXX | DDMMMYYYY<br>(X-) | DDMMMYYYY/hh:m<br>m<br>(-X) | | ,<br>≺es | o<br>Z |
| XXXXX | × | × | | DDMMMYYYY | | | No: 05, 13 | N <sub>O</sub> |
| XXXXX | × | × | | DDMMMYYYY | DDMMMYYYY/hh:m<br>m | | No: 02 | o<br>Z |
| XXXXX | ×× | | XXXXXX | DDMMMYYYY<br>(X-) | | DDMMMYYYY<br>(-X) | Yes | Yes: 02 |
| XXXXX | × | | XXXXXX | DDMMMYYYY<br>(X-) | DDMMMYYYY<br>(-X) | | Yes | o<br>Z |
| XXXXX | × | | XXXXXX | DDMMMYYYY<br>(-X) | DDMMMYYYY<br>(-X) | | Yes | o<br>Z |

Abbreviation: COVID-19 = novel coronavirus disease-19.

Note: Study day is calculated relative to the date of first application of study drug. If a subject is a rescreen, the latest date of screening and informed consent are presented. [1] 02 = Males and females ages 12 years and older (inclusive) at the time of consent or assent (for adolescents); 05 = A Psoriasis Scalp Severity Index (PSSI) score of at least 6 at Baseline; 13 = Subjects are considered reliable and capable of adhering to the Protocol and visit schedule according to the Investigator judgment. [2] 02 = Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED. Programming note: If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma as shown above. Decode any relevant criteria in the footnotes as shown in the example. If no criteria are present for a column, remove the [1] and/or [2] from the column header. Time is only collected for informed consent. If time is missing, display as shown in the shell. If subject rescreens, populate the latest date of screening and informed consent.





**premier** research

| Subject ID | Treatment<br>Received | Date of Protocol<br>Violation Collection<br>(Study Day) Event Type | Event Type | Violation<br>Level | iolation<br>Level Description | COVID-19<br>Related | COVID-19 COVID-19<br>Related Infection | COVID-19<br>Infection Action/Resolution |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | DDMONYYYY (XX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY (XX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor<br>Major | Minor XXXXXXXX<br>Major XXXXXXXXXXXXXX | | | |
| XXXXX | XXXXX | DDMONYYYY (XX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMONYYYY (XX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXX | XXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | × | × | |
| XXXXX | XXXXXX | DDMONYYYY (XX) XXXXXXXXXXXX | XXXXXXXXXX | XXXXX | xxxxx xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | × | × | |

Abbreviation: COVID-19 = novel coronavirus disease-19. Note: Study day is calculated relative to the date of first application of study drug.

Programming note: the structure of this listing may change depending on the information in the protocol deviations file.





Listing 16.2.3.1 Subject Randomization All Subjects

| l | | | Ra | Randomization | |
|---|---|---|---|---|---|
| ⊢ " | Treatment<br>Received | Randomized<br>Treatment | Date/Time | Number | Stratification ID |
| | XXXXX | XXXXX | DDMMMYYY/<br>hh:mm | XXXX | ××× |
| ^ | XXXXXX | XXXXX | DDMMMYYY/<br>hh:mm | XXXX | ××× |



Analysis Populations Listing 16.2.3.2 All Subjects

| Primary Reason(s) for Exclusion [7] | Subject missed Week 8 disease assessment specifically due to COVID-19 disruptions. | | Subject did not receive at least 1 dose of IP. |
|---|---|---|---|
| ¥ © | × | × | × |
| PRU4-mITT<br>[5] | ×× | × | × |
| PRU4-ITT<br>[5] | × | × | ×× |
| SPRU4-ITT SPRU4-mITT [4] | × | ×× | ×× |
| SPRU4-ITT<br>[4] | Yes | Yes | o<br>N |
| mITT<br>[3] | °Z | Yes | Š |
| <u> </u> | Yes | Yes | Yes |
| Safety<br>[1] | Yes | Yes | Š |
| Treatment<br>Received | XXXXXX | XXXXXXX | |
| Subject<br>ID | XXXXX | XXXXXX | XXXXX |

Abbreviations: COVID-19 = novel coronavirus disease-19; ITT = intent-to-treat; IP = investigational product; mITT = modified intent-to-treat; NA = not applicable; PK = pharmacokinetic; PRU4 = Subjects with WI-NRS Pruritus Score ≥4 at Baseline; SI-NRS = Scalp Itch – Numeric Rating Scale; SPRU4 = Subjects with WI-NRS Pruritus Score ≥4 at Baseline; WI-NRS = Worst Itch – Numeric Rating Scale.

[1] The Safety Population includes all subjects who are enrolled and received at least 1 confirmed dose of IP.
[2] The ITT Population includes all subjects who are randomized.
[3] The mitt population includes all subjects with the exception of subjects who missed the Week 8 S-IGA assessment specifically due to COVID-19 disruptions.
[3] The mitt population includes all randomized subjects with the exception of subjects who missed the Week 8 S-IGA assessment specifically due to COVID-19 disruptions.
[4] The SPRU4-ITT and SPRU4-mitt populations are subsets of the ITT and mitt populations, respectively, and include subjects with SI-NRS pruritus score ≥ 4 at Baseline. These populations will be used for the analyses of achievement of a 4-point reduction in SI-NRS pruritus score as compared to Baseline.

[5] The PRU4-ITT and PRU4-mITT populations are subsets of the ITT and mITT populations, respectively, and include subjects with WI-NRS pruritus score ≥ 4 at Baseline. These

populations will be used for the analyses of achievement of a 4-point reduction in WI-NRS pruritus score as compared to Baseline.
[6] The PK population includes all subjects receiving the active drug with sufficient plasma concentrations of roflumilast to define a profile, as determined by the pharmacokineticist.
[7] Applies to the Safety, ITT, and mITT populations only.





| PK Consent<br>Obtained/<br>Date of Consent | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | No | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | XXX |
|---|---|---|---|---|---|---|
| Photography<br>Consent Obtained/<br>Date of Consent | Yes/<br>DDMIMMYYYY | Yes/<br>DDMMMYYYY | o <sub>N</sub> | Yes/<br>DDMMMYYYY | Yes/<br>DDMMMYYYY | ×× |
| Race | XXXXXXX Yes/ | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| Ethnicity | XXXXXX | XXXXXX | XXXXXXX | XXXXXX | XXXXXXX | XXXXX |
| Age<br>(years)<br>[1] | × | × | × | × | × | × |
| Year of<br>Birth | <b>*</b> | *** | *** | *** | *** | * |
| Child-Bearing<br>Potential? If<br>Yes, Specify<br>Contraception | No | ON<br>N | | | N <sub>O</sub> | Yes:<br>XXXXXXX |
| Sex | × | XXXXXX No | ××× | XXX | XXXXX | XXX |
| Treatment<br>Received | XXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXX |
| Subject<br>ID | XXXXX | XXXXXX | XXXXXX | XXXXX | XXXXX | XXXXX |

Abbreviation: PK = pharmacokinetic. [1] Age at Screening.

Programming Note: If subject has multiple races, concatenate them. If child-bearing potential is Yes, concatenate type of contraception with "." as shown in the shell.



Listing 16.2.4.1.2 Baseline Characteristics All Subjects

| 3S [2] | × | × | × | × | × | × |
|---|---|---|---|---|---|---|
| WI-NRS [2] | × | × | × | × | × | × |
| SI-NRS [2] | × | × | × | × | × | × |
| B-IGA [1] | X = XXXXX | * XXXXX = X | X = XXXXX | X = X | X = X | X = XXXXX |
| S-IGA [1] | X = X | * XXXXX = X | X = X | X = X | X = X | X = XXXXX |
| BSA<br>(%) | × | × | × | × | × | ×× |
| Weight<br>(kg) | XX. | ×× | ×× | × | ×× | XXX |
| Height<br>(cm) | XX | ×× | ×× | ××× | ××× | XXX |
| Treatment<br>Received | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| Subject ID | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |

Abbreviations: B-IGA = body investigator global assessment; BSA = body surface area; S-IGA = scalp investigator global assessment; SI-NRS = Scalp Itch – Numeric Rating Scale; WI-NRS = Worst Itch – Numeric Rating Scale.

Note: Weight and % BSA affected by disease are the values at Screening. Height was collected at Baseline Day 0.

[1] For S-IGA and B-IGA, baseline is the last non-missing measurement taken before the first application of study drug. \* = Screening visit was used as baseline.

[2] For SI-NRS and WI-NRS, baseline is the last non-missing measurement taken on or before the day of first application of study drug.

Programming Note: For S-IGA and B-IGA scores, if VISIT is not Baseline Day 0 for the record where ABLFL=Y, then add a \* to the end of the concatenated numeric + text result, as shown in the shell.



**premier** research

| tory Conditions | Start Date (Study Day)/<br>End Date (Study Day) | DDMMMYYYY (X)/ DDMMMYYYY (X)/ DDMMMYYYY (X)/ DDMMMYYYY (X)/ DDMMMYYYY (X)/ | DDMMMYYYY (X)/<br>Ongoing |
|---|---|---|---|
| Other Medical History Conditions | System Organ Class/<br>Preferred Term/<br>Verbatim Term | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | Type of History | Topical Corticosteroids: Yes/<br>Topical Vitamin D Derivatives: No | Topical Corticosteroids: Yes/<br>Topical Vitamin D Derivatives: No |
| | Treatment Subject History of Psoriasis<br>Received Involvement | Knees/Elbow: Yes/<br>Genitalia: No | Knees/Elbow: Yes/<br>Genitalia: No |
| | Treatment<br>Received | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX XXXXXX |
| | Subject<br>ID | ××××××××××××××××××××××××××××××××××××××× | XXXXX |

Abbreviation: MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study day is calculated relative to the date of first application of study drug. Medical history was coded using MedDRA version 23.0. Only subjects with medical history recorded are listed.

Programming note: SOC & PT text should be presented as is from the dataset.



Listing 16.2.5.1 Study Drug Application at the Study Site All Subjects

| Kit Number/<br>Can ID | ××× | XXX<br>XXX | XXX | <b>{</b> | XXXX | ××× | ×××<br>××× |
|---|---|---|---|---|---|---|---|
| Reason Pre- and/or<br>Post-Application<br>Can Weight<br>Measurement not<br>Performed | | | | | | | XXXXXXXXXXXX |
| Applied<br>Dose<br>(g) | × | ×× | × | | × | × | |
| Post-Application<br>Can Weight (g)<br>Measurement | × | XX.X | × | | × | × | Not Done |
| Pre-Application<br>Can Weight (g)<br>Measurement | × | X.XX | × | | × | × | × |
| Date/Time of<br>Application<br>(Study Day) | DDMMMYYYY/HH:MM (X) | DDMMMYYYY/HH:MM (XX) | DDMMMYYYY/HH:MM (XX) | | DDMMMYYYY/HH:MM (X) | DDMMMYYYY/HH:MM (XX) | DDMMMYYYY/HH:MM (XX) |
| Study<br>Visit | XXXXX | XXXXX | XXXXXX | XXXXX | XXXXXX | XXXXX | XXXXX |
| Was Study<br>Drug<br>Application<br>Performed at<br>Study Site? | Yes | | | No: XXXXXX | Yes | | |
| Treatment<br>Received | XXXXXX Yes | | | | XXXXXX Yes | | |
| Subject<br>ID | ×× | | | | XXXX | | |

Note: Study day is calculated relative to the date of first application of study drug.

Programming note: For Pre & Post-Application Can Weight Measurement columns, if the weight measurement is not performed, set the value to be "Not Done". If drug not administered, concatenate reason (COVID-19 Disruption or other specify text) as shown in shell.



Listing 16.2.5.2 Cans All Subjects

| Subject ID | | Treatment Kit Number/<br>Received Can ID | Can Dispensed?<br>Reason if No | Can Dispensed? Date Dispensed<br>Reason if No (Study Day) | Dispense<br>Weight (g) | Dispense Can Returned?<br>Weight (g) Reason if No | Date Returned<br>(Study Day) | Return<br>Weight (g) |
|---|---|---|---|---|---|---|---|---|
| ×××× | XXXXXX | /xxxx | Yes | ррмммүүүү (X) | × | Yes | DDMMMYYYY (X) | ×:<br>×: |
| | | XXXXX<br>XXXXX | Yes | DDMMMYYYY (X) | ×× | Yes | DDMMMYYYY (X) | ××× |
| | | ××××× | Yes | DDMMMYYYY (X) | Q | Yes | DDMMMYYYY (X) | Q |
| XXXX | XXXXXX | XXXX | No: XXXXX | | | No: XXXXX | | |

Abbreviation: ND = not done. Note: Study day is calculated relative to the date of first application of study drug.

Programming note: within subject, sort by dispense date, return date, kit number and CANID.



Listing 16.2.5.3 Diary Dispensation All Subjects

| Date Returned<br>(Study Day) | DDMMMYYYY (X)<br>DDMMMYYYY (X) | | |
|---|---|---|---|
| Reason Diary<br>not Returned | | XXXXXXXXX | XXXXXXXX |
| Diary Returned Reason Diary<br>and Reviewed? not Returned | Yes | N <sub>o</sub> | ON N |
| Diary<br>Returned<br>Visit | XXXXXX | XXXXX | XXXXX |
| Date Dispensed<br>(Study Day) | DDMMMYYYY (X)<br>DDMMMYYYY (X) | DDMMMYYYY (X) | |
| Diary<br>Dispensed? | Yes | Yes | o<br>Z |
| Diary<br>Dispensation<br>Visit | XXXXXX | XXXXXX | XXXXX |
| Treatment<br>Received | XXXXX | | XXXXX |
| Subject ID | XXXX | | XXXX |

Note: Study day is calculated relative to the date of first application of study drug.



Listing 16.2.5.4 Compliance (CRF) All Subjects

| ubject ID | Treatment<br>Received | Study<br>Visit | Subject Compliant with<br>Medication? | Date of Compliance<br>Check (Study Day) | Compliance [1] | Overall<br>Compliance [2] | Overall Was Subject Retrained if not Check (Study Day) Compliance [1] Compliance [2] Compliant with Medication |
|---|---|---|---|---|---|---|---|
| | XXXXX | XXXXXX | XXX | DDMMMYYYY (X) | % % X X X X X X X X X X X X X X X X X X | %X:XX | |
| <i>\</i> | XXXXXX | XXXXX<br>XXXXX<br>XXXXX | × ×× | DDMMMYYYY (X) | % %%<br><: ×:×<br>×: × | %X:XX | |
| | | XXXXXXX | <b>*</b> × | | 87 47 | | XX |

Abbreviations: IP = investigational product; CRF = case report form. Note: Study day is calculated relative to the date of first application of study drug.

[1] This data comes from CRF page, unless otherwise specified.

[2] Overall compliance was calculated based on number of applications divided by the expected number of IP applications for each subject. Number of expected IP applications was calculated as number of days between first and last application of IP (last treatment date - first treatment date + 1). Number of IP applications was calculated as number of expected IP applications - missed IP applications as collected in the CRF.

Programming note: Populate overall compliance only for the first visit.



Listing 16.2.5.5 Missed Doses All Subjects

**premier** research

| Reason for Missed Dose | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|
| Missed Dose due to<br>COVID-19<br>Disruption? | 0 N<br>N | Yes | 0 Q |
| Date of Missed Dose<br>(Study Day) | DDMMMYYYY (X) | DDMMMYYYY (X) | DDMMMYYYY (X) |
| Study<br>Visit | ××××× | XXXXXX | XXXXXX<br>XXXXXX |
| Treatment<br>Received | XXXXX | XXXXXX | XXXXX |
| Subject ID | XXXXX | XXXXXX | ××××× |

Abbreviation: COVID-19 = novel coronavirus disease-19.

Note: Study day is calculated relative to the date of first application of study drug.

Programming note: Only subjects with missed doses should be presented in this listing.



| Subject<br>ID | PK Sa<br>Treatment at this<br>Received if No | PK Sample Collected Treatment at this Visit? Reason Received if No | Study Visit | PK Sample<br>Collected<br>Pre-Dose | PK Collection<br>Time Point | Date/Time of<br>Assessment<br>(Study Day) | Accession<br>Number | BSA Treated at<br>the Time of PK<br>Sample Collection | Roflumilast<br>Concentration<br>(unit) |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | XXXXXX | XX | XXXXX | DDMMMYYY/ | XXXXX | %X:XX | XXX |
| | | | XXXXXX | ×× | XXXXX | DDMMMYYY/ | XXXXX | % XX | XXX |
| | | | XXXXXX | ×× | XXXXX | DDMMMYYY/ | XXXXX | % XX | XXX |
| | | No: XXXXXXX | XXXXX | × | XXXXX | HH:MIMI (X) | | | |

Abbreviation: BLQ = Below the limit of quantification; BSA = body surface area; PK = pharmacokinetic. Note: Study day is calculated relative to the date of first application of study drug.




| Subject | Treatment | Study Visit | AUC <sub>0-t</sub> | AUC <sub>tau</sub> | T <sub>max</sub> | T <sub>lag</sub> | T <sub>last</sub> | C <sub>max</sub> | C <sub>min</sub> |
|---|---|---|---|---|---|---|---|---|---|
| D | Received | | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) | (unit) |
| XXXX | XXXXX | XXXXXX<br>XXXXXX<br>XXXXXX | *** | *** | *** | *** | *** | *** | *** |

Abbreviation: PK = pharmacokinetic.

Programming note: The above parameters are expected. However the final parameters provided by the pharmacokineticist will be listed and may be different than shown.



Listing 16.2.6.1 Scalp Investigator Global Assessment (S-IGA) All Subjects

| Subject<br>ID | Randomized<br>Treatment | Was Assessment<br>Completed? Reason<br>if No | If Yes, Telemedicine<br>or Delay in<br>Assessment<br>Collection [1] | Study Visit | Date/Time of<br>Assessment<br>(Study Day) | Result | Result Text Result | Change<br>from<br>Baseline | S-IGA<br>Success<br>[2] | 1 1 |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXXX | Yes | No | XXXXXXX | DDMMYYYY/hh:mm | × | XXXXXXXXX | | | |
| | | Yes | Yes: Delay in<br>Assessment<br>Collection | XXXXXX | DDMMMYYYY/hh:mm<br>(X) | × | XXXXXXXX | × | Yes | |
| | | No: COVID-19<br>Disruption | | XXXXXXX | | | | | | |
| | | Yes | °Z | XXXXXX | DDMMMYYYY/hh:mm<br>(X) | × | XXXXXXXX | × | Yes | |
| XXXXXX | XXXXXX | Yes | Yes: Assessment<br>Completed via<br>Telemedicine | XXXXXX | DDMMMYYYYY/hh:mm<br>(X) | × | XXXXXXXX | | | |
| | | No: XXXXXXXX | | XXXXXXX | DDMMMYYYY/hh:mm<br>(X) | | | | | |

Abbreviations: COVID-19 = novel coronavirus disease-19; S-IGA = scalp investigator global assessment.

Note: Study day is calculated relative to the date of first application of study drug. Baseline is the last non-missing measurement taken before the first application of study drug. Change from

baseline is calculated as Result – Baseline. [1] Due to COVID-19 disruption. [2] S-IGA Success ("Yes") is defined as an S-IGA score of "Clear" or "Almost Clear" plus a ≥2-grade improvement from baseline at Weeks 2, 4, 8, and 9; "No" otherwise.

Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell. For the "If Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".





Listing 16.2.6.2 Body Investigator Global Assessment (B-IGA) All Subjects

Programming note: Same as shell 16.2.6.1. Update any instances of S-IGA to B-IGA.



Listing 16.2.6.3 Psoriasis Scalp Severity Index (PSSI) All Subjects

| Subject<br>ID | Randomized<br>Treatment | Was<br>Assessment<br>Completed?<br>Reason if No | If Yes,<br>Telemedicine or<br>Delay in<br>Assesment<br>Collection [1] | Study<br>Visit | Date/Time of<br>Assessment<br>(Study Day) | Test | Numeric<br>Result | Text Result | Change<br>from<br>Baseline | PSSI-50 [3]/<br>PSSI-75 [4]/<br>PSSI-90 [5] |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | Yes | No | XXX | DDMMMYYYY/hh:mm | Erythema | 7 | XXXX | | |
| | | | | | (X) | Induration | 2.0 | XXXXX | | |
| | | | | | | Desquamation<br>Sum of Severity | N 0 | XXXX | | |
| | | | | | | Rating<br>Extent of Scalp | 2 | | | |
| | | | | | | Affected | ı | | | |
| | | | | | | PSSI Total Score [3] | 12 | | | |
| | | Yes | Yes: Delay in<br>Assessment | XXX | DDMMMYYYY/hh:mm<br>(X) | Erythema | 2 | XXXXX | × | |
| | | | | | | Induration | က | XXXX | × | |
| | | | | | | Desquamation | 2 | XXX | × | |
| | | | | | | Sum of Severity | 7 | | × | |
| | | | | | | Kating<br>Extent of Scalp | 2 | | × | |
| | | | | | | Affected<br>PSSI Total Score [2] | 41 | | × | XX/XX/XX |

Abbreviations: COVID-19 = novel coronavirus disease-19; PSSI = Psoriasis Scalp Severity Index.

Note: Study day is calculated relative to the date of first application of study drug. Baseline is the last non-missing measurement taken before the first application of study drug. Change from baseline is calculated as Result - Baseline.

[1] Due to COVID-19 disruption.
[2] PSSI total score is calculated as (erythema score + induration + desquamation) × extent of scale affected. The score ranges from 0 to 72. Erythema, induration, and desquamation are scored on a scale of 0 to 4, where 0 = absent and 4 = severest possible; extent of scale affected is scored on a scale of 0 to 6, where 0 = 0% of involved area and 6 = 90-100% of involved area.
[3] PSSI-50 is populated with "Yes" when there is an achievement of a 56% reduction in PSSI total score from baseline.
[4] PSSI-75 is populated with "Yes" when there is an achievement of a 76% reduction in PSSI total score from baseline.
[5] PSSI-90 is populated with "Yes" when there is an achievement of a 90% reduction in PSSI total score from baseline.

Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell for Listing 16.2.6.1. For the "if Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".

Only populate PSSI-50, PSSI-75, and PSSI-90 on PSSI Total Score row.



Listing 16.2.6.4 Scalp Itch – Numeric Rating Scale (SI-NRS) All Subjects

| SI-NRS<br>Success<br>(baseline ≥ 4)<br>[2] | Yes | Yes | Yes | |
|---|---|---|---|---|
| Change from (<br>Baseline | × | ×× | × | |
| Result | o× | ×× | × | × |
| Date/Time of<br>Assessment<br>(Study Day) | DDMIMMYYYY/hh:mm (X) | DDMMMYYYY/hh:mm (X) DDMMMYYYY/hh:mm (X) | DDMMMYYYY/hh:mm (X) | DDMMMYYYY/hh:mm (X) |
| Study Visit | XXXXXX<br>XXXXXX | XXXXXXX | XXXXXX | XXXXXXX |
| If Yes, Telemedicine or<br>Delay in Assessment<br>Collection [1] | 0 0<br>Z Z | No<br>Yes: Delay in | Assessment Collection<br>No | No |
| Was Assessment<br>Completed?<br>Reason if No | Yes<br>Yes | Yes<br>Yes | Yes | Yes<br>No: XXXXXX |
| Randomized<br>Treatment | XXXXXX | | | XXXXXX |
| Subject ID | XXXXX | | | XXXXXX |

Abbreviations: COVID-19 = novel coronavirus disease-19; SI-NRS = Scalp Itch – Numeric Rating Scale.

Note: Study day is calculated relative to the date of first application of study drug. Subjects rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher score indicates greater itch intensity. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as Result - Baseline.

[1] Due to COVID-19 disruption.
[2] SI-NRS Success is defined as achievement of a 4-point reduction in SI-NRS pruritus score at Weeks 2, 4, 8, and 9 compared to baseline, calculated only for subjects with a pruritus score of  $\geq 4$  at baseline.

Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection". Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell for Listing 16.2.6.1. For the "If Yes, Telemedicine or Delay in



Listing 16.2.6.5 Psoriasis Symptoms Diary (PSD) All Subjects

| Change from<br>Baseline | |
|---|---|
| Result | - 0 0 4 0 − 0 0 4 0 × |
| Question [2] | How severe was your psoriasis-related itching? How bothered were you by your psoriasis-related stinging? How severe was your psoriasis-related stinging? How bothered were you by your psoriasis-related burning? How bothered were you by your psoriasis-related burning? How bothered were you by your psoriasis-related burning? How bothered were you by your psoriasis-affected skin cracking? How bothered were you by your psoriasis-affected skin cracking? How severe was your psoriasis-related pain? How bothered were you by your psoriasis-affected pain? How bothered were you by your psoriasis scaling? How bothered were you by your psoriasis scaling? How noticeable did you think the color of your psoriasis-affected skin was? How much did you try to hide your psoriasis affected Skin? How much did your psoriasis cause you to avoid activities with other people? How embarrassed were you because of your psoriasis?? Total Score [3] |
| Date of Assessment<br>(Study Day) | DDMMMYYYY (XX) |
| Study<br>Visit | XXXXX |
| If Yes,<br>Telemedicine or<br>Delay in<br>Assessment<br>Collection [1] | <u>o</u> 2 |
| Assessment<br>Completed?<br>Reason if No | √es |
| Randomized<br>Treatment | XXXXX |
| Subject<br>ID | ×<br>× |

Abbreviations: COVID-19 = novel coronavirus disease-19; PSD = Psoriasis Symptoms Diary

Note: Study day is calculated relative to the date of first application of study drug. Subjects rate the severity of symptoms or how bothersome the symptoms are on an 11-point scale ranging from 0 to 10. Higher score indicates more severe symptoms. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is

calculated as Result - Baseline.

[1] Due to COVID-19 disruption.
[2] These questions are based on the psoriasis symptoms over the past 24 hours.
[3] Total score is calculated as sum of all 16 questions. The total score ranges from 0 to 160. If 1 or more items are missing, the score is not calculated.

Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell for Listing 16.2.6.1. For the "If Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".



## Listing 16.2.6.6 Psoriasis Area Severity Index (PASI)/Modified PASI (mPASI) All Subjects

| Change<br>from<br>Baseline | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Text Result | XXXX | XXXX | ××× | | | | | XXXX | XXX | XXXX | | | | | | |
| Numeric<br>Result | 2 | 2 | 2 | ××× | | | | 2 | 2 | 2 | ×:× | | | | | ×× |
| Test | Erythema | Induration | Desquamation | % Area Affected | Area Lesion score | Degree of Involvement | Head PASI Score | Erythema | Induration | Desquamation | % Area Affected | Area Lesion score | Degree of Involvement | Arm PASI Score | | PASI Total Score [2]<br>mPASI Total Score [3] |
| Area | Head | | | | | | | Arm | | | | | | | sba | ₹ |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/<br>hh:mm (X) | | | | | | | | | | | | | | Repeat the same for Trunk, Legs | |
| Study<br>Visit | XXX | | | | | | | | | | | | | | Repeat the | |
| If Yes,<br>Telemedicine or<br>Delay in<br>Assessment<br>Collection [1] | o <sub>N</sub> | | | | | | | | | | | | | | | |
| Was<br>Assessment<br>Completed?<br>Reason if No | Yes | | | | | | | | | | | | | | | |
| Randomized<br>Treatment | XXXXXX | | | | | | | | | | | | | | | |
| Subject<br>ID | XXXXX | | | | | | | | | | | | | | | |

Note: Study day is calculated relative to the date of first application of study drug. Baseline is the last non-missing measurement taken before the first application of study drug. Change Abbreviations: COVID-19 = novel coronavirus disease-19; mPASI = modified Psoriasis Area Severity Index; PASI = Psoriasis Area Severity Index. from baseline is calculated as Result – Baseline.

[1] Due to COVID-19 disruption.

[2] PASI total score is calculated as  $(0.1 \times [Eh + Th + Sh] \times Ah) + (0.2 \times [Ea + Ta + Sa] \times Aa) + (0.3 \times [Et + Tt + St] \times At) + (0.4 \times [El + Tl + Sl] \times Ah)$  where E, T, and S are erythema, thickness, and scaling, respectively, scored on a scale of 0 to 4, A is estimated area of skin involved, graded on a scale of 0 to 6, and h, e, t, and l are head, arms, trunk, and legs, respectively. The range of total score is 0 to 72.

[3] mPASI total score is calculated same as PASI above, except that for subjects with < 10% of any particular involved anatomic area, the mPASI will be calculated using the actual percentage of the anatomical area involved rather than the 0 to 6 estimated area score (e.g., 0.1 for 1%, 0.2 for 2%, 0.3 for 3%, ... 0.9 for 9%).

Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell for Listing 16.2.6.1. For the "If Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".

**premier** research



| | | ************************************** | If Yes, Telemedicine | | | | |
|---|---|---|---|---|---|---|---|
| | Randomized | Completed? | Or Delay III<br>Assessment | | Date/Time of | | Change from |
| Subject ID | Treatment | Reason if No | Collection [1] | Study Visit | Assessment (Study Day) | Result | Baseline |
| XXXXX | XXXXXX | Yes | No. | XXXXXX | DDMMMYYYY/hh:mm (X) | × | |
| | | Yes | No | XXXXXX | DDMMMYYYY/hh:mm (X) | × | × |
| | | Yes | Yes: Delay in | XXXXXX | DDMMMYYYY/hh:mm (X) | × | × |
| | | | Assessment | | | | |
| | | Yes | No | XXXXXXX | DDMMMYYYY/hh:mm (X) | × | × |
| XXXXX | XXXXXX | Yes | Yes: Assessment | XXXXXXX | DDMMMYYYY/hh:mm (X) | × | |
| | | | Telemedicine | | | | |
| | | No: XXXXXX | | XXXXXXX | DDMMMYYYY/hh:mm (X) | | |

Abbreviations: COVID-19 = novel coronavirus disease-19; WI-NRS = Worst Itch - Numeric Rating Scale.

Note: Study day is calculated relative to the date of first application of study drug. Subjects rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher score indicates greater itch intensity. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as Result – Baseline. [1] Due to COVID-19 disruption.

delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Collection".

Completed via Telemedicine; Delay in Assessment Collection". Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell for Listing 16.2.6.1. For the "If Yes,



## $\label{eq:local_local} \mbox{Listing 16.2.6.8} \\ \mbox{Dermatology Life Quality Index (DLQI)/Children's DLQI (CDLQI)} \\$ All Subjects

Form Name: DLQI

| ביום השוני הרצ | וק. דרב | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | lf Yes, | | | | | |
| | | | • | Telemedicine | Ë | | | | d |
| to aid I | Randomized | Sprit. | Assessment<br>Completed? | or Delay In | Date/Time of | | Nimeric | Text | Change |
| D D | Treatment | Visit | Reason if No | Collection [1] | (Study Day) | Question | Result | Result | Baseline |
| ××× | XXXXX | XXXX | Yes | CZ | /YYYYMMMQQ | 1. Over the last week how itchy sore painful | C | Not at all | |
| | | | | | hh:mm (XX) | or stinging has your skin been? | ) | | |
| | | | | | • | 2. Over the last week, how embarrassed or self | က | Very much | |
| | | | | | | conscious have you been because of your skin? | | | |
| | | | | | | 3. Over the last week, how much has your skin | က | Very much | |
| | | | | | | interfered with you going shopping or looking | | | |
| | | | | | | after your home or garden? | | | |
| | | | | | | 4. Over the last week, how much has your skin | က | Very much | |
| | | | | | | influenced the clothes you wear? | | | |
| | | | | | | 5. Over the last week, how much has your skin | 7 | A lot | |
| | | | | | | affected any social or leisure activities? | | | |
| | | | | | | 6. Over the last week, how much has your skin | _ | A little | |
| | | | | | | made it difficult for you to do any sport? | | | |
| | | | | | | 7. Over the last week, has your skin prevented | က | Yes | |
| | | | | | | you from working or studying? If "No", over the | | | |
| | | | | | | last week how much has your skin been a | | | |
| | | | | | | problem at work or studying? | | | |
| | | | | | | 8. Over the last week, how much has your skin | 0 | Not | |
| | | | | | | created problems with your partner or any of | | relevant | |
| | | | | | | your close friends or relatives? | | | |
| | | | | | | <ol><li>Over the last week, how much has your skin</li></ol> | 0 | Not | |
| | | | | | | caused any sexual difficulties? | | relevant | |
| | | | | | | 10. Over the last week, how much of a problem | ო | Very much | |
| | | | | | | has the treatment for your skin been, for | | | |
| | | | | | | example by making your home messy, or by | | | |
| | | | | | | taking up time? | | | |
| | | | | | | DLQI Total Score [2] | 18 | | |

Programming note: Continue for other visits. If form name=CDLQI, then refer to Protocol Appendix 7 for Questions. Replace DLQI total Score with CDLQI Total Score [1] in the body of listing. Footnote will remain as is.

Abbreviations: COVID-19 = novel coronavirus disease-19; DLQI = Dermatology Life Quality Index; CDLQI = Children's Dermatology Life Quality Index.

Note: Study day is calculated relative to the date of the first application of study drug. Baseline is the last non-missing measurement taken on or before the day of first application of study drug. Change from baseline is calculated as Result – Baseline.

[1] Due to COVID-19 disruption.
[2] The DLQI total score ranges between 0-30 and calculated as sum of all the 10 questions at each visit, where "Not relevant" was recoded to 0 before calculation of this score. If 1 item is missing, it is scored as 0 for that item. If 2 or more items are missing, the score was not calculated. The CDLQI total score is calculated similar to DLQI total score.





Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell for Listing 16.2.6.1. For the "If Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



Listing 16.2.6.9

Body Surface Area (BSA) (excluding Palms and Soles)
All Subjects

| Result | %<br>XX | **** |
|---|---|---|
| Test | Coverage Area (Head) | Coverage Area (Lower Limbs) Coverage Area (Upper Limbs) Coverage Area (Trunk) BSA Result [1] BSA CRF [2] Coverage Area (Head) Coverage Area (Lower Limbs) Coverage Area (Upper Limbs) Coverage Area (Upper Limbs) Coverage Area (Trunk) BSA Result [1] BSA CRF [2] |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/hh:mm | DDMMMYYYY (XX) |
| Study Visit | XXXXXX | ×××<br>×××<br>××× |
| If Assessment<br>Not Performed,<br>did COVID-19<br>disruption cause<br>or contribute to<br>missed BSA<br>Collection? | | × |
| If Assessment<br>Performed, did<br>COVID-19<br>disruption cause<br>or contribute to a<br>delay in BSA<br>Collection? | × | × |
| Assessment<br>Performed? | ×× | ×× |
| Randomized<br>Treatment | XXXXX | |
| Subject ID | XXXXX | |

Abbreviations: BSA = body surface area; COVID-19 = novel coronavirus disease-19; CRF = case report form; ePRO = electronic patient report outcome. Note: Study day is calculated relative to the date of first application of study drug.
[1] BSA result is calculated as sum of coverage areas of head, lower limbs, upper limbs and trunk. This is derived in the ePRO.
[2] BSA captured in the CRF data.



| kþr | | | |
|---|---|---|---|
| AE Lead to Study<br>D/C? | × | × | ×× |
| Serious?/<br>en Criteria Met | × | × | XXXXXXX |
| Outcome/<br>Action Taken/ Serious?/ AE Lo<br>Other Action Taken Criteria Met D/C? | /xxxxxxxxx<br>/xxxxxxxxxx | /xxxxxxxx<br>/xxxxxxxx | /xxxxxxxxxx/<br>/xxxxxxxxxxx/ |
| CTCAE Toxicity Grade/<br>Relationship | XXXXXXXXXX<br>/XXXXXXXXX | | /XXXXXXXXX<br>/XXXXXXXXXX |
| Outcome/<br>Start Date/Time (Study Day)/ CTCAE Toxicity Grade/ Action Taken/<br>End Date/Time (Study Day) Relationship Other Actior | DDMMMYYYYY/hh:mm (X)/<br>DDMMMYYYYY/ hh:mm (X) | DDMMYYYY/ hh:mm (X)/<br>DDMONYYYY/ hh:mm (X) | DDMONYYYY/ hh:mm (X)/<br>Ongoing |
| System Organ Class/<br>Preferred Tem/<br>Verbatim Term | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| TEAE? | × | × | × |
| Subject Treatment<br>ID Received | XXXXXX XXXXX | XXXXX | |
| Subject<br>ID | XXX | XXXX | |

Abbreviations: AE = adverse event; CTCAE = Common Terminology Criteria for Adverse Events; D/C = discontinuation; IP = investigational product; MedDRA = Medical Dictionary for Regulatory Activities; TEAE = treatment emergent adverse event.

Note: Study day is calculated relative to the date of first application of study drug. AEs were coded using MedDRA version 23.0. All AEs that occur after the date/time of first application of IP will be considered TEAEs. Severity grades are reported according to the CTCAE version 4.0.

Programming note: If time missing, display "---". If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. "Other Action Taken" will be either None, Concomitant Medication, Non-drug Therapy, Hospitalization or Prolongation of Hospitalization, Discontinued Study or Other; if specify text is needed, concatenate "Other:" with the text. If no events meet the criteria for display, present "No events are reported." SOC & PT text should be presented as is from the dataset.

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



Listing 16.2.8.1.1 Clinical Laboratory Data: Clinical Chemistry All Subjects

| Comments/<br>Reason not Done | | | | | | | | ××××× |
|---|---|---|---|---|---|---|---|---|
| Accession<br>Number | XXXX | ××× | XXXX | XXXX | XXXXX | XXXX | XXXXX | XXXX |
| Result<br>Interpretation;<br>Specify CS<br>Finding | Normal | Abnormal, NCS | Normal | Normal | Abnormal, CS;<br>XXXXXXX | XXXXX | XXXXX | XXXXX |
| Reference<br>Range<br>Flag | High | | Low | | | Low | | High |
| Reference<br>Range<br>[1] | XX - XX | XX - XX | XX – XX | XX - XX | XX - XX | XX - XX | XX - XX | × - × |
| Standard<br>Results | × | × | × | × | × | × | × | 8× |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm | DDMMMYYYY/hh:mm<br>(X) | DDMMMYYYY (X) | DDMMYYYYY/hh:mm/<br>hh:mm (X) | DDMMMYYYY/hh:mm (X) |
| Study<br>Visit | XXXXX | ×××× | XXXX | ×××× | XXXX | XXXXX | XXXX | XXXX |
| Parameter (unit) | Alanine | Ammotransierase (U/L) | | | | Alkaline | Phosphatase (U/L) | |
| Subject Treatment<br>ID Received | xxxxx xxxxx | | | | | | | |
| Subject<br>ID | XXXX | | | | | | | |

Abbreviations: CS = clinically significant; NCS = not clinically significant; ND = not done.

Note: Study day is calculated relative to the date of first application of study drug. Time of assessment was provided by the central laboratory (ACM).

[1] Reference range is used to identify potentially clinically significant laboratory values.





Listing 16.2.8.1.2 Clinical Laboratory Data: Hematology All Subjects

(Same shell as Listing 16.2.8.1.1)

Listing 16.2.8.1.3 Clinical Laboratory Data: Urinalysis All Subjects

(Same shell as Listing 16.2.8.1.1)

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



Listing 16.2.8.1.4 Clinical Laboratory Data: Serum and Urine Pregnancy Test Female Subjects

| Result | XXXXXXXX<br>XXXXXXXXX | ××××××××××××××××××××××××××××××××××××××× |
|---|---|---|
| Date/Time Performed<br>(Study Day) | DDMMMYYYY/hh:mm (XX) XXXXXXXX DDMMMYYYY/hh:mm (XX) XXXXXXXXX DDMMMYYYY/hh:mm (XX) XXXXXXXXX | DDMMMYYYYY/hh:mm (XX)<br>DDMMMYYYY/hh:mm (XX) |
| Type of Test | Serum<br>Urine<br>Urine | Serum<br>Urine<br>Urine |
| Study Visit | XXXXX<br>XXXXX | × ×× ×× ×× |
| Was Pregnancy<br>Test Performed?<br>Reason if No | Yes | Yes<br>No: XXXXXXXXX |
| Treatment<br>Received | XXXXX | XXXXX |
| Subject ID | XXXX | XXXXX |

Note: Study day is calculated relative to the date of first application of study drug. Time of assessment for serum pregnancy test was provided by the central laboratory (ACM).

Programming note: If time is missing, display it as --:--



**premier** research

| Subject<br>ID | Treatment<br>Received | Tolerability<br>Assessment<br>Performed? Reason if<br>No | If Yes, Telemedicine<br>or Delay in<br>Assessment<br>Collection [1] | Study Visit | Date/Time of<br>Assessment (Study<br>Day) | Dermal Response | Other Effects |
|---|---|---|---|---|---|---|---|
| XXXXX | xxxxx xxxxx | Yes | No<br>ON | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXX = X | X = XXXXXXXX |
| | | Yes | Yes: Delay in<br>Assessment<br>Collection | XXXXX | DDMMMYYYY/hh:mm<br>(XX) | XXXXXXXX = X | XXXXXXXX = X |
| | | Yes | No | XXXXXX | DDMMMYYYY/hh:mm<br>(XX) | X = XXXXXXXX | X = XXXXXXXX |
| XXXXX | XXXXX | Yes | No | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXXX = X | XXXXXXXX = X |
| | | Yes | No | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXXX = X | XXXXXXXX = X |
| | | Yes | Yes: Assessment<br>Completed via<br>Telemedicine | XXXXX | DDMMMYYYY/hh:mm<br>(XX) | XXXXXXXX = X | XXXXXXXX = X |
| XXXXX | xxxxxx xxxxxx | Yes | No | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXXX = X | XXXXXXXX = X |
| | | Yes | No | XXXXXX | DDMMMYYYY/hh:mm | XXXXXXX = X | XXXXXXXX = X |
| | | No: COVID-19<br>Disruption | | XXXXX | (XX) | | |

Abbreviations: COVID-19 = novel coronavirus disease-19; IP = investigational product.

Note: Study day is calculated relative to the date of the first application of study drug. This assessment will be conducted by the investigator prior to the application of IP in the study site.

[1] Due to COVID-19 disruption.

Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell. For the "If Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only was COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".



| Subject<br>ID | Treatment<br>Received | Tolerability<br>Assessment<br>Performed?<br>Reason if No | If Yes,<br>Telemedicine or<br>Delay in<br>Assessment<br>Collection [1] | Study Visit | Date/Time of<br>Assessment (Study<br>Day) | Grade | Sensation Following the Application of IP |
|---|---|---|---|---|---|---|---|
| XXXXX | xxxxxx xxxxxx | Yes | o N | XXXXXX | DDMMMYYYY/hh:mm | 0 = None | No sensation |
| | | Yes | Yes: Delay in<br>Assessment<br>Collection | XXXXX | DDMMMYYYY/hh:mm<br>(XX) | 1 = Mild | Slight warm, tingling sensation; not really bothersome |
| | | Yes | No | XXXXX | DDMMMYYYY/hh:mm<br>(XX) | 2 = Moderate | Definite warm, tingling sensation that is somewhat bothersome |
| XXXXX | XXXXXX XXXXXX | Yes | No | XXXXX | DDMMMYYYY/hh:mm | 0 = None | No sensation |
| | | Yes | Yes: Assessment<br>Completed via<br>Telemedicine | XXXXX | DDMMMYYYY/hh:mm<br>(XX) | 3 = Severe | Hot tingling/stinging sensation that has caused definite discomfort |
| | | No: COVID-19<br>Disruption | | XXXXXX | | | |

Abbreviations: COVID-19 = novel coronavirus disease-19; IP = investigational product.

Note: Study day is calculated relative to the date of the first application of study drug. This assessment will be performed at baseline visit 10 to 15 minutes after the application of IP in the study site.

[1] Due to COVID-19 disruption.

**Programming note:** Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell. For the "If Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No", if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".

Statistical Analysis Plan, Sponsor Arcutis Biotherapeutics, Inc. Protocol Number ARQ-154-204 PCN Number ARCU210101



**premier** research

| Abnormal Findings/<br>Clinically Significant/<br>Description of Finding | } | × | /XXX | XXXXXX |
|---|---|---|---|---|
| BMI<br>(kg/m²) | × | × | × | |
| Height (cm) | × | | × | |
| Blood<br>Pressure (mmHg)<br>Systolic Diastolic | × | × | × | |
| Blood<br>Pressure (mmHg)<br>Systolic Diast | × | × | × | |
| Position | XX | XXXXX | XXXX | |
| Heart<br>Rate<br>(bpm) | × | × | × | |
| Temp<br>(°C) | × | × | ×× | |
| Date of<br>Assessment<br>(Study Day) | DDMMMYYYY | DDMMMYYYY | (X)<br>DDMMMYYYY | 8 |
| Study<br>Visit | XXXX | XXXX | XXX<br>XXX | |
| Vital Signs<br>Collected?<br>Reason if No | Yes | Yes | No: XXXXXX<br>Yes | |
| Treatment<br>Received | ××××× | | | |
| Subject<br>ID | XXXX | | | |

Abbreviation: BMI = body mass index; Temp = temperature.

Note: Study day is calculated relative to the date of first application of study drug.

[1] BMI is derived as (weight in kg)/[(height in cm/100)<sup>2</sup>]. Weight is collected at all visits. For visits up to Week 4, Baseline Day 0 height is used for BMI derivation. Week 8 and Week 9 BMI is derived using Week 8 height.

Programming note: Concatenate reason not done as shown in the shell.



Listing 16.2.9.3.2 Vital Signs - Weight All Subjects

**premier** research

| Abnormal Findings/<br>Clinically Significant/<br>Description of Finding | × | XXXXXX<br>XXXXX |
|---|---|---|
| Underlying Reason<br>for Weight Loss | Weight loss was a result of dieting | |
| Weight Loss<br>due to<br>Complications<br>Associated with<br>COVID-19 | 0 C<br>Z | 2 |
| Was Weight<br>Loss<br>Intentional? | X Yes | |
| Percent<br>Change in<br>Weight<br>Since<br>Baseline | × × | { |
| Weight<br>(kg) | × × | |
| Date of<br>Assessment<br>(Study Day) | DDMMMYYYY (X) | $\otimes$ |
| Study<br>Visit | XXXX | X<br>X<br>X |
| Vital Signs<br>Collected?<br>Reason if No | Kes × | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Treatment<br>Received | XXXXX | XXXXX |
| Subject<br>ID | ××× | × |

Abbreviation: COVID-19 = novel coronavirus disease-19. Note: Study day is calculated relative to the date of first application of study drug.

Programming note: Concatenate reason not done as shown in the shell. If reason for weight loss is "Other", concatenate reason as shown in the shell.



Listing 16.2.9.4 Physical Examination All Subjects

| Treatment<br>Received | Physical<br>Examination<br>Performed?<br>Reason if No | Study Visit | Date of<br>Assessment<br>(Study Day) | Body System | Result | Abnormal Findings | Clinically Significant? |
|---|---|---|---|---|---|---|---|
| XXXXXXX | Yes | XXXXXXX | DDMMMYYYY | Skin | Normal | | |
| | | | ( <del>)</del> | Lungs<br>Heart | Abnormal<br>Normal | XXXXXXX | No |
| | Yes | XXXXXXX | DDMMMYYYY | Skin | Normal | | |
| | | | ( <del>x</del> ) | Lungs<br>Heart | Abnormal<br>Normal | XXXXXXX | No |
| | No: XXXXXXX | XXXXXXX | | | | | |

Note: Study day is calculated relative to the date of first application of study drug.

Programming note: Concatenate reason not done as shown in the shell.

Listing 16.2.9.5 Medical Photography All Subjects

| Date of Assessment<br>(Study Day) | DDMMMYYYY (XX) | DDMMMYYYY (XX) | DDMMMYYYY (XX) | | DDMMMYYYY (XX) | |
|---|---|---|---|---|---|---|
| Study Visit | XXXXXX | XXXXXX | XXXXX | | XXXXXX | XXXXXX |
| If Yes, Delay in<br>Assessment<br>Collection [1] | o <sub>N</sub> | No | Yes: Delay in | Assessment<br>Collection | No | |
| Photography<br>Performed?<br>Reason if No | Yes | Yes | Yes | | Yes | No: XXXXXX |
| Treatment<br>Received | XXXXXX | | | | | |
| Subject ID | XXXXXX | | | | | |

Abbreviation: COVID-19 = novel coronavirus disease-19.

Note: Study day is calculated relative to the date of first application of study drug.

[1] Due to COVID-19 disruption.

Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell. For the "If Yes, Delay in Assessment Collection" column, do the following: if the answer to did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection".





Listing 16.2.9.6 Prior and Concomitant Medications All Subjects

| <br> | | | |
|---|---|---|---|
| Route/<br>Frequency | XXXXXXX<br>XXXXXXX | XXXXXXX | )<br>> |
| Dose (unit) | (XXX) XXX | (XXX) XXX | (XXX) XXX |
| Start Date (Study Day)/<br>End Date (Study Day) | DDMMMYYYY (X)/<br>DDMMMYYYY (X) | DDMMMYYYY (X)/<br>Ongoing | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |
| ATC Class (Level 4)/<br>Preferred Term/<br>Verbatim Term | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ************************************** |
| Indication | ××××××××××××××××××××××××××××××××××××××× | XXXXXX | XXXXX |
| Prior/<br>Freatment Concomitant<br>Received [1] | Prior | Both | Concomitant |
| | XXXXX | | |
| Country | ×××××××××××××××××××××××××××××××××××××× | | |
| Subject<br>ID | ×××× | | |

Abbreviation: ATC = anatomic therapeutic chemical; NA = Not applicable; WHO-DDE = World Health Organization-Drug Dictionary Enhanced.

Note: Study day is calculated relative to the date of first application of study drug. Medications were coded using WHO-DDE Global B3 version September 2019.

[1] Prior indicates medication that was started and stopped prior to dosing of study drug. Concomitant indicates medication that started during the treatment period. Both indicates medication that was started prior to dosing of study drug and continued during the treatment period.

Programming note: If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXXX" but just "XXXXXXX"" on the back of the standard of the control of the c





## Listing 16.2.9.7 Patient Health Questionnaire (PHQ-8)/Modified PHQ-Adolescents (PHQ-A) All Subjects

| | | | the | | яý | | | | the | | яý | | | | | ession | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Text Result | Not at all | Several days | More than half the | days | Nearly every day | Not at all | Several days | | More than half the | days | Nearly every day | | | | | Moderate depression | |
| Result | 0 | <del>-</del> | 7 | | က | 0 | _ | | 7 | | က | | | | × | 12 | |
| Question [3] | PHQ-8 1. Little interest or pleasure in doing things | 2. Feeling down, depressed, or hopeless | 3. Trouble falling or staying asleep, or sleeping | too much | <ol> <li>Feeling tired or having little energy</li> </ol> | <ol><li>Poor appetite or overeating</li></ol> | <ol><li>Feeling bad about yourself, or that you are a</li></ol> | failure, or have let yourself or your family down | 7. Trouble concentrating on things, such as | reading the newspaper or watching television | 8. Moving or speaking so slowly that other | people could have noticed. Or the opposite- | being so fidgety or restless that you have been | moving around a lot more than usual | CRF-Calculated Total Score | Total Score [4] | |
| Form<br>Name<br>[2] | PHQ-8 | | | | | | | | | | | | | | | | |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/<br>hh:mm (XX) | | | | | | | | | | | | | | | | DDMMMYYYY/<br>hh:mm (XX) |
| Study<br>Visit | XXX | | | | | | | | | | | | | | | | XXX |
| If Yes, Telemedicine<br>or Delay in<br>Assessment<br>Collection [1] | Yes: Delay in<br>Assessment<br>Collection | | | | | | | | | | | | | | | | |
| Assessment<br>Completed?<br>Reason If No | Yes | | | | | | | | | | | | | | | | No: XXXXX |
| Treatment<br>Received | ×××× | | | | | | | | | | | | | | | | |
| Subject<br>ID | ××× | | | | | | | | | | | | | | | | |

Abbreviations: COVID-19 = novel coronavirus disease-19; CRF = case report form; PHQ-8 = patient health questionnaire-8 questions; PHQ-A = patient health questionnaire-adolescents. Note: Study day is calculated relative to the date of the first application of study drug.

- [1] Due to ĆOVÍD-19 disruption.

- [2] Form name will be PHQ-8 for adults and Modified PHQ-A for adolescents.
  [3] These questions are based on the "Over the last 2 weeks, how often have you been bothered by any of the following problems?" prompt.
  [4] The total score is calculated as sum of all the 8 questions. If more than 1 item is missing the total score should not be calculated. If 1 item is missing, the total score is calculated as sum of all the 8 questions. If more than 1 item is categorized as None Minimal depression; 5-9 = Mild depression; 10-14 = Moderate depression; 15-19 = Moderately severe depression; 20-24 = Severe depression.

Programming note: Concatenate reason not done (COVID-19 Disruption or other specify text) as shown in the shell. For the "if Yes, Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Assessment Completed via Telemedicine"; if the answer to only did COVID-19 disruption cause/contribute to delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection"



**premier** research

| 1 1 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Result | × | × | × | × | ; | × | × | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | 1 = Less than | once a week<br>1 = Fleeting –<br>few seconds or | minutes<br>1 = Easily able to<br>control thoughts |
| Assessment | 1. Wish to be dead | If yes, describe: 2. Non-Specific Active Suicidal Thoughts | 3. Active Suicidal Ideation with Any Methods (not | Figure 1 Mithout Intent to Act<br>If yes, describe:<br>4. Active Suicidal Ideation<br>with Some Intent to Act | without Specific Plan If yes, describe: | 5. Active Suicidal Ideation with Specific Plan and Intent | If yes, describe:<br>Most Severe Ideation Type<br># (1-5) | Description of Ideation | Frequency | Duration | Controllability |
| Category | Suicidal<br>Ideation | | | | | | Intensity of<br>Ideation | | | | |
| Telemedicine<br>or Delay in<br>Assessment<br>Collection [1] | Yes: Delay in<br>Assessment<br>Collection | | | | | | | | | | |
| Reference<br>Period | Baseline/<br>Screening | | | | | | | | | | |
| Date/Time of<br>Assessment<br>(Study Day) | DDMMMYYYY/<br>hh:mm (XX) | | | | | | | | | | |
| Study Visit | XXXXX | | | | | | | | | | |
| Treatment<br>Received | XXXXXX | | | | | | | | | | |
| Subject<br>ID | XXXXX | | | | | | | | | | |

Programming note: Reference period will be either Baseline/Screening or Since Last Visit. Display the results following the order of C-SSRS questionnaire for all categories.

Abbreviations: COVID-19 = novel coronavirus disease-19; C-SSRS = Columbia-Suicide Severity Rating Scale.

Note: Study day is calculated relative to the date of first application of study drug. Assessments that are marked as Not Done are not included in the listing.

[1] Due to COVID-19 disruption.





Programming note: For the "Telemedicine or Delay in Assessment Collection" column, do the following: if the answer to both questions (was assessment completed via telemedicine or was delayed) is No, display "No"; if the answer to only was assessment completed via telemedicine is yes, set to "Yes: Assessment Completed via Telemedicine; if the answer to only did COVID-19 disruption cause/contribute to delay, set to "Yes: Delay in Assessment Collection"; if both are yes, set to "Yes: Assessment Completed via Telemedicine; Delay in Assessment Collection".



## **Appendix 1: Premier Research Library of Abbreviations**

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| AE | adverse event |
| ANCOVA | analysis of covariance |
| ATC | anatomical therapeutic chemical |
| B-IGA | body investigator global assessment |
| BMI | body mass index |
| BSA | body surface area |
| CDISC | Clinical Data Interchange Standards Consortium |
| CDLQI | Children's Dermatology Life Quality Index |
| CI | confidence interval |
| СМН | Cochran-Mantel-Haenszel |
| COVID-19 | novel coronavirus disease-19 |
| CRF | case report form |
| CS | clinically significant |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| DBP | diastolic blood pressure |
| DLQI | Dermatology Life Quality Index |
| eCRF | electronic case report form |
| ePRO | electronic patient report outcomes |
| FDA | Food and Drug Administration |



| Abbreviation | Definition |
|------------------|-----------------------------------------------|
| HR | heart rate |
| ICH | International Council for Harmonisation |
| ITT | intent-to-treat |
| LS | least-squares |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mPASI | Modified Psoriasis Scalp Severity Index |
| NA | not applicable |
| NCS | nonclinically significant |
| PASI | Psoriasis Scalp Severity Index |
| PD | protocol deviation |
| PE | physical examination |
| PHQ-A | Modified PHQ-9 for Adolescents |
| PHQ-8 | Patient Health Questionnaire depression scale |
| PK | pharmacokinetic |
| PP | per-protocol |
| PSD | Psoriasis Symptoms Diary |
| PSSI | Psoriasis Scalp Severity Index |
| RR | respiratory rate |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS <sup>®</sup> | a software system used for data analysis |





| Abbreviation | Definition |
|--------------|-------------------------------------------|
| SBP | systolic blood pressure |
| SD | standard deviation |
| S-IGA | scalp investigator global assessment |
| SI-NRS | scalp itch – numeric rating scale |
| SOC | system organ class |
| TEAE | treatment emergent adverse event |
| TLFs | tables, listings, and figures |
| WHO | World Health Organization |
| WHO-DD | world health organization drug dictionary |
| WI-NRS | worst itch – numeric rating scale |